Rivaroxaban versus Warfarin in Patients with Atrial Fibrillation (ROCKET AF Trial)

**DUPLICATE-ROCKET AF** 

September 14, 2021

NCT04593056

#### 1. RCT Details

#### 1.1 Title

Rivaroxaban versus Warfarin in Patients with Atrial Fibrillation (ROCKET AF trial)

#### 1.2 Intended aim(s)

To compare the risk of stroke or systemic embolism in nonvalvular atrial fibrillation (AF) patients at increased risk for stroke with rivaroxaban versus warfarin use.

## 1.3 Primary endpoint for replication

The primary outcome of the study was composite of stroke (ischemic or hemorrhage) and systemic embolism.

## 1.3.1 Required power for primary endpoint and noninferiority margin (if applicable)

The test was designed for noninferiority. The most conservative approach was chosen, selecting the lower limit, 1.46 to obtain a 95% power with a 1-sided  $\alpha$  equal to 0.025. With expected study duration was 40 months, project event rate of 2.3% per 100 patient years in the warfarin group, and 14% annual attrition rate, 405 events were selected as the prespecified target to ensure a robust statistical result.

# 1.4 Secondary endpoint for replication (assay sensitivity) and RCT finding

Major bleeding; HR = 1.04 (95% CI 0.90-1.20)

## 1.5 Trial estimate

HR = 0.79 (95% CI 0.66-0.96) comparing rivaroxaban vs warfarin (Patel et al., 2011)

## 2. Person responsible for implementation of replication in Aetion

Dureshahwar Jawaid, MPH, Ajinkya Pawar, Ph.D., and Hemin Lee, MD, MPH implemented the study design in the Aetion Evidence Platform. They are not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

# 3. Data Source(s)

United/Optum, Truven/MarketScan, Medicare

# 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

## **Design Diagram – ROCKET AF TRIAL REPLICATION**



#### 5. Cohort Identification

## 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing rivaroxaban (at a daily dose of 20mg or 15 mg) to warfarin users. The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of rivaroxaban or warfarin (index date). We will restrict the analyses to patients with a diagnosis of atrial fibrillation with risk factors for stroke or systemic embolism.

## 5.2 Important steps for cohort formation

New users (defined as no use in 180 days prior to index date) of an exposure and a comparator drug will be identified.

# 5.2.1 Eligible cohort entry dates

Rivaroxaban was approved for non-valvular atrial fibrillation on November 4, 2011.

- For Marketscan: November 4, 2011 -December 31, 2018 (end of data availability).
- For Medicare: November 4, 2011 -December 31, 2017 (end of data availability).
- For Optum: November 4, 2011 -December 31, 2019 (end of data availability).

# 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

# 5.3 Flowchart of the study cohort assembly

For rivaroxaban vs. warfarin

| | Optum | | Truven | | Medicare | |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 75,894,642 | | 200,203,908 | | 6,886,908 |
| Did not meet cohort entry criteria | -74,960,282 | 934,360 | -199,073,812 | 1,130,096 | -2,028,461 | 4,858,447 |
| Excluded due to insufficient enrollment | -92,301 | 842,059 | -95,091 | 1,035,005 | -1,551,114 | 3,307,333 |

| Excluded due to prior use of referent | -482,398 | 359,661 | -622,538 | 412,467 | -2,080,069 | 1,227,264 |
|---|---|---|---|---|---|---|
| Excluded due to prior use of exposure | -205,565 | 154,096 | -204,425 | 208,042 | -660,796 | 566,468 |
| Excluded because patient qualified in >1 exposure category | -7 | 154,089 | -26 | 208,016 | -81 | 566,387 |
| Excluded based on Age | -624 | 153,465 | 0 | 208,016 | -155 | 566,232 |
| Excluded based on Gender | 0 | 153,465 | 0 | 208,016 | 0 | 566,232 |
| Excluded based on Inclusion #1 - Age >=18 | -86 | 153,379 | -264 | 207,752 | -65 | 566,167 |
| Excluded based on Inclusion #2 & 3 - Atrial fibrillation | -83,438 | 69,941 | -129,172 | 78,580 | -348,521 | 217,646 |
| Excluded based on Inclusion #4 | -13,297 | 56,644 | -16,046 | 62,534 | -36,136 | 181,510 |
| Excluded based on Exclusion #1a - Mitral stenosis | -275 | 56,369 | -154 | 62,380 | -399 | 181,111 |
| Excluded based on Exclusion #1b - Prosthetic heart valve | -1,238 | 55,131 | -789 | 61,591 | -3,016 | 178,095 |
| Excluded based on Exclusion #1e - atrial myxoma or left ventricular thrombus | -158 | 54,973 | -35 | 61,556 | -234 | 177,861 |
| Excluded based on Exclusion #1f - Active infective endocarditis | -279 | 54,694 | -138 | 61,418 | -401 | 177,460 |
| Excluded based on Exclusion #2a - Active bleeding or bleeding history | -3,413 | 51,281 | -2,716 | 58,702 | -8,256 | 169,204 |
| Excluded based on Exclusion #2b.1 - Major Surgery | -1,564 | 49,717 | -1,561 | 57,141 | -6,484 | 162,720 |
| Excluded based on Exclusion #2b.2 - Bleeding diathesis | -1,235 | 48,482 | -885 | 56,256 | -3,832 | 158,888 |
| Excluded based on Exclusion #2b.3 - Intracranial neoplasm, AV malformation, cerebral aneurysm | -259 | 48,223 | -283 | 55,973 | -422 | 158,466 |
| Excluded based on Exclusion #2d - Thrombocytopenia | 0 | 48,223 | 0 | 55,973 | 0 | 158,466 |
| Excluded based on Exclusion #2e - Uncontrolled hypertension | -47 | 48,176 | -105 | 55,868 | -300 | 158,166 |
| Excluded based on Exclusion #3a.1 - stroke plus disabling stroke effects | -257 | 47,919 | -152 | 55,716 | -847 | 157,319 |
| Excluded based on Exclusion # 3a.2 - stroke | -103 | 47,816 | -88 | 55,628 | -642 | 156,677 |
| Excluded based on Exclusion #3b - TIA | -17 | 47,799 | -25 | 55,603 | -123 | 156,554 |
| Excluded based on Exclusion #3c - DVT & PE | -1,095 | 46,704 | -853 | 54,750 | -3,185 | 153,369 |
| Excluded based on Exclusion #3d.1 - Use of aspirin > 100 mg, #3d.2 - Use of fibrinolytic agents, #3d.3 - Use of Aspirin + thienopyridines, #3d.4 - Use of cangrelor, #3f – Use of CYP inhibitors, #3g - Use of CYP inducers | -1,020 | 45,684 | -1,024 | 53,726 | -4,503 | 148,866 |
| Excluded based on Exclusion #3h – Anemia & #3i - Pregnancy | -1,382 | 44,302 | -1,294 | 52,432 | -6,940 | 141,926 |
| Excluded based on Exclusion #3k - HIV infection | -13 | 44,289 | -7 | 52,425 | -12 | 141,914 |

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Excluded based on Exclusion #3l - Severe renal impairment | -3,281 | 41,008 | -2,012 | 50,413 | -7,391 | 134,523 |
|---|---|---|---|---|---|---|
| Excluded based on Exclusion #3m - Liver disease | -192 | 40,816 | -170 | 50,243 | -466 | 134,057 |
| Excluded based on Exclusion #4a - CCI (180 days)- ICD9 and ICD10 v2 | -40 | 40,776 | -31 | 50,212 | -400 | 133,657 |
| Excluded based on Exclusion #4b - drug addiction or alcohol abuse | -157 | 40,619 | -106 | 50,106 | -231 | 133,426 |
| Excluded based on Exclusion #4f - Non-compliance | -15 | 40,604 | -21 | 50,085 | -196 | 133,230 |
| Final cohort | | 40,604 | | 50,085 | | 133,230 |

Due to CMS cell suppression policy, all values less than 11 are denoted with \*\*

#### 6. Variables

#### 6.1 Exposure-related variables:

## Study drug:

The study exposure of interest is initiation of rivaroxaban. Initiation will be defined by no use of rivaroxaban or a comparator in the prior 6 months before treatment initiation (washout period).

# Comparator agents-

- Initiators of rivaroxaban will be compared to initiators of-
  - Warfarin

#### 6.2 Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B).

<sup>\*</sup> Medicare database includes all patients using a novel oral anticoagulant and a subset of patients using warfarin during 2011-2017.

## 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Primary Effectiveness outcomes of interest (definitions provided in **Appendix A**):

- Primary outcome: stroke (hemorrhagic, ischemic) and systemic embolism
- Secondary outcome: Individual components
  - Hospital admission for stroke (principal diagnosis position)
  - Hospital admission for systemic embolism (principal diagnosis position)

Control outcomes of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted):

1. Major bleeding

## 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the primary analysis, as it targets the relative hazard of outcomes on treatment.

For the as-treated analyses, the follow-up will start the day after initiation of rivaroxaban and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.

- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug
  (rivaroxaban and comparator) plus a defined grace period (i.e., 10 days after the end of the last prescription's days' supply in
  main analyses).
- The date of augmentation or switching from exposure to comparator or vice versa or augmentation/switching to any other NOAC (e.g. switching from rivaroxaban or warfarin to apixaban would be a censoring event);
  - o A dosage change on the index treatment does not fulfill this criterion
  - o An added treatment that is not part of the exposure or comparator group does not fulfill this criterion

For the intention-to-treat (ITT) analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

## 7. Initial Feasibility Analysis

#### **Aetion report name:**

#### For rivaroxaban vs. warfarin

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1310/results/58054/result/0">https://bwh-dope.aetion.com/projects/details/1310/results/58054/result/0</a>
Truven- <a href="https://bwh-dope.aetion.com/projects/details/1341/results/58058/result/0">https://bwh-dope.aetion.com/projects/details/1313/results/58058/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/projects/details/1341/results/58058/result/0">https://bwh-dope.aetion.com/projects/details/1313/results/58058/result/0</a>

<u>Date conducted:</u> 09/02/2020

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of study population
- Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

#### **Aetion report name:**

For rivaroxaban vs. warfarin

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1310/results/58056/result/0">https://bwh-dope.aetion.com/projects/details/1310/results/58056/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/projects/details/1341/results/58059/result/0">https://bwh-dope.aetion.com/projects/details/1310/results/58056/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/projects/details/1341/results/58059/result/0">https://bwh-dope.aetion.com/projects/details/1310/results/58056/result/0</a>

Date conducted: 09/02/2020

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 6/3/20 |
|-------------------------|------------------|----------------|---------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 6/30/20 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

## Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1310/results/57933/result/0">https://bwh-dope.aetion.com/projects/details/1310/results/57933/result/0</a>
Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/1313/results/57934/result/0">https://bwh-dope.aetion.com/projects/details/1313/results/57934/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/projects/details/1341/results/57981/result/0">https://bwh-dope.aetion.com/projects/details/1313/results/57934/result/0</a>

# Date conducted: 8/27/2020 (Medicare 8/30/2020)

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to **Appendix B**.

• Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 1,879 (1.83%) | 946 (1.84%) | 933 (1.82%) |
| Start of an additional exposure | 3,238 (3.15%) | 1,642 (3.20%) | 1,596 (3.11%) |
| End of index exposure | 71,983 (70.13%) | 36,022 (70.19%) | 35,961<br>(70.07%) |
| Specified date reached (Dec 17/Dec 18/Dec 19) | 6,822 (6.65%) | 3,196 (6.23%) | 3,626 (7.07%) |
| End of patient enrollment | 5,237 (5.10%) | 2,408 (4.69%) | 2,829 (5.51%) |
| Switch to other NOACs (for censoring) + nursing home admission | 13,477 (13.13%) | 7,104 (13.84%) | 6,373 (12.42%) |

Effectiveness research with Real World Data to support FDA's regulatory decision making

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | | |
|---|---|---|---|
| Patient Group Optum Truven Medicare | | | |
| Overall Patient Population | 98 [38-209] | 98 [44-236] | 98 [38-206] |
| Referent | 98 [38-190] | 98 [44-192] | 98 [38-188] |
| Exposure | 98 [38-231] | 119 [44-281] | 98 [38-228] |

• Report overall risk of the primary outcome.

| | Optum | MarketScan | Medicare | Pooled |
|-------------------------|-------|------------|----------|--------|
| Risk per 1,000 patients | 7.00 | 7.33 | 12.05 | 10.08 |

# **10. Final Power Assessment**

# Date conducted:

- Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.
  - For rivaroxaban vs. warfarin

# o Pooled

| Curaniania, Analysis | | | |
|---|---|---|---|
| Superiority Analysis | | Non-inferiority Analysis | |
| Number of patients matched | 102,636 | Number of patients matched | 102.626 |
| Reference | 51,318 | | 102,636 |
| | | Reference | 51,318 |
| Exposed | 51,318 | Exposed | 51,318 |
| Risk per 1,000 patients | 10.08 | Risk per 1,000 patients | - |
| Desired HR from RCT | 0.79 | | 10.08 |
| Desired in their their | 0.73 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.46 |
| Number of events expected | 1034.57088 | Number of events expected | 1034.57088 |
| Power | 0.966450516 | Power | 0.999981559 |

# o Optum

| O Optum | | | |
|---|---|---|---|
| Superiority Analysis | | Non-inferiority Analysis | |
| Number of patients matched | 17,900 | Number of patients matched | 17,900 |
| Reference | 8,950 | Reference | 8,950 |
| Exposed | 8,950 | Exposed | 8,950 |
| Risk per 1,000 patients | 7.00 | Risk per 1,000 patients | 7.00 |
| Desired HR from RCT | 0.79 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.46 |
| Number of events expected | 125.3 | Number of events expected | 125.3 |
| Power | 0.261393559 | Power | 0.562809862 |

# MarketScan

| | | • | |
|---|---|---|---|
| Superiority Analysis | | Non-inferiority Analysis | |
| Number of patients matched | 22,600 | Number of patients matched | 22,600 |
| Reference | 11,300 | | 11,300 |
| Exposed | 11,300 | Exposed | 11,300 |
| Risk per 1,000 patients | 7.33 | Risk per 1,000 patients | 7.33 |
| Desired HR from RCT | 0.79 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.46 |
| Number of events expected | 165.658 | Number of events expected | 165.658 |
| Power | 0.329138572 | Power | 0.682759594 |

## Medicare

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | 62,136 | Number of patients matched | 62,136 |
| Reference | 31,068 | Reference | 31,068 |
| Exposed | 31,068 | Exposed | 31,068 |
| Risk per 1,000 patients | 12.05 | Risk per 1,000 patients | 12.05 |
| Desired HR from RCT | 0.79 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.46 |
| Number of events expected | 748.7388 | Number of events expected | 748.7388 |
| Power | 0.897079133 | Power | 0.999353731 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 9/8/20 |
|-------------------------|------------------|----------------|---------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 9/29/20 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

# 11. Study Confidence and Concerns

<u>Deadline for voting on study confidence and listing concerns:</u>
<u>Date votes and concerns are summarized:</u>

• If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.

- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.
- After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

## 12. Register study protocol on clinicalTrials.gov

## Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

## 13. Comparative Analyses

Aetion report name:

Date conducted:

- 13.1 For primary analysis:
- 13.2 For sensitivity analyses:

# 14. Requested Results

# 14.1 <u>Table 1: Baseline characteristics before and after adjustment</u>

| Variable | Before adjus | tment | | After adjustment | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | i |
| Age categories | | | | | | |

# 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

# 14.3 <u>Table 3: Censoring events</u>

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

# 14.4 <u>Table 4: Results from primary analyses;</u>

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

# 14.5 <u>Table 5: Results from secondary analyses;</u>

Effectiveness research with Real World Data to support FDA's regulatory decision making

# 15. References

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. New England Journal of Medicine. 2011; 365(10):883-91.

| # | ROCKET-AF trial definitions | Implementation in routine care | References/Rationale | Color coding |
|---|---|---|---|---|
| | Trial details- Primary indication, 4a- Unintended S with label change | HR = 0.79 (95% CI 0.66-0.96) | Please see the following Google Drive for further details or any missing information:<br>https://drive.google.com/open?id=1WD618wrvwYiEaXzfLTcuK-VCcnb6b-gV | Criteria |
| | EXPOSURE vs. COMPARISON | | ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive Folder [link above]. ICD-9 to ICD-10 code conversions were completed using a SAS macro that implements forward/backward mapping based on the CMSICD-9 to ICD-10 mapping: <a href="https://www.nber.org/data/icd9-icd-10-cm-and-pos-crosswalk-eeneral-mutwalence-mapping.htm">https://www.nber.org/data/icd9-icd-10-cm-and-pos-crosswalk-eeneral-mutwalence-mapping.htm</a> . | Adequate mapping in claims |
| | Rivaroxaban vs. Warfarin PRIMARY OUTCOME | Rivaroxaban 20mg OR 15mg daily (if low GFR) vs. adjusted-dose warfarin | | Intermediate mapping in claims |
| | PRIMARY OUTCOME Primary endpoint of stroke (ischemic or hemorrhagic) and systemic embolism. | Measured 1 day after drug initiation in primary diagnosis position specified below and inpatient care setting: Stroke: ICD-9 discharge diagnosis codes: 430.xx Subarachnoid hemorrhage (SAH) 431.xx Intracerebral hemorrhage (ICH) 431.xx Intracerebral hemorrhage (ICH) 431.xx (excluding 434.x0) Occlusion and stenosis of precerebral arteries with cerebral infarction 434.xx (excluding 434.x0) Occlusion and stenosis of cerebral arteries with cerebral infarction 436.x Acute, but ill-defined cerebrovascular events Systemic embolism: ICD-9 discharge diagnosis code: 444.xx Arterial embolism ICD-10 discharge diagnosis code: 174.x Arterial embolism and thrombosis | For stroke: PPV of 85% or higher for ischemic stroke PPV ranging from 80% to 98% for hemorrhagic stroke PPV ranging from 80% to 98% for hemorrhagic stroke → Andrade SE, Harrold LR, Tjia J, et al. A systematic review of validated methods for identifying cerebrovascular accident or transient ischemic attack using administrative data. Pharmacoepidemiology and Drug Safety 2012;21 Suppl 1:100- 28.] → Tirischwell DL, Longstreth WT, Jr. Validating administrative data in stroke research. Stroke; a journal of cerebral circulation 2002;33:2465-70.] → Roumie CL, Mitchel E, Gideon PS, Varas-Lorenzo C, Castellsague J, Griffin MR. Validation of ICO-9 codes with a high positive predictive value for incident strokes resulting in hospitalization using Medicaid health data. Pharmacoepidemiology and drug safety 2008;17:20-6.] | Poor mapping or cannot be measured in claims Can't be measured in claims but not important for the analysis |
| | INCLUSION CRITERIA | <u>I</u> | | |
| 2 | Men or women aged ≥18 years Non-valvular Atrial fibrillation Atrial fibrillation must be documented by ECG evidence (e.g., 12-lead ECG, rhythm strip, Holter, pacemaker interrogation) within 30 days before randomization. In addition, subjects must have medical evidence of atrial fibrillation within 1 year before and at least one day before the qualifying ECG evidence. This could be obtained from a notation in the subject's record (e.g., medical chart, hospital discharge summary). | Measured on the day of drug initiation: Age >= 18 Measured 12 months prior to and including day of drug initiation, with >2 diagnoses separated by at least 14 days, in any diagnosis position and inpatient or outpatient care setting: Atrial fibrillation: ICD-9 diagnosis: 427.31 ICD-10 diagnosis: 48.0x, I48.1x, I48.2x, I48.9x | | |
| 3 | Non-valvular Atrial fibrillation Subjects with newly diagnosed atrial fibrillation are eligible provided that: - there is evidence that the atrial fibrillation is non-valvular - cardioversion is not planned - there is ECG evidence on 2 occasions 24 hours apart demonstrating atrial fibrillation For Inclusion Criteria 4 It is either A) History of ischemic stroke or TIA or arterial embolism OR- B) 2 of the following 4 1) Heart failure 2) Hypertension 3) Age >= 75 | | | |
| 4 | A) Diabetes History of prior ischemic stroke, TIA or non-CNS systemic embolism believed to be cardioembolic in origin | Measured any time prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Ischemic stroke: ICD-9 diagnosis: 433.x, 434.x, 436.xx IIA: ICD-9 diagnosis: 435.xx Systemic embolism: ICD-9 diagnosis: 444.xx | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 | |
| | OR 2 or more of the following risk factors | | | |
| 4a | - Heart failure and/or left ventricular ejection fraction ≤35% | Measured anytime prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Heart failure: ICD-9 diagnosis: 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagaliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 | |

| Measured 10 May prior to and inlocating day of drug initiation in any diagnosis position and impatient or outpatient care setting: Hopertension (defined as use of antihypertensive medications within 6 months before the screening visit or pensistent systolic blood pressure above 140 mmHg or diastolic blood pressure above 140 | ion based cohort study." BMU of Heart Failure Hospitalization pagliflozin Comparative on. 2019 Apr 8. doi: ssociated with canagliflozin ion based cohort study." BMU of Heart Failure Hospitalization pagliflozin Comparative |
|---|---|
| Age 275 years Measured any time prior to and including day of drug initiation in diagnosis position and inpatient or outpatient care setting: Methy top 2; ICD-9 diagnosis: 250.x0 or 250.x2 ICD-10 diagnosis: 250.x0 or 250.x2 ICD-10 diagnosis: E11.x Diabetes mellitus (defined as a history of type 1 or type 2 diabetes mellitus or use of antidiabetic drugs: populatic 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Add medications within 6 months before screening visit) Patorno, Elisabetta et al. "Cardiovascular outcomes as versus other non-piliflozin antidiabetic drugs: populatic 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk in Routine Clinical Care: A First Analysis from the Emp Effectiveness and Safety (EMPRISE) Study." Groulatic 10.1161/CIRCULATIONAHA.118.039177 Following drug dispensing within 6 months of drug initiation: Refer to the 'Diabetes meds' sheet for list of DM Drugs Female subjects must be postmenopausal (for at least 2 years), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study, and, for those of childbearing potential, have a negative serum β-hCG pregnancy test at screening. Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures | ion based cohort study." BMJ of Heart Failure Hospitalization pagliflozin Comparative |
| Inpatient or outpatient care setting: M type 2: ICD-9 diagnosis: 250:x0 or 250:x2 ICD-10 diagnosis: E11:x DM type 1: ICD-9 diagnosis: 250:x0 or 250:x3 ICD-10 diagnosis: 250:x0 or 250:x3 ICD-10 diagnosis: 250:x0 or 250:x3 ICD-10 diagnosis: 250:x1 or 250:x3 ICD-10 diagnosis: 250:x1 or 250:x3 ICD-10 diagnosis: 250:x1 or 250:x3 ICD-10 diagnosis: E10:x ICD-9 diagnosis: 250:x1 or 250:x3 ICD-10 diagnosis: E10:x ICD-1 | ion based cohort study." BMJ of Heart Failure Hospitalization pagliflozin Comparative |
| 5 an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study; and, for those of childbearing potential, have a negative serum β-hCG pregnancy test at screening. 6 Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures | · |
| | ien below. |
| required for the study and are willing to participate in the study | |
| In order to participate in the optional pharmacogenomic component, subjects must have signed the informed consent for DNA 7 research document indicating willingness to participate in the pharmacogenomics component of the study (where local regulations permit) | |
| EXCLUSION CRITERIA 1 Cardiac-Related Conditions | |
| Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Mitral stenosis: ICD-9 diagnosis: 396.0x, 396.1x ICD-10 diagnosis: 134.2x, 105.1x, 105.2x | |
| Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: ICD-9 diagnosis: V43.3x ICD-10 diagnosis: 295.2x CPT procedure: (TAVR with prosthetic valve) 33361, 33362, 33363, 33364, 33365, 33368, 33369, 33477, 0483T, 0684T, 0569T, 0570T | |
| 1c Planned cardioversion (electrical or pharmacological) N/A Will not capture 'planned' procedures | |
| 1c Planned cardioversion (electrical or pharmacological) N/A Will not capture 'planned' procedures Transient AF would not be well captured in claims. | |
| | r the hospitalist." Hospital |

| 2 | Active endocarditis Hemorrhage Risk-Related Criteria Active internal bleeding | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Endocarditis: ICD-9 diagnosis: 421.xx , 424.9x ICD-10 diagnosis: 133.xx, 138.xx, 139.xx Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Refer to the 'Bleeding' sheet for detailed codes (includes GI bleeding, intracranial, intra-articular bleeding mentioned in exclusion 2b) Measured 30 days prior to and including day of drug initiation in diagnosis position and inpatient or outpatient care setting: 11 Major surgery: Major surgery selected from procedure codes range 40.x-84.x -OR- | Tan, Charlie et al. "Accuracy of administrative data for identification of patients with infective endocarditis." International Journal of cardiology vol. 224 (2016): 162-164. doi:10.1016/j.ijcard.2016.09.030 |
|---|---|---|---|
| 2b | History of or condition associated with increased bleeding risk including, but not limited to: - Major surgical procedure or trauma within 30 days before the randomization visit - Clinically significant gastrointestinal bleeding within 6 months before the randomization visit - History of intracranial, intraccular, spinal, or atraumatic intra-articular bleeding - Chronic hemorrhagic disorder - Known intracranial neoplasm, arteriovenous malformation, or aneurysm | 21 Hemorrhagic disorder (Bleeding diathesis) 286.x Coagulation defects 287.x Purpura and other hemorrhagic conditions -OR- 31 Intracranial neoplasm, AV malformation, aneurysm Intracranial neoplasm ICD-9 diagnosis: 225.xx ICD-10 diagnosis: D33.xx AV malformation ICD-9 diagnosis: 747.81 ICD-10 diagnosis: 747.81 ICD-10 diagnosis: 47.3x ICD-10 diagnosis: 47.3x ICD-10 diagnosis: 47.3x ICD-10 diagnosis: 47.3x ICD-10 diagnosis: 47.3x | |
| 2c | Planned invasive procedure with potential for uncontrolled bleeding, including major surgery | N/A | |
| 2d | Platelet count < <90,000/μL at the screening visit | Measured 30 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Thrombocytopenia: ICD-9 diagnosis: 287.3x, 287.4x, 287.5x Measured 180 days prior to and including day of drug initiation in any diagnosis position | |
| | Sustained uncontrolled hypertension: systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥100 mmHg | and Inpatient care or ED setting: Malignant hypertension: ICD-9 diagnosis: 401.0x Hypertensive urgency/Hypertensive crisis: ICD-10 diagnosis: 116.xx | |
| 3 | Concomitant Conditions and Therapies | | |
| 3а | Severe, disabling stroke (modified Rankin score of 4 to 5, inclusive) within 3 months or any stroke within<br>14 days before the randomization visit | 1) Measured 30 days prior to and including day of drug initiation in position and care setting specified below: Stroke(primary diagnosis position, inpatient care setting): ICD-9 diagnosis: 430.xx, 431.xx, 433.xx, 434.xx, 436.xx, -PLUS- Disabling stroke effects (any position, any care setting, with 7-83 days between the strokes) ICD-9 diagnosis: 438.xx Late effects of cerebrovascular disease ICD-10 diagnosis: IGD-10 diagnosis: IGD-10 care to the stroke of the strokes of the strok | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| 3b | Transient ischemic attack within 3 days before the randomization visit | Measured 3 days prior to and including day of drug initiation in primary diagnosis position and inpatient care or ED setting: TIA: ICD-9 diagnosis: 435.xx | |

| 30 | Indication for anticoagulant therapy for a condition other than atrial fibrillation (e.g., VTE) | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: 1) Pulmonary embolism (PE): ICD-9 diagnosis: 415.vx (LCD-10 diagnosis: 126.vx, 2) Deep vein thrombosis (DVT): ICD-9 diagnosis: 451.vx, 453.vx ICD-10 diagnosis: 126.vx, 180.vx, 181.vx, 182.vx, 126.vx | |
|---|---|---|---|
| 30 | Treatment with: — Aspirin >100 mg daily — Aspirin in combination with thienopyridines within S days before randomization — Intravenous antiplatelets within S days before randomization — Fibrinolytics within 10 days before randomization — Note: Aspirin ≤100 mg monotherapy is allowed and thienopyridine monotherapy is allowed. | Measured 180 days prior to and including day of drug initiation: <u>Aspirin dose &gt;100mg</u> : (Only prescription use is captured.) Measured 10 days prior to and including day of drug initiation: <u>Fibrinolytic agents</u> : Alteplase, reteplase, tenecteplase, streptokinase, urokinase Measured 5 days prior to and including day of drug initiation: <u>Aspirin (any dose) + thienopyridines</u> (clopidogrel or prasugrel or ticlopidine) Measured 5 days prior to and including day of drug initiation: <u>Cangrelor</u> | |
| 36 | Anticipated need for chronic treatment with a non-steroidal anti-inflammatory drug | | |
| 31 | Systemic treatment with a strong inhibitor of cytochrome P450 3A4, such as ketoconazole or protease inhibitors, within 4 days before randomization, or planned treatment during the time period of the study | Measured 4 days prior to and including day of drug initiation as a dispensing of the following: <u>CYP inhibitors</u> (selected): | |
| 3g | Treatment with a strong inducer of cytochrome P450 3A4, such as rifampin/rifampicin, within 4 days before randomization, or planned treatment during the time period of the study | ketoconazole, metronidazole, amiodarone, cimetidine, omeprazole, fluoxetine, indinavir, ritonavir <u>CYP inducers</u> (selected): carbamazepine, phenytoin, rifampin/rifampicin, phenobarbital | |
| 31 | Anemia (hemoglobin <10 g/dL) at the screening visit | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Anemia (non-deficiency)/neoplastic/chemotherapy/hemorrhagic assoicated): ICD-9 diagnosis: 282.x, 283.x, 284.x, 285.0, 285.2 (acute posthemorrhagic anemia), 285.22 (anemia of neoplastic disease), 285.3 (antineoplastic chemotherapy induced anemia) ICD-10 diagnosis: D55 - D62, D63.0 | |
| 3 | Pregnancy or breast-feeding | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Refer to the 'Pregnancy' sheet. | |
| 3, | Any other contraindication to warfarin | N/A | |
| 34 | Known HIV infection at time of screening | Following diagnosis or drugs measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: HIV Infection: 024 Human immunodeficiency virus [HIV] disease 079.53 Human immunodeficiency virus, type 2 [HIV-2] V08 Asymptomatic human immunodeficiency virus [HIV] infection status -OR- Filled prescription for HIV treatment 180 days prior to drug initiation: Refer to the 'HIV treatment' sheet for list of treatments | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |

| 31 | Calculated CLCR <30 mL/min at the screening visit (refer to Attachment 4 for calculating CLCR) | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: CKD stage 4/5/ESRD; ICD-9 diagnosis: 585.4x, 585.5x, 585.6x ICD-10 diagnosis: N18.4x, N18.5x, N18.6x -OR- Dialysis/ Renal transplant; Refer to the 'Dialysis' sheet for list of codes | |
|---|---|---|---|
| 3m | Known significant liver disease (e.g., acute clinical hepatitis, chronic active hepatitis, cirrhosis), or ALT >3x the ULN | Measured 180 days prior to and including day of drug initiation in any diagnosis/procedure position and inpatient or outpatient care setting: Liver disease: ICD-9 diagnosis: 070.xx, 570.xx-573.xx 456.0x-456.2x, 576.8x, 782.4x, 789.5x ICD-9 procedure: 39.1x, 42.91 | |
| 4 | Study Participation and Follow-up-Related Criteria | | |
| $\Box$ | and a region of the second sec | Measured 180 days prior to and including day of drug initiation: | |
| 4a | Serious concomitant illness associated with a life expectancy of less than 2 years | CCI>=10 | |
| 4b | Drug addiction or alcohol abuse within 3 years before the randomization visit | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Alcohol abuse or dependence: 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence: 292.xx, 304.xx, 305.2x-305.9x, 648.3x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Groulation. 2019 Apr 8. doi: 10.1161/CRCUATIONAHALISA.039177 |
| 4c | Have received an experimental drug or used an experimental medical device within 30 days before the | N/A | |
| 24 | planned start of treatment Previous randomization in the present study or other study of rivaroxaban | N/A | |
| | Previous randomization in the present study of other study of notine study of nutro procession of the following th | N/A | |
| 4f | Inability or unwillingness to comply with study-related procedures | Measured 180 days hospitalization prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Non-compliance: ICD-9 diagnosis: V15.81 PERSONAL HISTORY OF NONCOMPLIANCE WITH MEDICAL TREATMENT PRESENTING HAZARDS TO HEALTH; V45.12 NONCOMPLIANCE WITH RENAL DIALYSIS | |
| | Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator. | N/A | |

| Trial ID | pNDA27 |
|---|---|
| Trial Name (with web links) | ROCKET AF |
| Trial Name (with pdf links) | ROCKET AF |
| NCT | NCT00403767 |
| Trial category | Primary indication |
| Therapeutic Area | Cardiology/Vascular Diseases |
| Study batch | NOACs |
| RCT Category | 4a- Unintended S with label change |
| <b>Brand Name</b> | <u>Xarelto</u> |
| <b>Generic Name</b> | rivaroxaban |
| <u>Sponsor</u> | Janssen Pharmaceuticals |
| <u>Year</u> | 2011 |
| Measurable endpoint | Primary endpoint of stroke and systemic embolism |
| <u>Exposure</u> | Rivaroxaban |
| <u>Comparator</u> | Warfarin |
| | patients with nonvalvular atrial fibrillation who were at increased risk |
| <u>Population</u> | for stroke |
| <u>Trial finding</u> | HR = 0.79 (95% CI 0.66–0.96) |
| No. of Patients | 14,264 |
| Non-inferiority margin | HR = 1.46 |
| | 0.95 power of 95% to calculate a noninferiority margin of 1.46 with a |
| <u>Power</u> | one-sided alpha level of 0.025. |
| Blinding | Double-blinded |
| | Alternative hypothesis of non-inferiority (NI) by a NI margin of 1.46 in hazard ratio (HR) based on on-treatment data from the per protocol population. The required number of primary efficacy endpoint events was determined based on the following assumptions: NI margin of 1.46, 1-sided alpha of 0.025, power of >95% when true HR is 1, and exponential distributions. The margin was selected based on clinical appropriateness and quantitative analysis of relevant studies in Hart et |
| Statistical Method | al. |
| | For the reduction in the risk of stroke and systemic embolism |
| Approval indication | resulting from atrial fibrillation |

#### **Dialysis codes**

ESRD, defined as 2 codes (either inpatient or outpatient), separated by at least 30 days

Codes include:

- ICD9 prox codes:

39.95, Hemodialysis

54.98, Peritoneal dialysis

- ICD9 dx codes:

585.5x, Chronic kidney disease, Stage V (for ESRD with no mention of dialysis)

585.6x, End stage renal disease (for ESRD with dialysis)

V56.0x, encounter for dialysis NOS

V56.8x, encounter for peritoneal dialysis

V45.1x, renal dialysis status

- CPT4 codes:

90957, 90960, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 4 or more face-to-face physician visits per month

90958, 90961, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 2-3 face-to-face physician visits per month

90959, 90962, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 1 face-to-face physician visit per month

90920, 90921, ESRD related services per full month; for patients 12-19 and twenty years of age and over

90924, 90925, ESRD related services (less than full month), per day; for patients 12-19 and twenty years of age and over

90935, Hemodialysis procedure with single physician evaluation

90937, Hemodialysis procedure requiring repeated evaluation(s) with or without substantial revision of dialysis prescription

90945, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies), with single physician evaluation

90947, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies) requiring repeated physician evaluations, with or without substantial revision of dialysis prescription

90965, 90966, ESRD related services for home dialysis per full month, for patients 12-19 and 20 years of age and older

90969, 90970, ESRD related services for dialysis less than a full month of service, per day; for patients 12-19 and 20 years of age and older

90989, Dialysis training, patient, including helper where applicable, any mode, completed course

90993, Dialysis training, patient, including helper where applicable, any mode, course not completed, per training session

90999, Unlisted dialysis procedure, inpatient or outpatient

99512, Home visit for hemodialysis

- HCPCS codes:

G0257, Unscheduled or emergency dialysis treatment for ESRD patient in a hospital outpatient dept. that is not certified as an ESRD facility G0314, G0317, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age an over to include monitoring for the adequacy of nutrition, etc. w/4 or more physician visit per month

G0315, G0318, ESRD related services during the course of treatment, for patients 12-19 and 20yrs of age and over to include monitoring for the adequacy of putrition, etc. w/2 or 3 physician visit per month

aucquacy of fluctition, etc. w/2 of 3 physician visit per month

G0316, G0319, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/1 physician visit per month

G0322, G0323, ESRD related services for home dialysis patients per full month: for patients 12-19 and 20 yrs of age and over to include monitoring for adequacy of nutrition and etc.

G0326, G0327, ESRD related services for home dialysis (less than full month), per day; for patients 12-19 and 20 yrs of age and over S9335, Home therapy, hemodialysis; administrative services, professional pharmacy services, care coordination, and all necessary supplies and equipment (drugs and nursing services coded separately), per diem

S9339, Home therapy, peritoneal dialysis, administrative services, care coordination and all necessary supplies and equipment, per diem

OR

Kidney transplant, defined as either 1 inpatient or 1 outpatient code

Codes include:

-ICD9 dx codes:

V42.0x, Kidney transplant status

996.81 Complications of transplanted kidney

-ICD9 prox codes:

55.6x, Transplant of kidney (Exclude 55.61)

- CPT4 codes:

50360, Renal allotransplantation, implantation, graft, w/o donor & recipient nephrectomy

# **Bleeding Codes** 423.0 - (ICD9) HEMOPERICARDIUM 430 - (ICD9) SUBARACHNOID HEMORRHAGE 431 - (ICD9) INTRACEREBRAL HEMORRHAGE 432.0 - (ICD9) NONTRAUMATIC EXTRADURAL HEMORRHAGE 432.1 - (ICD9) SUBDURAL HEMORRHAGE 432.9 - (ICD9) UNSPECIFIED INTRACRANIAL HEMORRHAGE 459.0 - (ICD9) HEMORRHAGE UNSPECIFIED 531.0 - (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE 531.00 - (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 531.01 - (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION 531.2 - (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION 531.20 - (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.21 - (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 531.4 - (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE 531.40 - (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 531.41 - (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION 531.6 - (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION 531.60 - (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.61 - (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 532.0 - (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE 532.00 - (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 532.01 - (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.2 - (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION 532.20 - (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 532.21 - (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 532.4 - (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE 532.40 - (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 532.41 - (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.6 - (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION 532.60 - (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 532.61 - (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.0 - (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE 533.00 - (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.01 - (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.2 - (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.20 - (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 533.21 - (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.4 - (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE 533.40 - (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION

533.41 - (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.6 - (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.60 - (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 533.61 - (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 534.0 - (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.00 - (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.01 - (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 534.2 - (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.20 - (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 534.21 - (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 534.4 - (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.40 - (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.41 - (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 534.6 - (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.60 - (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 534.61 - (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 562.02 - (ICD9) DIVERTICULOSIS OF SMALL INTESTINE WITH HEMORRHAGE 562.03 - (ICD9) DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.12 - (ICD9) DIVERTICULOSIS OF COLON WITH HEMORRHAGE 562.13 - (ICD9) DIVERTICULITIS OF COLON WITH HEMORRHAGE 568.81 - (ICD9) HEMOPERITONEUM (NONTRAUMATIC) 569.3 - (ICD9) HEMORRHAGE OF RECTUM AND ANUS 569.83 - (ICD9) PERFORATION OF INTESTINE 569.85 - (ICD9) ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 569.86 - (ICD9) DIEULAFOY LESION (HEMORRHAGIC) OF INTESTINE 578.0 - (ICD9) HEMATEMESIS 578.1 - (ICD9) BLOOD IN STOOL 578.9 - (ICD9) HEMORRHAGE OF GASTROINTESTINAL TRACT UNSPECIFIED 719.1 - (ICD9) HEMARTHROSIS 719.10 - (ICD9) HEMARTHROSIS SITE UNSPECIFIED 719.11 - (ICD9) HERARTHROSIS INVOLVING SHOULDER REGION 719.12 - (ICD9) HEMARTHORSIS INVOLVING UPPER ARM 719.13 - (ICD9) HEMARTHROSIS INVOLVING FOREARM 719.14 - (ICD9) HEMARTHROSIS INVOLVING HAND 719.15 - (ICD9) HEMARTHROSIS INVOLVING PELVIC REGION AND THIGH 719.16 - (ICD9) HEMARTHROSIS INVOLVING LOWER LEG 719.17 - (ICD9) HEMARTHROSIS INVOLVING ANKLE AND FOOT

1/19.18 - (ICD9) HEMARTHROSIS INVOLVING OTHER SPECIFIED SITES 719.19 - (ICD9) HEMARTHROSIS INVOLVING MULTIPLE SITES 131.2 - (ICD10) Hemopericardium, not elsewhere classified 160.00 - (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified carotid siphon and bifurcation 160.01 - (ICD10) Nontraumatic subarachnoid hemorrhage from right carotid siphon and bifurcation 160.02 - (ICD10) Nontraumatic subarachnoid hemorrhage from left carotid siphon and bifurcation 160.10 - (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified middle cerebral artery 160.11 - (ICD10) Nontraumatic subarachnoid hemorrhage from right middle cerebral artery I60.12 - (ICD10) Nontraumatic subarachnoid hemorrhage from left middle cerebral artery 160.2 - (ICD10) Nontraumatic subarachnoid hemorrhage from anterior communicating artery 160.30 - (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified posterior communicating artery 160.31 - (ICD10) Nontraumatic subarachnoid hemorrhage from right posterior communicating artery 160.32 - (ICD10) Nontraumatic subarachnoid hemorrhage from left posterior communicating artery I60.4 - (ICD10) Nontraumatic subarachnoid hemorrhage from basilar artery I60.50 - (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified vertebral artery I60.51 - (ICD10) Nontraumatic subarachnoid hemorrhage from right vertebral artery 160.52 - (ICD10) Nontraumatic subarachnoid hemorrhage from left vertebral artery 160.6 - (ICD10) Nontraumatic subarachnoid hemorrhage from other intracranial arteries 160.7 - (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified intracranial artery 160.8 - (ICD10) Other nontraumatic subarachnoid hemorrhage 160.9 - (ICD10) Nontraumatic subarachnoid hemorrhage, unspecified 161.0 - (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, subcortical I61.1 - (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, cortical 161.2 - (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, unspecified 161.3 - (ICD10) Nontraumatic intracerebral hemorrhage in brain stem 161.4 - (ICD10) Nontraumatic intracerebral hemorrhage in cerebellum I61.5 - (ICD10) Nontraumatic intracerebral hemorrhage, intraventricular 161.6 - (ICD10) Nontraumatic intracerebral hemorrhage, multiple localized 161.8 - (ICD10) Other nontraumatic intracerebral hemorrhage 161.9 - (ICD10) Nontraumatic intracerebral hemorrhage, unspecified 162.00 - (ICD10) Nontraumatic subdural hemorrhage, unspecified 162.01 - (ICD10) Nontraumatic acute subdural hemorrhage 162.02 - (ICD10) Nontraumatic subacute subdural hemorrhage 162.03 - (ICD10) Nontraumatic chronic subdural hemorrhage I62.1 - (ICD10) Nontraumatic extradural hemorrhage 162.9 - (ICD10) Nontraumatic intracranial hemorrhage, unspecified K25.0 - (ICD10) Acute gastric ulcer with hemorrhage K25.2 - (ICD10) Acute gastric ulcer with both hemorrhage and perforation K25.4 - (ICD10) Chronic or unspecified gastric ulcer with hemorrhage

| K25.6 - (ICD10) Chronic or unspecified gastric ulcer with both hemorrhage and perforation |
|---|
| K26.0 - (ICD10) Acute duodenal ulcer with hemorrhage |
| K26.2 - (ICD10) Acute duodenal ulcer with both hemorrhage and perforation |
| K26.4 - (ICD10) Chronic or unspecified duodenal ulcer with hemorrhage |
| K26.6 - (ICD10) Chronic or unspecified duodenal ulcer with both hemorrhage and perforation |
| K27.0 - (ICD10) Acute peptic ulcer, site unspecified, with hemorrhage |
| K27.2 - (ICD10) Acute peptic ulcer, site unspecified, with both hemorrhage and perforation |
| K27.4 - (ICD10) Chronic or unspecified peptic ulcer, site unspecified, with hemorrhage |
| K27.6 - (ICD10) Chronic or unspecified peptic ulcer, site unspecified, with both hemorrhage and perforation |
| K28.0 - (ICD10) Acute gastrojejunal ulcer with hemorrhage |
| K28.2 - (ICD10) Acute gastrojejunal ulcer with both hemorrhage and perforation |
| K28.4 - (ICD10) Chronic or unspecified gastrojejunal ulcer with hemorrhage |
| K28.6 - (ICD10) Chronic or unspecified gastrojejunal ulcer with both hemorrhage and perforation |
| K55.21 - (ICD10) Angiodysplasia of colon with hemorrhage |
| K56.60 - (ICD10) Unspecified intestinal obstruction |
| K57.01 - (ICD10) Diverticulitis of small intestine with perforation and abscess with bleeding |
| K57.11 - (ICD10) Diverticulosis of small intestine without perforation or abscess with bleeding |
| K57.13 - (ICD10) Diverticulitis of small intestine without perforation or abscess with bleeding |
| K57.21 - (ICD10) Diverticulitis of large intestine with perforation and abscess with bleeding |
| K57.31 - (ICD10) Diverticulosis of large intestine without perforation or abscess with bleeding |
| K57.33 - (ICD10) Diverticulitis of large intestine without perforation or abscess with bleeding |
| K57.41 - (ICD10) Diverticulitis of both small and large intestine with perforation and abscess with bleeding |
| K57.51 - (ICD10) Diverticulosis of both small and large intestine without perforation or abscess with bleeding |
| K57.53 - (ICD10) Diverticulitis of both small and large intestine without perforation or abscess with bleeding |
| K57.81 - (ICD10) Diverticulitis of intestine, part unspecified, with perforation and abscess with bleeding |
| K57.91 - (ICD10) Diverticulosis of intestine, part unspecified, without perforation or abscess with bleeding |
| K57.93 - (ICD10) Diverticulitis of intestine, part unspecified, without perforation or abscess with bleeding |
| K62.5 - (ICD10) Hemorrhage of anus and rectum |
| K63.1 - (ICD10) Perforation of intestine (nontraumatic) |

| K63.81 - (ICD10) Dieulatoy lesion of intestine |
|----------------------------------------------------------|
| K66.1 - (ICD10) Hemoperitoneum |
| K92.0 - (ICD10) Hematemesis |
| K92.1 - (ICD10) Melena |
| K92.2 - (ICD10) Gastrointestinal hemorrhage, unspecified |
| M25.00 - (ICD10) Hemarthrosis, unspecified joint |
| M25.011 - (ICD10) Hemarthrosis, right shoulder |
| M25.012 - (ICD10) Hemarthrosis, left shoulder |
| M25.019 - (ICD10) Hemarthrosis, unspecified shoulder |
| M25.021 - (ICD10) Hemarthrosis, right elbow |
| M25.022 - (ICD10) Hemarthrosis, left elbow |
| M25.029 - (ICD10) Hemarthrosis, unspecified elbow |
| M25.031 - (ICD10) Hemarthrosis, right wrist |
| M25.032 - (ICD10) Hemarthrosis, left wrist |
| M25.039 - (ICD10) Hemarthrosis, unspecified wrist |
| M25.041 - (ICD10) Hemarthrosis, right hand |
| M25.042 - (ICD10) Hemarthrosis, left hand |
| M25.049 - (ICD10) Hemarthrosis, unspecified hand |
| M25.051 - (ICD10) Hemarthrosis, right hip |
| M25.052 - (ICD10) Hemarthrosis, left hip |
| M25.059 - (ICD10) Hemarthrosis. unspecified hip |

M25.061 - (ICD10) Hemarthrosis, right knee
M25.062 - (ICD10) Hemarthrosis, left knee
M25.069 - (ICD10) Hemarthrosis, unspecified knee
M25.071 - (ICD10) Hemarthrosis, right ankle
M25.072 - (ICD10) Hemarthrosis, left ankle
M25.073 - (ICD10) Hemarthrosis, unspecified ankle
M25.073 - (ICD10) Hemarthrosis, inspecified ankle
M25.074 - (ICD10) Hemarthrosis, right foot
M25.075 - (ICD10) Hemarthrosis, unspecified foot
M25.076 - (ICD10) Hemarthrosis, unspecified foot
M25.08 - (ICD10) Hemarthrosis, other specified site
R58 - (ICD10) Hemorrhage, not elsewhere classified

Legacy Attribute - Procedure Code (Any Confinement Position):
0W.3P8ZZ - (ICD10) 0W3P8ZZ, Control Bleeding in Gastrointestinal Tract, Via Natural or Artificial Opening Endoscopic
44.43 - (ICD9) ENDOSCOPIC CONTROL OF GASTRIC OR DUODENAL BLEEDING

# **HIV Treatment**

Abacavir

Amprenavir

Atazanavir

Darunavir

Delavirdine

Didanosine

Efavirenz

Emtricitabine

Enfuvirtide

Etravirine

Fosamprenavir

Indinavir

Lamivudine-Zidovudine

Maraviroc

Nelfinavir

Nevirapine

Raltegravir

Rilpivirine

Ritonavir

Ritonavir-Lopinavir

Saquinavir

Stavudine

Tipranavir

Zalcitabine

Zidovudine

#### **Diabetes Medications**

ALOGLIPTIN BENZOATE/PIOGLITAZONE HCL

DAPAGLIFLOZIN PROPANEDIOL

DAPAGLIFLOZIN PROPANEDIOL/SAXAGLIPTIN HCL

ERTUGLIFLOZIN PIDOLATE

**EXENATIDE MICROSPHERES** 

INSULIN ASPART PROTAMINE HUMAN/INSULIN ASPART

**INSULIN DETEMIR** 

INSULIN GLARGINE, HUMAN RECOMBINANT ANALOG/LIXISENATIDE

INSULIN NPH HUMAN AND INSULIN REGULAR HUMAN SEMI-SYNTHETIC

INSULIN ZINC HUMAN RECOMBINANT

LIXISENATIDE

PIOGLITAZONE HCL/GLIMEPIRIDE

REPAGLINIDE/METFORMIN HCL

ALOGLIPTIN BENZOATE

CANAGLIFLOZIN

CANAGLIFLOZIN/METFORMIN HCL

DULAGLUTIDE

INSULIN DEGLUDEC

INSULIN, PORK PURIFIED

LINAGLIPTIN

ROSIGLITAZONE MALEATE/GLIMEPIRIDE

SAXAGLIPTIN HCL/METFORMIN HCL

**ALBIGLUTIDE** 

DAPAGLIFLOZIN PROPANEDIOL/METFORMIN HCL

ERTUGLIFLOZIN PIDOLATE/METFORMIN HCL

**EXENATIDE** 

INSULIN ASPART

MIGLITOL

PRAMLINTIDE ACETATE

SEMAGLUTIDE

**EMPAGLIFLOZIN** 

INSULIN LISPRO PROTAMINE AND INSULIN LISPRO

INSULIN ZINC EXTENDED HUMAN RECOMBINANT

SAXAGLIPTIN HCL

EMPAGLIFLOZIN/LINAGLIPTIN

ERTUGLIFLOZIN PIDOLATE/SITAGLIPTIN PHOSPHATE

INSULIN DEGLUDEC/LIRAGLUTIDE

LIRAGLUTIDE

ALOGLIPTIN BENZOATE/METFORMIN HCL

INSULIN LISPRO

EMPAGLIFLOZIN/METFORMIN HCL

LINAGLIPTIN/METFORMIN HCL

INSULIN GLARGINE, HUMAN RECOMBINANT ANALOG

NATEGLINIDE

SITAGLIPTIN PHOSPHATE

INSULIN GLULISINE

ROSIGLITAZONE MALEATE/METFORMIN HCL

SITAGLIPTIN PHOSPHATE/METFORMIN HCL

INSULIN NPH HUMAN ISOPHANE/INSULIN REGULAR, HUMAN

INSULIN REGULAR, HUMAN

GLIPIZIDE/METFORMIN HCL

PIOGLITAZONE HCL/METFORMIN HCL

REPAGLINIDE

ACETOHEXAMIDE

ROSIGLITAZONE MALEATE
ACARBOSE
GLYBURIDE,MICRONIZED
TOLBUTAMIDE
GLYBURIDE/METFORMIN HCL
GLIMEPIRIDE
PIOGLITAZONE HCL
TOLAZAMIDE

GLYBURIDE

GLIPIZIDE

METFORMIN HCL

CHLORPROPAMIDE
# Appendix A

| Нур | ertension medications |
|---|---|
| ACE inhibitor | Benazepril, captopril, enalapril, fosinopril, lisinopril, moexipril, perindopril, quinapril, ramipril, trandolapril |
| ARB | Azilsartan, candesartan, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan |
| Beta blocker | Acebutolol, atenolol, betaxolol, bisoprolol, carteolol, carvedilol, esmolol, labetalol, metoprolol tartrate, metoprolol succinate, propranolol, penbutolol, pindolol, nadolol, nebivolol, sotalol, timolol |
| Calcium channel blocker | Diltiazem, mibefradil, verapamil, amlodipine, clevidipine, bepridil, felodipine, isradipine, nicardipine, nifedipine, nimodipine, nisoldipine |
| Other hypertension drugs | Doxazosin, eplerenone, prazosin, terazosin, clonidine, guanabenz, guanadrel, guanethidine, guanfacine, hydralazine, methyldopa, metyrosine, reserpine, minoxidil, aliskiren |
| Thiazides | Benzthiazide, chlorothiazide, chlorthalidone, cyclothiazide, hydrochlorothiazide, hydroflumethiazide, indapamide, methyclothiazide, metolazone, polythiazide, quinethazone, trichlormethiazide, bendroflumethiazide |
| Loop diuretics | Furosemide, bumetanide, torsemide, ethacrynic acid |
| Other diuretics | Amiloride, eplerenone, spironolactone, triamterene |

72.3 HIGH FORCEPS OPERATION

# **Pregnancy** Diagnosis codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN+A2:J81 V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY Procedure codes 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION

#### Appendix A

- 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY
- 72.39 OTHER HIGH FORCEPS OPERATION
- 72.4 FORCEPS ROTATION OF FETAL HEAD
- 72.5 BREECH EXTRACTION
- 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.52 OTHER PARTIAL BREECH EXTRACTION
- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION

#### Appendix A

- 74.1 LOW CERVICAL CESAREAN SECTION
- 74.2 EXTRAPERITONEAL CESAREAN SECTION
- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS

Appendix B: Rivaroxaban vs Warfarin



| | | | | | Unmatched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Optu | | | MarketS | | | Medicare | | | | POOLED | |
| Variable | Reference-warfarin | Exposure - rivaroxaban<br>(15 or 20 mg) | St. Diff. | Reference-warfarin | Exposure - rivaroxaban<br>(15 or 20 mg) | St. Diff. | Reference- warfarin | Exposure - | St. Diff. | Reference-warfarin | Exposure - rivaroxaban<br>(15 or 20 mg) | St. Diff. |
| Number of patients | 25,701 | (15 of 20 flig)<br>14,869 | St. Dill. | 32,295 | (15 of 20 mg)<br>17,748 | St. Dill. | 92,403 | 40,652 | St. Dill. | 150,399 | 73,269 | St. Dill. |
| Age | 23,701 | 14,005 | | 32,233 | 17,740 | | 32,403 | 40,032 | | 130,333 | 73,203 | |
| mean (sd) | 76.81 (7.78) | 74.48 (9.36) | 0.27 | 76.99 (10.15) | 72.74 (11.18) | 0.40 | 79.76 (7.99) | 78.49 (8.07) | 0.16 | 78.66 (8.47) | 76.28 (9.18) | 0.27 |
| median [IQR] | 78.00 [73.00, 82.00] | 76.00 [69.00, 82.00] | 0.23 | 79.00 [72.00, 84.00] | 75.00 [64.00, 81.00] | 0.37 | 80.00 [76.00, 85.00] } | , , | 0.12 | 79.44 (8.47) | 77.42 (9.18) | 0.23 |
| Age categories without zero category | 70.00 [73.00, 02.00] | 70.00 [03.00, 02.00] | 0.25 | 75.00 [72.00,01.00] | 75.00 [01.00,02.00] | 0.57 | 00.00 (, 0.00, 05.00), | .00 [/ 1.00, 0 1.00] | 0.12 | 73.11(0.17) | 77.12 (3.20) | 0.23 |
| 18 - 54; n (%) | 395 (1.5%) | 556 (3.7%) | -0.14 | 906 (2.8%) | 1,010 (5.7%) | -0.14 | 738 (0.8%) | 423 (1.0%) | -0.02 | 2,039 (1.4%) | 1989 (2.7%) | -0.09 |
| 55 - 64; n (%) | 1,596 (6.2%) | 1,657 (11.1%) | -0.17 | 3,653 (11.3%) | 3,754 (21.2%) | -0.27 | 2,322 (2.5%) | 1,256 (3.1%) | -0.04 | 7,571 (5.0%) | 6,667 (9.1%) | -0.16 |
| 65 - 74; n (%) | 5,501 (21.4%) | 3,823 (25.7%) | -0.10 | 5,619 (17.4%) | 3,840 (21.6%) | -0.11 | 16,731 (18.1%) | 9,029 (22.2%) | -0.10 | 27,851 (18.5%) | 16,692 (22.8%) | -0.11 |
| >= 75; n (%) | 18,209 (70.8%) | 8,833 (59.4%) | 0.24 | 22,117 (68.5%) | 9,144 (51.5%) | 0.35 | 72,612 (78.6%) | 29,944 (73.7%) | 0.12 | 112,938 (75.1%) | 47,921 (65.4%) | 0.21 |
| Gender without zero category- United | | | | | | | | | | | | |
| Males; n (%) | 13,338 (51.9%) | 7,726 (52.0%) | 0.00 | 17,422 (53.9%) | 9,827 (55.4%) | -0.03 | 39,860 (43.1%) | 16,739 (41.2%) | 0.04 | 70,620 (47.0%) | 34,292 (46.8%) | 0.00 |
| Females; n (%) | 12,363 (48.1%) | 7,143 (48.0%) | 0.00 | 14,873 (46.1%) | 7,921 (44.6%) | 0.03 | 52,543 (56.9%) | 23,913 (58.8%) | -0.04 | 79,779 (53.0%) | 38,977 (53.2%) | 0.00 |
| Race | | | | | | | | | | | | |
| White; n (%) | | | | | | | 85,842 (92.9%) | 36,882 (90.7%) | | 85,842 (92.9%) | 36,882 (90.7%) | 0.00 |
| Black; n (%) | | | | | | | 3,514 (3.8%) | 1,923 (4.7%) | | 3,514 (3.8%) | 1,923 (4.7%) | 0.00 |
| Asian; n (%) | | | | | | | 767 (0.8%) | 513 (1.3%) | | 767 (0.8%) | 513 (1.3%) | 0.00 |
| Hispanic; n (%) | | | | | | | 998 (1.1%) | 596 (1.5%) | | 998 (1.1%) | 596 (1.5%) | 0.00 |
| North American Native; n (%) | | | | | | | 339 (0.4%) | 159 (0.4%) | | 339 (0.4%) | 159 (0.4%) | 0.00 |
| Other/Unknown; n (%) Region without zero category- United v3 (lumping | | | | | | | 943 (1.0%) | 579 (1.4%) | | 943 (1.0%) | 579 (1.4%) | 0.00 |
| missing&other category with West) | 3,626 (14.1%) | 2,178 (14.6%) | -0.01 | 7,778 (24.1%) | 4,155 (23.4%) | 0.02 | 21,665 (23.4%) | 8,259 (20.3%) | 0.08 | 33,069 (22.0%) | 14,592 (19.9%) | 0.05 |
| Northeast; n (%) | 3,626 (14.1%)<br>8,341 (32.5%) | 2,178 (14.6%)<br>6,178 (41.5%) | -0.01<br>-0.19 | 7,778 (24.1%)<br>10,408 (32.2%) | 4,155 (23.4%)<br>4,919 (27.7%) | 0.02 | 21,665 (23.4%) 28,585 (30.9%) | 8,259 (20.3%)<br>16,109 (39.6%) | -0.18 | 47,334 (31.5%) | 14,592 (19.9%)<br>27,206 (37.1%) | -0.12 |
| South; n (%) | 5,845 (22.7%) | 2,875 (19.3%) | 0.08 | 8,928 (27.6%) | 6,242 (35.2%) | -0.16 | 27,907 (30.2%) | 10,396 (25.6%) | 0.10 | 42,680 (28.4%) | 19,513 (26.6%) | 0.04 |
| Midwest; n (%)<br>West; n (%) | 7,889 (30.7%) | 3,638 (24.5%) | 0.08 | 5,055 (15.7%) | 2,317 (13.1%) | 0.16 | 14,246 (15.4%) | 5,888 (14.5%) | 0.10 | 27,190 (18.1%) | 11,843 (16.2%) | 0.04 |
| Unknown+missing; n (%) | 7,885 (30.7%)<br>N/A | 3,038 (24.5%)<br>N/A | #VALUE! | 126 (0.4%) | 115 (0.6%) | -0.03 | 14,240 (13.4%)<br>N/A | 0,888 (14.5%)<br>N/A | #VALUE! | 126 (0.4%) | 11,843 (10.2%) | -0.03 |
| CV Covariates | 19/5 | 14/15 | #VALUE: | 120 (0.470) | 113 (0.070) | 0.03 | 19/5 | 14/7 | #VALUE: | 120 (0.470) | 113 (0.070) | 0.03 |
| Ischemic heart disease; n (%) | 9,344 (36.4%) | 5,576 (37.5%) | -0.02 | 11,325 (35.1%) | 6.317 (35.6%) | -0.01 | 37.684 (40.8%) | 17.950 (44.2%) | -0.07 | 58.353 (38.8%) | 29.843 (40.7%) | -0.04 |
| Acute MI; n (%) | 682 (2.7%) | 450 (3.0%) | -0.02 | 729 (2.3%) | 476 (2.7%) | -0.03 | 2,949 (3.2%) | 1,572 (3.9%) | -0.04 | 4360 (2.9%) | 2498 (3.4%) | -0.03 |
| ACS/unstable angina; n (%) | 582 (2.3%) | 465 (3.1%) | -0.05 | 680 (2.1%) | 509 (2.9%) | -0.05 | 2,657 (2.9%) | 1,599 (3.9%) | -0.06 | 3919 (2.6%) | 2573 (3.5%) | -0.05 |
| Old MI; n (%) | 1,268 (4.9%) | 859 (5.8%) | -0.04 | 949 (2.9%) | 543 (3.1%) | -0.01 | 6,575 (7.1%) | 3,525 (8.7%) | -0.06 | 8792 (5.8%) | 4927 (6.7%) | -0.04 |
| Stable angina; n (%) | 1,103 (4.3%) | 862 (5.8%) | -0.07 | 1,016 (3.1%) | 756 (4.3%) | -0.06 | 3,424 (3.7%) | 2,051 (5.0%) | -0.06 | 5,543 (3.7%) | 3,669 (5.0%) | -0.06 |
| Coronary atherosclerosis and other forms of chronic | | | | | | | | | | | | |
| ischemic heart disease; n (%) | 8,620 (33.5%) | 5,100 (34.3%) | -0.02 | 10,565 (32.7%) | 5,774 (32.5%) | 0.00 | 35,060 (37.9%) | 16,501 (40.6%) | -0.06 | 54,245 (36.1%) | 27,375 (37.4%) | -0.03 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) | 459 (1.8%) | 229 (1.5%) | 0.02 | 612 (1.9%) | 282 (1.6%) | 0.02 | 1,748 (1.9%) | 698 (1.7%) | 0.02 | 2819 (1.9%) | 1209 (1.7%) | 0.02 |
| Previous cardiac procedure (CABG or PTCA or Stent) | | | | | | | | | | | | |
| v4; n (%) | 210 (0.8%) | 147 (1.0%) | -0.02 | 294 (0.9%) | 131 (0.7%) | 0.02 | 1,098 (1.2%) | 509 (1.3%) | -0.01 | 1602 (1.1%) | 787 (1.1%) | 0.00 |
| History of CABG or PTCA; n (%) | 2,059 (8.0%) | 1,491 (10.0%) | -0.07 | 1,375 (4.3%) | 879 (5.0%) | -0.03 | 12,032 (13.0%) | 6,338 (15.6%) | -0.07 | 15,466 (10.3%) | 8,708 (11.9%) | -0.05 |
| Any stroke; n (%) | 4,563 (17.8%) | 3,218 (21.6%) | -0.10 | 5,295 (16.4%) | 3,292 (18.5%) | -0.06 | 18,172 (19.7%) | 9,000 (22.1%) | -0.06 | 28,030 (18.6%) | 15,510 (21.2%) | -0.07 |
| Ischemic stroke (w and w/o mention of cerebral infarction); n (%) | 4,563 (17.8%) | 3,218 (21.6%) | -0.10 | 5,295 (16.4%) | 3,292 (18.5%) | -0.06 | 18,114 (19.6%) | 8,981 (22.1%) | -0.06 | 27,972 (18.6%) | 15,491 (21.1%) | -0.06 |
| Hemorrhagic stroke; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 226 (0.2%) | 97 (0.2%) | 0.00 | 27,972 (18.6%) | 97 (0.1%) | 0.03 |
| TIA; n (%) | 1,646 (6.4%) | 1,300 (8.7%) | -0.09 | 1,863 (5.8%) | 1,452 (8.2%) | -0.09 | 5,231 (5.7%) | 2,791 (6.9%) | -0.05 | 8740 (5.8%) | 5543 (7.6%) | -0.07 |
| Other cerebrovascular disease; n (%) | 887 (3.5%) | 674 (4.5%) | -0.05 | 944 (2.9%) | 581 (3.3%) | -0.03 | 4,120 (4.5%) | 2,059 (5.1%) | -0.03 | 5951 (4.0%) | 3314 (4.5%) | -0.07 |
| Late effects of cerebrovascular disease; n (%) | 992 (3.9%) | 563 (3.8%) | 0.01 | 948 (2.9%) | 445 (2.5%) | 0.02 | 5,242 (5.7%) | 2,344 (5.8%) | 0.00 | 7182 (4.8%) | 3352 (4.6%) | 0.01 |
| Cerebrovascular procedure; n (%) | 36 (0.1%) | 24 (0.2%) | -0.03 | 56 (0.2%) | 32 (0.2%) | 0.00 | 255 (0.3%) | 138 (0.3%) | 0.00 | 347 (0.2%) | 194 (0.3%) | -0.02 |
| Heart failure (CHF); n (%) | 6,985 (27.2%) | 3,669 (24.7%) | 0.06 | 8,000 (24.8%) | 3,790 (21.4%) | 0.08 | 33,361 (36.1%) | 15,107 (37.2%) | -0.02 | 48,346 (32.1%) | 22,566 (30.8%) | 0.03 |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2; | | | | | | | | | | | | |
| n (%) | 2,542 (9.9%) | 1,530 (10.3%) | -0.01 | 2,939 (9.1%) | 1,390 (7.8%) | 0.05 | 10,824 (11.7%) | 4,854 (11.9%) | -0.01 | 16,305 (10.8%) | 7,774 (10.6%) | 0.01 |
| Atrial fibrillation; n (%) | 24,905 (96.9%) | 14,554 (97.9%) | -0.06 | 30,559 (94.6%) | 17,422 (98.2%) | -0.19 | 89,565 (96.9%) | 39,491 (97.1%) | -0.01 | 145,029 (96.4%) | 71,467 (97.5%) | -0.06 |
| Other cardiac dysrhythmia; n (%) | 13,569 (52.8%) | 10,907 (73.4%) | -0.44 | 10,549 (32.7%) | 8,843 (49.8%) | -0.35 | 44,238 (47.9%) | 24,562 (60.4%) | -0.25 | 68,356 (45.4%) | 44,312 (60.5%) | -0.31 |
| Cardiac conduction disorders; n (%) | 2,156 (8.4%) | 1,560 (10.5%) | -0.07 | 2,075 (6.4%) | 1,362 (7.7%) | -0.05 | 8,105 (8.8%) | 4,354 (10.7%) | -0.06 | 12336 (8.2%) | 7276 (9.9%) | -0.06 |
| Other CVD; n (%) | 8,898 (34.6%) | 5,631 (37.9%) | -0.07 | 10,301 (31.9%) | 6,111 (34.4%) | -0.05 | 32,880 (35.6%) | 15,926 (39.2%) | -0.07 | 52,079 (34.6%) | 27,668 (37.8%) | -0.07 |
| Diabetes-related complications | | | | | | | | | | | | |
| Diabetic retinopathy; n (%) | 509 (2.0%) | 251 (1.7%) | 0.02 | 567 (1.8%) | 234 (1.3%) | 0.04 | 1,748 (1.9%) | 714 (1.8%) | 0.01 | 2,824 (1.9%) | 1,199 (1.6%) | 0.02 |
| Diabetes with other ophthalmic manifestations; n | | | | | | | | | | | | |
| (%) | 38 (0.1%) | 37 (0.2%) | -0.03 | 433 (1.3%) | 168 (0.9%) | 0.04 | 1,127 (1.2%) | 458 (1.1%) | 0.01 | 1598 (1.1%) | 663 (0.9%) | 0.02 |
| Retinal detachment, vitreous hemorrhage, | 40 (0.0-1) | 25 (0.20() | 2.25 | 04 (0.000) | 25 (0.200) | 0.00 | 475 (0.5-0) | 76 (0.20() | 2.22 | 201/02-11 | 4.5 (0.20) | 2.25 |
| vitrectomy; n (%) | 48 (0.2%) | 35 (0.2%) | 0.00 | 81 (0.3%) | 35 (0.2%) | 0.02<br>0.02 | 175 (0.2%) | 76 (0.2%) | 0.00<br>0.00 | 304 (0.2%) | 146 (0.2%) | 0.00 |
| Retinal laser coagulation therapy; n (%) | 33 (0.1%) | 14 (0.1%) | 0.00 | 84 (0.3%) | 27 (0.2%) | 0.02 | 179 (0.2%) | 76 (0.2%) | -0.01 | 296 (0.2%) | 117 (0.2%) | 0.00 |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 1,737 (6.8%) | 892 (6.0%) | 0.03 | 1,633 (5.1%) | 840 (4.7%) | 0.02 | 6,290 (6.8%) | 2,868 (7.1%) | -0.01 | 9660 (6.4%) | 4600 (6.3%) | 0.00 |

| Occurrence of diabetic nephropathy V3 with ICD10 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Copy; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1,264 (1.4%) | 565 (1.4%) | 0.00 | 1,264 (0.8%) | 565 (0.8%) | 0.00 |
| Hypoglycemia v2; n (%) | 267 (1.0%) | 118 (0.8%) | 0.02 | 460 (1.4%) | 194 (1.1%) | 0.03 | 2,229 (2.4%) | 1,198 (2.9%) | -0.03 | 2956 (2.0%) | 1510 (2.1%) | -0.01 |
| Hyperglycemia; n (%) | 1,205 (4.7%) | 912 (6.1%) | -0.06 | 701 (2.2%) | 569 (3.2%) | -0.06 | 4,983 (5.4%) | 2,695 (6.6%) | -0.05 | 6889 (4.6%) | 4176 (5.7%) | -0.05 |
| Disorders of fluid electrolyte and acid-base balance; n | 2 270 (0 20/) | 4 524 (40 00) | 2.25 | 2 276 /7 00/) | 4 400 (0 40() | 0.05 | 44 744 (42 70/) | 5 425 (42 50/) | 0.00 | 4.53.50 (4.0.00() | 0247/44 20/ | |
| (%) | 2,379 (9.3%) | 1,624 (10.9%) | -0.05<br>-0.03 | 2,276 (7.0%) | 1,498 (8.4%) | -0.05<br>0.00 | 11,714 (12.7%) | 5,125 (12.6%) | 0.00 | 16369 (10.9%) | 8247 (11.3%) | -0.01<br>0.00 |
| Diabetic ketoacidosis; n (%) Hyperosmolar hyperglycemic nonketotic syndrome | 28 (0.1%) | 24 (0.2%) | -0.03 | 35 (0.1%) | 24 (0.1%) | 0.00 | 168 (0.2%) | 81 (0.2%) | 0.00 | 231 (0.2%) | 129 (0.2%) | 0.00 |
| (HONK); n (%) | 26 (0.1%) | 23 (0.2%) | -0.03 | 25 (0.1%) | 19 (0.1%) | 0.00 | 147 (0.2%) | 86 (0.2%) | 0.00 | 198 (0.1%) | 128 (0.2%) | -0.03 |
| Diabetes with peripheral circulatory disorders with | 20 (0.270) | 25 (0.270) | 0.03 | 25 (0:270) | 13 (0.170) | 0.00 | 117 (0.270) | 00 (0.270) | 0.00 | 130 (0.170) | 120 (0.270) | 0.05 |
| ICD-10 v2 Copy; n (%) | 863 (3.4%) | 413 (2.8%) | 0.03 | 810 (2.5%) | 339 (1.9%) | 0.04 | 4,632 (5.0%) | 1,893 (4.7%) | 0.01 | 6305 (4.2%) | 2645 (3.6%) | 0.03 |
| Diabetic Foot; n (%) | 641 (2.5%) | 259 (1.7%) | 0.06 | 864 (2.7%) | 329 (1.9%) | 0.05 | 4,161 (4.5%) | 1,511 (3.7%) | 0.04 | 5666 (3.8%) | 2099 (2.9%) | 0.05 |
| Gangrene v2; n (%) | 32 (0.1%) | 25 (0.2%) | -0.03 | 53 (0.2%) | 14 (0.1%) | 0.03 | 251 (0.3%) | 80 (0.2%) | 0.02 | 336 (0.2%) | 119 (0.2%) | 0.00 |
| Lower extremity amputation; n (%) | 103 (0.4%) | 47 (0.3%) | 0.02 | 66 (0.2%) | 33 (0.2%) | 0.00 | 577 (0.6%) | 221 (0.5%) | 0.01 | 746 (0.5%) | 301 (0.4%) | 0.01 |
| Osteomyelitis; n (%) | 89 (0.3%) | 43 (0.3%) | 0.00 | 130 (0.4%) | 65 (0.4%) | 0.00 | 642 (0.7%) | 264 (0.6%) | 0.01 | 861 (0.6%) | 372 (0.5%) | 0.01 |
| Skin infections v2; n (%) | 1,508 (5.9%) | 777 (5.2%) | 0.03 | 2,170 (6.7%) | 1,006 (5.7%) | 0.04 | 7,041 (7.6%) | 2,925 (7.2%) | 0.02 | 10719 (7.1%) | 4708 (6.4%) | 0.03 |
| Erectile dysfunction; n (%) | 400 (1.6%) | 301 (2.0%) | -0.03 | 363 (1.1%) | 327 (1.8%) | -0.06 | 577 (0.6%) | 320 (0.8%) | -0.02 | 1340 (0.9%) | 948 (1.3%) | -0.04 |
| Diabetes with unspecified complication; n (%) | 345 (1.3%) | 282 (1.9%) | -0.05 | 355 (1.1%) | 254 (1.4%) | -0.03 | 1,374 (1.5%) | 754 (1.9%) | -0.03 | 2074 (1.4%) | 1290 (1.8%) | -0.03 |
| Diabetes mellitus without mention of complications; | | | | | | | | | | | | |
| n (%) | 9,288 (36.1%) | 5,120 (34.4%) | 0.04 | 10,733 (33.2%) | 6,006 (33.8%) | -0.01 | 40,275 (43.6%) | 18,008 (44.3%) | -0.01 | 60,296 (40.1%) | 29,134 (39.8%) | 0.01 |
| Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) | 21,744 (84.6%) | 12,927 (86.9%) | -0.07 | 23,292 (72.1%) | 14,059 (79.2%) | -0.17 | 85,616 (92.7%) | 38,411 (94.5%) | -0.07 | 130,652 (86.9%) | 65,397 (89.3%) | -0.07 |
| Hyperlipidemia v2; n (%) | 15,725 (61.2%) | 9,844 (66.2%) | -0.10 | 14,454 (44.8%) | 9,966 (56.2%) | -0.23 | 53,237 (57.6%) | 26,192 (64.4%) | -0.14 | 83,416 (55.5%) | 46,002 (62.8%) | -0.15 |
| Edema; n (%) | 2,694 (10.5%) | 1,703 (11.5%) | -0.03 | 2,678 (8.3%) | 1,441 (8.1%) | 0.01 | 10,081 (10.9%) | 4,546 (11.2%) | -0.01 | 15453 (10.3%) | 7690 (10.5%) | -0.01 |
| Renal Dysfunction (non-diabetic) v2; n (%) | 17 (0.1%) | 7 (0.0%) | 0.04 | 19 (0.1%) | 12 (0.1%) | 0.00 | 4,118 (4.5%) | 1,550 (3.8%) | 0.04 | 4,154 (2.8%) | 1,569 (2.1%) | 0.05 |
| Occurrence of acute renal disease v2; n (%) | 13 (0.1%) | 6 (0.0%) | 0.04 | 19 (0.1%) | 12 (0.1%) | 0.00 | 466 (0.5%) | 199 (0.5%) | 0.00 | 498 (0.3%) | 217 (0.3%) | 0.00 |
| Occurrence of chronic renal insufficiency; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 2,595 (2.8%) | 832 (2.0%) | 0.05 | 2,595 (1.7%) | 832 (1.1%) | 0.05 |
| Chronic kidney disease v2; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 2,451 (2.7%) | 775 (1.9%) | 0.05 | 2,451 (1.6%) | 775 (1.1%) | 0.04 |
| CKD Stage 3-4; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1,885 (2.0%) | 538 (1.3%) | 0.05 | 1,885 (1.3%) | 538 (0.7%) | 0.06 |
| Occurrence of hypertensive nephropathy; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 530 (0.6%) | 239 (0.6%) | 0.00 | #VALUE! | 239 (0.3%) | #VALUE! |
| Occurrence of miscellaneous renal insufficiency v2; n | | | | | | | | | | | | |
| (%) | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1,435 (1.6%) | 642 (1.6%) | 0.00 | 1,436 (1.0%) | 643 (0.9%) | 0.01 |
| Glaucoma or cataracts v2; n (%) | 5,562 (21.6%) | 3,146 (21.2%) | 0.01 | 7,173 (22.2%) | 3,770 (21.2%) | 0.02 | 1,558 (1.7%) | 741 (1.8%) | -0.01 | 14,293 (9.5%) | 7,657 (10.5%) | -0.03 |
| Cellulitis or abscess of toe; n (%) | 337 (1.3%) | 241 (1.6%) | -0.03 | 280 (0.9%) | 179 (1.0%) | -0.01 | 3,729 (4.0%) | 1,328 (3.3%) | 0.04 | 4346 (2.9%) | 1748 (2.4%) | 0.03 |
| Foot ulcer; n (%) | 650 (2.5%) | 262 (1.8%) | 0.05 | 891 (2.8%) | 336 (1.9%) | 0.06 | 78 (0.1%) | 47 (0.1%) | 0.00 | 1619 (1.1%) | 645 (0.9%) | 0.02 |
| Bladder stones; n (%)<br>Kidney stones; n (%) | 23 (0.1%)<br>197 (0.8%) | 12 (0.1%)<br>170 (1.1%) | 0.00<br>-0.03 | 28 (0.1%)<br>297 (0.9%) | 15 (0.1%)<br>201 (1.1%) | 0.00<br>-0.02 | 1,249 (1.4%)<br>14,547 (15.7%) | 656 (1.6%)<br>6,671 (16.4%) | -0.02<br>-0.02 | 1300 (0.9%)<br>15041 (10.0%) | 683 (0.9%)<br>7042 (9.6%) | 0.00<br>0.01 |
| Urinary tract infections (UTIs); n (%) | 2,316 (9.0%) | 1,299 (8.7%) | 0.01 | 2,410 (7.5%) | 1,240 (7.0%) | 0.02 | 33,456 (36.2%) | 16,172 (39.8%) | -0.02 | 38,182 (25.4%) | 18,711 (25.5%) | 0.00 |
| Dipstick urinalysis; n (%) | 6,881 (26.8%) | 4,590 (30.9%) | -0.09 | 6,443 (20.0%) | 4,127 (23.3%) | -0.08 | 14,331 (15.5%) | 6,373 (15.7%) | -0.01 | 27,655 (18.4%) | 15,090 (20.6%) | -0.06 |
| Non-dipstick urinalysis; n (%) | 3,469 (13.5%) | 2,020 (13.6%) | 0.00 | 1,948 (6.0%) | 1,256 (7.1%) | -0.04 | 3,642 (3.9%) | 1,643 (4.0%) | -0.01 | 9,059 (6.0%) | 4,919 (6.7%) | -0.03 |
| Urine function test; n (%) | 661 (2.6%) | 362 (2.4%) | 0.01 | 1,148 (3.6%) | 580 (3.3%) | 0.02 | 1,909 (2.1%) | 900 (2.2%) | -0.01 | 3718 (2.5%) | 1842 (2.5%) | 0.00 |
| Cytology; n (%) | 219 (0.9%) | 155 (1.0%) | -0.01 | 382 (1.2%) | 167 (0.9%) | 0.03 | 1,916 (2.1%) | 842 (2.1%) | 0.00 | 2517 (1.7%) | 1164 (1.6%) | 0.01 |
| Cystoscopy; n (%) | 257 (1.0%) | 131 (0.9%) | 0.01 | 504 (1.6%) | 210 (1.2%) | 0.03 | #REF! | #REF! | #REF! | #REF! | #REF! | #REF! |
| Other Covariates | | | | | | | | | | | | |
| Liver disease; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 938 (1.0%) | 501 (1.2%) | -0.02 | 938 (0.6%) | 501 (0.7%) | -0.01 |
| Osteoarthritis; n (%) | 4,861 (18.9%) | 3,135 (21.1%) | -0.06 | 5,140 (15.9%) | 3,000 (16.9%) | -0.03 | 20,522 (22.2%) | 10,442 (25.7%) | -0.08 | 30523 (20.3%) | 16577 (22.6%) | -0.06 |
| Other arthritis, arthropathies and musculoskeletal | | | | | | | | | | | | |
| pain; n (%) | 9,456 (36.8%) | 6,010 (40.4%) | -0.07 | 11,557 (35.8%) | 6,608 (37.2%) | -0.03 | 37,694 (40.8%) | 17,578 (43.2%) | -0.05 | 58707 (39.0%) | 30196 (41.2%) | -0.04 |
| Dorsopathies; n (%) | 5,242 (20.4%) | 3,469 (23.3%) | -0.07 | 5,958 (18.4%) | 3,826 (21.6%) | -0.08 | 20,625 (22.3%) | 10,095 (24.8%) | -0.06 | 31825 (21.2%) | 17390 (23.7%) | -0.06 |
| Fractures; n (%) | 1,067 (4.2%) | 569 (3.8%) | 0.02 | 1,475 (4.6%) | 655 (3.7%) | 0.05 | 5,670 (6.1%) | 2,346 (5.8%) | 0.01 | 8212 (5.5%) | 3570 (4.9%) | 0.03 |
| Falls v2; n (%) Osteoporosis; n (%) | 1,290 (5.0%)<br>2,120 (8.2%) | 750 (5.0%)<br>1,174 (7.9%) | 0.00<br>0.01 | 625 (1.9%)<br>2,196 (6.8%) | 333 (1.9%)<br>977 (5.5%) | 0.00<br>0.05 | 2,916 (3.2%)<br>9,398 (10.2%) | 1,273 (3.1%)<br>4,284 (10.5%) | 0.01<br>-0.01 | 4831 (3.2%)<br>13714 (9.1%) | 2356 (3.2%)<br>6435 (8.8%) | 0.00<br>0.01 |
| Hyperthyroidism; n (%) | 301 (1.2%) | 1,174 (7.5%) | -0.01 | 2,196 (0.8%) | 192 (1.1%) | -0.03 | 1,116 (1.2%) | 562 (1.4%) | -0.01 | 1679 (1.1%) | 944 (1.3%) | -0.02 |
| Hypothyroidism v2; n (%) | 4,578 (17.8%) | 2,866 (19.3%) | -0.01 | 3,919 (12.1%) | 2,552 (14.4%) | -0.03 | 14,603 (15.8%) | 5,985 (14.7%) | 0.03 | 23100 (15.4%) | 11403 (15.6%) | -0.02 |
| Other disorders of thyroid gland V2; n (%) | 785 (3.1%) | 608 (4.1%) | -0.05 | 861 (2.7%) | 677 (3.8%) | -0.06 | 3,132 (3.4%) | 1,569 (3.9%) | -0.03 | 4778 (3.2%) | 2854 (3.9%) | -0.04 |
| Depression; n (%) | 1,966 (7.6%) | 1,253 (8.4%) | -0.03 | 1,876 (5.8%) | 1,092 (6.2%) | -0.02 | 9,551 (10.3%) | 4,998 (12.3%) | -0.06 | 13393 (8.9%) | 7343 (10.0%) | -0.04 |
| Anxiety; n (%) | 1,921 (7.5%) | 1,548 (10.4%) | -0.10 | 1,417 (4.4%) | 1,206 (6.8%) | -0.10 | 7,883 (8.5%) | 4,932 (12.1%) | -0.12 | 11221 (7.5%) | 7686 (10.5%) | -0.10 |
| Sleep_Disorder; n (%) | 2,242 (8.7%) | 1,139 (7.7%) | 0.04 | 3,395 (10.5%) | 2,017 (11.4%) | -0.03 | 8,029 (8.7%) | 3,474 (8.5%) | 0.01 | 13666 (9.1%) | 6630 (9.0%) | 0.00 |
| Dementia; n (%) | 1,801 (7.0%) | 1,125 (7.6%) | -0.02 | 1,911 (5.9%) | 830 (4.7%) | 0.05 | 8,977 (9.7%) | 4,265 (10.5%) | -0.03 | 12689 (8.4%) | 6220 (8.5%) | 0.00 |
| Delirium; n (%) | 416 (1.6%) | 261 (1.8%) | -0.02 | 521 (1.6%) | 228 (1.3%) | 0.03 | 2,706 (2.9%) | 1,367 (3.4%) | -0.03 | 3643 (2.4%) | 1856 (2.5%) | -0.01 |
| Psychosis; n (%) | 319 (1.2%) | 176 (1.2%) | 0.00 | 441 (1.4%) | 190 (1.1%) | 0.03 | 2,089 (2.3%) | 961 (2.4%) | -0.01 | 2849 (1.9%) | 1327 (1.8%) | 0.01 |
| Obesity; n (%) | 2,962 (11.5%) | 2,712 (18.2%) | -0.19 | 2,363 (7.3%) | 2,324 (13.1%) | -0.19 | 11,623 (12.6%) | 6,894 (17.0%) | -0.12 | 16948 (11.3%) | 11930 (16.3%) | -0.15 |
| Overweight; n (%) | 887 (3.5%) | 894 (6.0%) | -0.12 | 356 (1.1%) | 426 (2.4%) | -0.10 | 2,338 (2.5%) | 1,512 (3.7%) | -0.07 | 3581 (2.4%) | 2832 (3.9%) | -0.09 |
| Smoking; n (%) | 3,155 (12.3%) | 2,794 (18.8%) | -0.18 | 1,598 (4.9%) | 1,423 (8.0%) | -0.13 | 19,504 (21.1%) | 11,882 (29.2%) | -0.19 | 24257 (16.1%) | 16099 (22.0%) | -0.15 |
| Alcohol abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 51 (0.1%) | 32 (0.1%) | 0.00 | 51 (0.0%) | 32 (0.0%) | #DIV/0! |
| Drug abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 123 (0.1%) | 108 (0.3%) | -0.04 | 123 (0.1%) | 108 (0.1%) | 0.00 |

| COPD; n (%) | 4,309 (16.8%) | 2,430 (16.3%) | 0.01 | 4,571 (14.2%) | 2,352 (13.3%) | 0.03 | 18,074 (19.6%) | 8,952 (22.0%) | -0.06 | 26954 (17.9%) | 13734 (18.7%) | -0.02 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Asthma; n (%) | 1,542 (6.0%) | 1,081 (7.3%) | -0.05 | 1,625 (5.0%) | 1,171 (6.6%) | -0.07 | 6,360 (6.9%) | 3,495 (8.6%) | -0.06 | 9527 (6.3%) | 5747 (7.8%) | -0.06 |
| Obstructive sleep apnea; n (%) | 2,457 (9.6%) | 1,923 (12.9%) | -0.10 | 2,936 (9.1%) | 2,260 (12.7%) | -0.12 | 7,564 (8.2%) | 4,077 (10.0%) | -0.06 | 12957 (8.6%) | 8260 (11.3%) | -0.09 |
| Pneumonia; n (%) | 1,531 (6.0%) | 901 (6.1%) | 0.00 | 1,914 (5.9%) | 1,034 (5.8%) | 0.00 | 8,764 (9.5%) | 4,313 (10.6%) | -0.04 | 12209 (8.1%) | 6248 (8.5%) | -0.01 |
| Imaging; n (%) | 36 (0.1%) | 27 (0.2%) | -0.03 | 44 (0.1%) | 15 (0.1%) | 0.00 | 3,729 (4.0%) | 1,328 (3.3%) | 0.04 | 3809 (2.5%) | 1370 (1.9%) | 0.04 |
| Other Medications | 50 (0.170) | 27 (0.270) | 0.05 | 11(0.270) | 13 (0.170) | 0.00 | 3,723 (1.070) | 1,520 (5.570) | 0.01 | 3003 (2.374) | 1370 (1.370) | 0.01 |
| Use of ACE inhibitors; n (%) | 9,773 (38.0%) | 5,230 (35.2%) | 0.06 | 11,540 (35.7%) | 6,215 (35.0%) | 0.01 | 35,261 (38.2%) | 15,477 (38.1%) | 0.00 | 56574 (37.6%) | 26922 (36.7%) | 0.02 |
| Use of ARBs; n (%) | 5,359 (20.9%) | 3,889 (26.2%) | -0.13 | 7,683 (23.8%) | 4,892 (27.6%) | -0.09 | 20,854 (22.6%) | 10,920 (26.9%) | -0.10 | 33896 (22.5%) | 19701 (26.9%) | -0.10 |
| Use of Loop Diuretics - United; n (%) | 7,760 (30.2%) | 3,674 (24.7%) | 0.12 | 10,702 (33.1%) | 3,963 (22.3%) | 0.24 | 40,069 (43.4%) | 15,255 (37.5%) | 0.12 | 58531 (38.9%) | 22892 (31.2%) | 0.16 |
| Use of other diuretics- United; n (%) | 1,535 (6.0%) | 731 (4.9%) | 0.05 | 2,341 (7.2%) | 878 (4.9%) | 0.10 | 7,877 (8.5%) | 2,806 (6.9%) | 0.06 | 11753 (7.8%) | 4415 (6.0%) | 0.07 |
| Use of nitrates-United; n (%) | 2,055 (8.0%) | 1,038 (7.0%) | 0.04 | 3,094 (9.6%) | 1,354 (7.6%) | 0.07 | 10,921 (11.8%) | 4,642 (11.4%) | 0.01 | 16070 (10.7%) | 7034 (9.6%) | 0.04 |
| Use of other hypertension drugs; n (%) | 2,028 (7.9%) | 1,125 (7.6%) | 0.01 | 2,574 (8.0%) | 1,303 (7.3%) | 0.03 | 7,958 (8.6%) | 3,455 (8.5%) | 0.00 | 12560 (8.4%) | 5883 (8.0%) | 0.01 |
| Use of digoxin- United; n (%) | 4,005 (15.6%) | 1,311 (8.8%) | 0.21 | 6,378 (19.7%) | 1,975 (11.1%) | 0.24 | 17,796 (19.3%) | 5,477 (13.5%) | 0.16 | 28179 (18.7%) | 8763 (12.0%) | 0.19 |
| Use of Anti-arrhythmics; n (%) | 2,453 (9.5%) | 2,071 (13.9%) | -0.14 | 3,881 (12.0%) | 2,847 (16.0%) | -0.12 | 10,257 (11.1%) | 6,110 (15.0%) | -0.12 | 16591 (11.0%) | 11028 (15.1%) | -0.12 |
| Use of COPD/asthma meds-United; n (%) | 4,206 (16.4%) | 2,858 (19.2%) | -0.07 | 5,916 (18.3%) | 3,513 (19.8%) | -0.04 | 18,597 (20.1%) | 9,406 (23.1%) | -0.07 | 28719 (19.1%) | 15777 (21.5%) | -0.06 |
| Use of statins; n (%) | 15,187 (59.1%) | 9,008 (60.6%) | -0.03 | 19,252 (59.6%) | 10,616 (59.8%) | 0.00 | 56,100 (60.7%) | 25,111 (61.8%) | -0.02 | 90539 (60.2%) | 44735 (61.1%) | -0.02 |
| Use of other lipid-lowering drugs; n (%) | 1,698 (6.6%) | 959 (6.4%) | 0.01 | 3,164 (9.8%) | 1,658 (9.3%) | 0.02 | 6,803 (7.4%) | 2,989 (7.4%) | 0.00 | 11665 (7.8%) | 5606 (7.7%) | 0.00 |
| Use of antiplatelet agents; n (%) | 2,667 (10.4%) | 2,234 (15.0%) | -0.14 | 4,187 (13.0%) | 2,985 (16.8%) | -0.11 | 12,151 (13.2%) | 7,088 (17.4%) | -0.12 | 19005 (12.6%) | 12307 (16.8%) | -0.12 |
| Use of heparin and other low-molecular weight | | | | | | | | | | | | |
| heparins; n (%) | 1,027 (4.0%) | 48 (0.3%) | 0.26 | 13 (0.0%) | 2 (0.0%) | #DIV/0! | 5,378 (5.8%) | 271 (0.7%) | 0.29 | 6418 (4.3%) | 321 (0.4%) | 0.26 |
| Use of NSAIDs; n (%) | 2,211 (8.6%) | 1,854 (12.5%) | -0.13 | 2,679 (8.3%) | 2,192 (12.4%) | -0.13 | 8,445 (9.1%) | 5,496 (13.5%) | -0.14 | 13335 (8.9%) | 9542 (13.0%) | -0.13 |
| Use of oral corticosteroids; n (%) | 4,525 (17.6%) | 3,114 (20.9%) | -0.08 | 5,871 (18.2%) | 3,585 (20.2%) | -0.05 | 20,413 (22.1%) | 10,417 (25.6%) | -0.08 | 30809 (20.5%) | 17116 (23.4%) | -0.07 |
| Use of bisphosphonate (United); n (%) | 1,032 (4.0%) | 504 (3.4%) | 0.03 | 1,328 (4.1%) | 488 (2.7%) | 0.08 | 3,634 (3.9%) | 1,530 (3.8%) | 0.01 | 5994 (4.0%) | 2522 (3.4%) | 0.03 |
| Use of opioids- United; n (%) | 5,799 (22.6%) | 3,261 (21.9%) | 0.02 | 7,739 (24.0%) | 4,176 (23.5%) | 0.01 | 25,851 (28.0%) | 11,903 (29.3%) | -0.03 | 39389 (26.2%) | 19340 (26.4%) | 0.00 |
| Use of antidepressants; n (%) | 4,895 (19.0%) | 3,065 (20.6%) | -0.04 | 6,023 (18.6%) | 3,323 (18.7%) | 0.00 | 22,801 (24.7%) | 10,978 (27.0%) | -0.05 | 33719 (22.4%) | 17366 (23.7%) | -0.03 |
| Use of antipsychotics; n (%) | 375 (1.5%) | 238 (1.6%) | -0.01 | 504 (1.6%) | 250 (1.4%) | 0.02 | 2,418 (2.6%) | 1,335 (3.3%) | -0.04 | 3297 (2.2%) | 1823 (2.5%) | -0.02 |
| Use of anticonvulsants; n (%) | 2,989 (11.6%) | 1,777 (12.0%) | -0.01 | 3,445 (10.7%) | 1,742 (9.8%) | 0.03 | 13,599 (14.7%) | 6,653 (16.4%) | -0.05 | 20033 (13.3%) | 10172 (13.9%) | -0.02 |
| Use of lithium- United; n (%) | 13 (0.1%) | 12 (0.1%) | 0.00 | 23 (0.1%) | 18 (0.1%) | 0.00 | 29 (0.0%) | 30 (0.1%) | -0.04 | 65 (0.0%) | 60 (0.1%) | -0.04 |
| Use of Benzos- United; n (%) | 2,295 (8.9%) | 1,810 (12.2%) | -0.11 | 4,007 (12.4%) | 2,389 (13.5%) | -0.03 | 10,742 (11.6%) | 6,233 (15.3%) | -0.11 | 17044 (11.3%) | 10432 (14.2%) | -0.09 |
| Use of anxiolytics/hypnotics-United; n (%) | 1,231 (4.8%) | 865 (5.8%) | -0.04 | 2,019 (6.3%) | 1,221 (6.9%) | -0.02 | 5,918 (6.4%) | 3,005 (7.4%) | -0.04 | 9168 (6.1%) | 5091 (6.9%) | -0.03 |
| Use of dementia meds- United; n (%) | 988 (3.8%) | 571 (3.8%) | 0.00 | 1,481 (4.6%) | 546 (3.1%) | 0.08 | 5,159 (5.6%) | 2,315 (5.7%) | 0.00 | 7628 (5.1%) | 3432 (4.7%) | 0.02 |
| Use of antiparkinsonian meds- United; n (%) | 695 (2.7%) | 399 (2.7%) | 0.00 | 923 (2.9%) | 441 (2.5%) | 0.02 | 3,529 (3.8%) | 1,659 (4.1%) | -0.02 | 5147 (3.4%) | 2499 (3.4%) | 0.00 |
| Any use of pramlintide; n (%) | 3 (0.0%) | 3 (0.0%) | #DIV/0! | 4 (0.0%) | 2 (0.0%) | #DIV/0! | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Any use of 1st generation sulfonylureas; n (%) | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 14 (0.0%) | 1 (0.0%) | #DIV/0! | | | #VALUE! | #VALUE! | #VALUE! | 0.00 |
| Entresto (sacubitril/valsartan); n (%) | 64 (0.2%) | 67 (0.5%) | -0.05 | 18 (0.1%) | 29 (0.2%) | -0.03 | 87 (0.1%) | 88 (0.2%) | -0.03 | 169 (0.1%) | 184 (0.3%) | 0.00 |
| | | | | | | | | | | | 22.547 | |
| Labs | 2 444 (42 40/) | 2 COE (10 10/) | 0.43 | 45.6 (4.40/) | 242 (4 40/) | 0.00 | N1/A | N1/A | 49/411151 | 57,996 | 32,617 | 0.00 |
| Lab values-HbA1c (%) v3; n (%) | 3,444 (13.4%) | 2,695 (18.1%) | -0.13 | 456 (1.4%) | 242 (1.4%) | 0.00 | N/A | N/A | #VALUE! | 3,900 (6.7%) | 2,937 (9.0%) | -0.09 |
| Lab values- HbA1c (%) v3; n (%)<br>Lab values- HbA1c (%) (within 3 months) v3; n (%) | 2,217 (8.6%) | 1,747 (11.7%) | -0.10 | 321 (1.0%) | 170 (1.0%) | 0.00 | N/A | N/A | #VALUE! | 3,900 (6.7%)<br>2,538 (4.4%) | 2,937 (9.0%)<br>1,917 (5.9%) | -0.07 |
| Lab values- HbA1c (%) v3; n (%)<br>Lab values- HbA1c (%) (within 3 months) v3; n (%)<br>Lab values- HbA1c (%) (within 6 months) v3; n (%) | 2,217 (8.6%)<br>3,444 (13.4%) | 1,747 (11.7%)<br>2,695 (18.1%) | -0.10<br>-0.13 | 321 (1.0%)<br>456 (1.4%) | 170 (1.0%)<br>242 (1.4%) | 0.00<br>0.00 | N/A<br>N/A | N/A<br>N/A | #VALUE!<br>#VALUE! | 3,900 (6.7%)<br>2,538 (4.4%)<br>3,900 (6.7%) | 2,937 (9.0%)<br>1,917 (5.9%)<br>2,937 (9.0%) | -0.07<br>-0.09 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-HbA1c (%) (within 6 months) v3; n (%) Lab values-BNP; n (%) | 2,217 (8.6%)<br>3,444 (13.4%)<br>401 (1.6%) | 1,747 (11.7%)<br>2,695 (18.1%)<br>281 (1.9%) | -0.10<br>-0.13<br>-0.02 | 321 (1.0%)<br>456 (1.4%)<br>35 (0.1%) | 170 (1.0%)<br>242 (1.4%)<br>28 (0.2%) | 0.00<br>0.00<br>-0.03 | N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE!<br>#VALUE! | 3,900 (6.7%)<br>2,538 (4.4%)<br>3,900 (6.7%)<br>436 (0.8%) | 2,937 (9.0%)<br>1,917 (5.9%)<br>2,937 (9.0%)<br>309 (0.9%) | -0.07<br>-0.09<br>-0.01 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-HbA1c (%) (within 6 months) v3; n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) | 2,217 (8.6%)<br>3,444 (13.4%)<br>401 (1.6%)<br>281 (1.1%) | 1,747 (11.7%)<br>2,695 (18.1%)<br>281 (1.9%)<br>224 (1.5%) | -0.10<br>-0.13<br>-0.02<br>-0.04 | 321 (1.0%)<br>456 (1.4%)<br>35 (0.1%)<br>28 (0.1%) | 170 (1.0%)<br>242 (1.4%)<br>28 (0.2%)<br>18 (0.1%) | 0.00<br>0.00<br>-0.03<br>0.00 | N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE!<br>#VALUE! | 3,900 (6.7%)<br>2,538 (4.4%)<br>3,900 (6.7%)<br>436 (0.8%)<br>309 (0.5%) | 2,937 (9.0%)<br>1,917 (5.9%)<br>2,937 (9.0%)<br>309 (0.9%)<br>242 (0.7%) | -0.07<br>-0.09<br>-0.01<br>-0.03 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-HbA1c (%) (within 6 months) v3; n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 6 months); n (%) | 2,217 (8.6%)<br>3,444 (13.4%)<br>401 (1.6%)<br>281 (1.1%)<br>401 (1.6%) | 1,747 (11.7%)<br>2,695 (18.1%)<br>281 (1.9%)<br>224 (1.5%)<br>281 (1.9%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02 | 321 (1.0%)<br>456 (1.4%)<br>35 (0.1%)<br>28 (0.1%)<br>35 (0.1%) | 170 (1.0%)<br>242 (1.4%)<br>28 (0.2%)<br>18 (0.1%)<br>28 (0.2%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03 | N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE!<br>#VALUE!<br>#VALUE! | 3,900 (6.7%)<br>2,538 (4.4%)<br>3,900 (6.7%)<br>436 (0.8%)<br>309 (0.5%)<br>436 (0.8%) | 2,937 (9.0%)<br>1,917 (5.9%)<br>2,937 (9.0%)<br>309 (0.9%)<br>242 (0.7%)<br>309 (0.9%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-HbA1c (%) (within 6 months) v3; n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) | 2,217 (8.6%)<br>3,444 (13.4%)<br>401 (1.6%)<br>281 (1.1%)<br>401 (1.6%)<br>6,014 (23.4%) | 1,747 (11.7%)<br>2,695 (18.1%)<br>281 (1.9%)<br>224 (1.5%)<br>281 (1.9%)<br>4,675 (31.4%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18 | 321 (1.0%)<br>456 (1.4%)<br>35 (0.1%)<br>28 (0.1%)<br>35 (0.1%)<br>409 (1.3%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07 | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE!<br>#VALUE!<br>#VALUE!<br>#VALUE! | 3,900 (6.7%)<br>2,538 (4.4%)<br>3,900 (6.7%)<br>436 (0.8%)<br>309 (0.5%)<br>436 (0.8%)<br>6,423 (11.1%) | 2,937 (9.0%)<br>1,917 (5.9%)<br>2,937 (9.0%)<br>309 (0.9%)<br>242 (0.7%)<br>309 (0.9%)<br>5,065 (15.5%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-HbA1c (%) (within 6 months) v3; n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) | 2,217 (8.6%)<br>3,444 (13.4%)<br>401 (1.6%)<br>281 (1.1%)<br>401 (1.6%)<br>6,014 (23.4%)<br>4,107 (16.0%) | 1,747 (11.7%)<br>2,695 (18.1%)<br>281 (1.9%)<br>224 (1.5%)<br>281 (1.9%)<br>4,675 (31.4%)<br>3,320 (22.3%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16 | 321 (1.0%)<br>456 (1.4%)<br>35 (0.1%)<br>28 (0.1%)<br>35 (0.1%)<br>409 (1.3%)<br>282 (0.9%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06 | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! | 3,900 (6.7%)<br>2,538 (4.4%)<br>3,900 (6.7%)<br>436 (0.8%)<br>309 (0.5%)<br>436 (0.8%)<br>6,423 (11.1%)<br>4,389 (7.6%) | 2,937 (9.0%)<br>1,917 (5.9%)<br>2,937 (9.0%)<br>309 (0.9%)<br>242 (0.7%)<br>309 (0.9%)<br>5,065 (15.5%)<br>3,610 (11.1%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.12 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP; n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) | 2,217 (8.6%)<br>3,444 (13.4%)<br>401 (1.6%)<br>281 (1.1%)<br>401 (1.6%)<br>6,014 (23.4%)<br>4,107 (16.0%)<br>6,014 (23.4%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16<br>-0.18 | 321 (1.0%)<br>456 (1.4%)<br>35 (0.1%)<br>28 (0.1%)<br>35 (0.1%)<br>409 (1.3%)<br>282 (0.9%)<br>409 (1.3%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06<br>-0.07 | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE! | 3,900 (6.7%)<br>2,538 (4.4%)<br>3,900 (6.7%)<br>436 (0.8%)<br>309 (0.5%)<br>436 (0.8%)<br>6,423 (11.1%)<br>4,389 (7.6%)<br>6,423 (11.1%) | 2,937 (9.0%)<br>1,917 (5.9%)<br>2,937 (9.0%)<br>309 (0.9%)<br>242 (0.7%)<br>309 (0.9%)<br>5,065 (15.5%)<br>3,610 (11.1%)<br>5,065 (15.5%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.12<br>-0.13 |
| Lab values- HbA1c (%) v3; n (%) Lab values- HbA1c (%) (within 3 months) v3; n (%) Lab values- HbA1c (%) (within 6 months) v3; n (%) Lab values- BNP; n (%) Lab values- BNP (within 3 months); n (%) Lab values- BNP (within 6 months); n (%) Lab values- BUN (mg/dl); n (%) Lab values- BUN (mg/dl) (within 3 months); n (%) Lab values- BUN (mg/dl) (within 6 months); n (%) Lab values- Creatinine (mg/dl) v2; n (%) | 2,217 (8.6%)<br>3,444 (13.4%)<br>401 (1.6%)<br>281 (1.1%)<br>401 (1.6%)<br>6,014 (23.4%)<br>4,107 (16.0%) | 1,747 (11.7%)<br>2,695 (18.1%)<br>281 (1.9%)<br>224 (1.5%)<br>281 (1.9%)<br>4,675 (31.4%)<br>3,320 (22.3%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16 | 321 (1.0%)<br>456 (1.4%)<br>35 (0.1%)<br>28 (0.1%)<br>35 (0.1%)<br>409 (1.3%)<br>282 (0.9%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06 | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! | 3,900 (6.7%)<br>2,538 (4.4%)<br>3,900 (6.7%)<br>436 (0.8%)<br>309 (0.5%)<br>436 (0.8%)<br>6,423 (11.1%)<br>4,389 (7.6%) | 2,937 (9.0%)<br>1,917 (5.9%)<br>2,937 (9.0%)<br>309 (0.9%)<br>242 (0.7%)<br>309 (0.9%)<br>5,065 (15.5%)<br>3,610 (11.1%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.12 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP; n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) | 2,217 (8.6%)<br>3,444 (13.4%)<br>401 (1.6%)<br>281 (1.1%)<br>401 (1.6%)<br>6,014 (23.4%)<br>4,107 (16.0%)<br>6,014 (23.4%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16<br>-0.18 | 321 (1.0%)<br>456 (1.4%)<br>35 (0.1%)<br>28 (0.1%)<br>35 (0.1%)<br>409 (1.3%)<br>282 (0.9%)<br>409 (1.3%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06<br>-0.07 | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE! | 3,900 (6.7%)<br>2,538 (4.4%)<br>3,900 (6.7%)<br>436 (0.8%)<br>309 (0.5%)<br>436 (0.8%)<br>6,423 (11.1%)<br>4,389 (7.6%)<br>6,423 (11.1%) | 2,937 (9.0%)<br>1,917 (5.9%)<br>2,937 (9.0%)<br>309 (0.9%)<br>242 (0.7%)<br>309 (0.9%)<br>5,065 (15.5%)<br>3,610 (11.1%)<br>5,065 (15.5%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.12<br>-0.13 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP, n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNN (mg/dl); n (%) Lab values-BNN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months); v2; | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 6,112 (23.8%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16<br>-0.18<br>-0.20 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06<br>-0.07<br>-0.08 | N/A | N/A | #VALUE! | 3,900 (6.7%)<br>2,538 (4.4%)<br>3,900 (6.7%)<br>436 (0.8%)<br>309 (0.5%)<br>436 (0.8%)<br>6,423 (11.1%)<br>4,389 (7.6%)<br>6,423 (11.1%)<br>6,535 (11.3%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.12<br>-0.13<br>-0.14 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP; n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 6,112 (23.8%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16<br>-0.18<br>-0.20 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06<br>-0.07<br>-0.08 | N/A | N/A | #VALUE! | 3,900 (6.7%)<br>2,538 (4.4%)<br>3,900 (6.7%)<br>436 (0.8%)<br>309 (0.5%)<br>436 (0.8%)<br>6,423 (11.1%)<br>4,389 (7.6%)<br>6,423 (11.1%)<br>6,535 (11.3%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.12<br>-0.13<br>-0.14 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP; n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) (vithin 3 months); n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 6,112 (23.8%) 4,168 (16.2%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16<br>-0.18<br>-0.20 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06<br>-0.07<br>-0.08 | N/A | N/A | #VALUE! | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 436 (0.8%) 6,423 (11.1%) 4,389 (7.6%) 6,423 (11.1%) 6,535 (11.3%) 4,461 (7.7%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,055 (15.5%) 5,252 (16.1%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.12<br>-0.13<br>-0.14 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP( (%) (within 6 months) v3; n (%) Lab values-BNP, m(%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Etrainine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-HDL level (mg/dl); n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 6,112 (23.8%) 4,168 (16.2%) 6,112 (23.8%) 4,306 (16.8%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16<br>-0.18<br>-0.20<br>-0.18 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) 293 (0.9%) 423 (1.3%) 373 (1.2%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) 412 (2.3%) 270 (1.5%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06<br>-0.07<br>-0.08<br>-0.07 | N/A | N/A | #VALUE! | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 309 (0.5%) 436 (0.8%) 6,423 (11.1%) 4,389 (7.6%) 6,423 (11.1%) 6,535 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) 3,762 (11.5%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.12<br>-0.13<br>-0.14<br>-0.13 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP; n (%) Lab values-BNP; (within 6 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 4,112 (23.8%) 4,168 (16.2%) 6,112 (23.8%) 4,306 (16.8%) 2,689 (10.5%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16<br>-0.18<br>-0.20<br>-0.18<br>-0.20<br>-0.15 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 409 (1.3%) 409 (1.3%) 423 (1.3%) 423 (1.3%) 423 (1.3%) 373 (1.2%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) 308 (1.7%) 412 (2.3%) 270 (1.5%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06<br>-0.07<br>-0.08<br>-0.07<br>-0.08 | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 309 (0.5%) 436 (0.8%) 6,423 (11.1%) 6,535 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 5,065 (15.5%) 5,252 (16.1%) 3,762 (11.5%) 5,252 (16.1%) 3,679 (11.3%) 2,307 (7.1%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.12<br>-0.13<br>-0.14<br>-0.13 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP; n (%) Lab values-BNP; n (%) Lab values-BNP (within 6 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 3 months); n (%) Lab values-HDL level (mg/dl) (within 3 months); n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 6,112 (23.8%) 4,168 (16.2%) 6,112 (23.8%) 4,306 (16.8%) 2,689 (10.5%) 4,306 (16.8%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) 3,409 (22.9%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16<br>-0.18<br>-0.20<br>-0.18<br>-0.20<br>-0.15 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) 293 (0.9%) 423 (1.3%) 373 (1.2%) 373 (1.2%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) 308 (1.7%) 412 (2.3%) 270 (1.5%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06<br>-0.07<br>-0.08<br>-0.07<br>-0.08<br>-0.03 | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 436 (0.8%) 436 (0.8%) 6,423 (11.1%) 6,423 (11.1%) 6,535 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) 4,679 (8.1%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) 3,762 (11.5%) 5,252 (16.1%) 3,679 (11.3%) 2,307 (7.1%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.14<br>-0.13<br>-0.14<br>-0.11<br>-0.08 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP( (%) (within 6 months) v3; n (%) Lab values-BNP, m(%) Lab values-BNP (within 3 months); n (%) Lab values-BNN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 3 months); n (%) Lab values-HDL level (mg/dl) (within 3 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 4,112 (23.8%) 4,168 (16.2%) 6,112 (23.8%) 4,306 (16.8%) 2,689 (10.5%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16<br>-0.18<br>-0.20<br>-0.18<br>-0.20<br>-0.15 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 409 (1.3%) 409 (1.3%) 423 (1.3%) 423 (1.3%) 423 (1.3%) 373 (1.2%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) 308 (1.7%) 412 (2.3%) 270 (1.5%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06<br>-0.07<br>-0.08<br>-0.07<br>-0.08 | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 309 (0.5%) 436 (0.8%) 6,423 (11.1%) 6,535 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 5,065 (15.5%) 5,252 (16.1%) 3,762 (11.5%) 5,252 (16.1%) 3,679 (11.3%) 2,307 (7.1%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.12<br>-0.13<br>-0.14<br>-0.13 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP; n (%) Lab values-BNP; n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-LDL level (mg/dl) (vithin 6 months); n (%) Lab values-LDL level (mg/dl) (vithin 6 months); n (%) Lab values-LDL level (mg/dl) (vithin 6 months); n (%) Lab values-LDL level (mg/dl) (within 6 months); n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 4,107 (16.2%) 6,112 (23.8%) 4,168 (16.2%) 6,112 (23.8%) 4,306 (16.8%) 4,306 (16.8%) 4,523 (17.6%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) 3,409 (22.9%) 3,538 (23.8%) | 0.10<br>0.13<br>0.02<br>0.04<br>0.02<br>0.18<br>0.16<br>0.18<br>0.20<br>0.18<br>-0.20<br>-0.15<br>-0.12 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 409 (1.3%) 423 (1.3%) 423 (1.3%) 423 (1.3%) 373 (1.2%) 452 (1.4%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) 308 (1.7%) 412 (2.3%) 270 (1.5%) 270 (1.5%) 279 (1.6%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06<br>-0.07<br>-0.08<br>-0.07<br>-0.08<br>-0.03<br>-0.03 | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 436 (0.8%) 436 (0.8%) 6,423 (11.1%) 6,535 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) 4,679 (8.1%) 4,975 (8.6%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 309 (0.9%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) 3,762 (11.5%) 5,252 (16.1%) 3,679 (11.3%) 2,307 (7.1%) 3,679 (11.3%) 3,817 (11.7%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.12<br>-0.13<br>-0.14<br>-0.13<br>-0.14<br>-0.11<br>-0.08 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP; n (%) Lab values-BNP; n (%) Lab values-BNP (within 6 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 3 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-LDL level (mg/dl) (within 6 months); n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) Lab values-LDL level (mg/dl) (within 3 months) v2; n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 6,112 (23.8%) 4,168 (16.2%) 6,112 (23.8%) 4,306 (16.8%) 2,689 (10.5%) 4,306 (16.8%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) 3,409 (22.9%) | -0.10<br>-0.13<br>-0.02<br>-0.04<br>-0.02<br>-0.18<br>-0.16<br>-0.18<br>-0.20<br>-0.18<br>-0.20<br>-0.15 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) 293 (0.9%) 423 (1.3%) 373 (1.2%) 373 (1.2%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) 308 (1.7%) 412 (2.3%) 270 (1.5%) | 0.00<br>0.00<br>-0.03<br>0.00<br>-0.03<br>-0.07<br>-0.06<br>-0.07<br>-0.08<br>-0.07<br>-0.08<br>-0.03 | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 436 (0.8%) 436 (0.8%) 6,423 (11.1%) 6,423 (11.1%) 6,535 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) 4,679 (8.1%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) 3,762 (11.5%) 5,252 (16.1%) 3,679 (11.3%) 2,307 (7.1%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.14<br>-0.13<br>-0.14<br>-0.11<br>-0.08 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP, n (%) Lab values-BNP, within 3 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-HDL level (mg/dl); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 3 months); n (%) Lab values-HDL level (mg/dl) (within 3 months); n (%) Lab values-LDL level (mg/dl) (vithin 6 months); n (%) Lab values-LDL level (mg/dl) (within 3 months) v2; n (%) Lab values-LDL level (mg/dl) (within 3 months) v2; n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 6,112 (23.8%) 4,168 (16.2%) 6,112 (23.8%) 4,306 (16.8%) 2,689 (10.5%) 4,306 (16.8%) 4,2835 (11.0%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) 3,409 (22.9%) 3,538 (23.8%) 2,212 (14.9%) | -0.10 -0.13 -0.02 -0.04 -0.02 -0.18 -0.16 -0.18 -0.20 -0.18 -0.20 -0.15 -0.12 -0.15 -0.12 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) 293 (0.9%) 423 (1.3%) 373 (1.2%) 452 (1.4%) 296 (0.9%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 330 (2.2%) 412 (2.3%) 412 (2.3%) 270 (1.5%) 270 (1.5%) 279 (1.6%) 185 (1.0%) | 0.00 0.00 -0.03 0.00 -0.03 -0.07 -0.08 -0.07 -0.08 -0.07 -0.08 -0.03 -0.02 -0.03 -0.02 | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 436 (0.8%) 6,423 (11.1%) 4,389 (7.6%) 6,423 (11.1%) 6,535 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) 4,975 (8.6%) 3,131 (5.4%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) 3,679 (11.3%) 2,307 (7.1%) 3,679 (11.3%) 3,817 (11.7%) 2,397 (7.3%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.14<br>-0.13<br>-0.14<br>-0.11<br>-0.08 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP1c (%) (within 6 months) v3; n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNN (mig/dl); n (%) Lab values-BNN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-LDL level (mg/dl) (vithin 6 months); n (%) Lab values-LDL level (mg/dl) (vithin 6 months) v2; n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 2811 (1.1%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.8%) 4,168 (16.2%) 6,112 (23.8%) 4,306 (16.8%) 2,689 (10.5%) 4,306 (16.8%) 2,835 (11.0%) 4,523 (17.6%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) 3,538 (23.8%) 2,212 (14.9%) 3,538 (23.8%) | -0.10 -0.13 -0.02 -0.04 -0.02 -0.18 -0.16 -0.18 -0.20 -0.18 -0.20 -0.15 -0.15 -0.15 -0.15 -0.15 -0.15 -0.15 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) 293 (0.9%) 421 (1.3%) 373 (1.2%) 452 (1.4%) 452 (1.4%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) 412 (2.3%) 270 (1.5%) 181 (1.0%) 279 (1.6%) 185 (1.0%) | 0.00 0.00 -0.03 -0.07 -0.08 -0.07 -0.08 -0.03 -0.07 -0.08 -0.07 -0.08 -0.01 -0.02 | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 436 (0.8%) 436 (0.8%) 6,423 (11.1%) 6,323 (11.1%) 6,535 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) 2,940 (5.1%) 4,975 (8.6%) 4,975 (8.6%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) 3,762 (11.5%) 5,252 (16.1%) 3,679 (11.3%) 2,307 (7.1%) 3,817 (11.7%) 2,397 (7.3%) 3,817 (11.7%) | -0.07 -0.09 -0.01 -0.03 -0.01 -0.13 -0.12 -0.13 -0.14 -0.13 -0.14 -0.11 -0.08 -0.10 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP; n (%) Lab values-BNP; (within 6 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 4,107 (16.0%) 6,112 (23.8%) 4,168 (16.2%) 6,112 (23.8%) 2,689 (10.5%) 4,306 (16.8%) 4,523 (17.6%) 2,835 (11.0%) 4,523 (17.6%) 4,60.2%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) 3,409 (22.9%) 3,538 (23.8%) 2,212 (14.9%) 3,538 (23.8%) 41 (0.3%) | -0.10 -0.13 -0.02 -0.04 -0.02 -0.18 -0.16 -0.18 -0.20 -0.15 -0.12 -0.15 -0.12 -0.15 -0.12 -0.15 -0.12 -0.15 -0.12 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) 293 (0.9%) 423 (1.3%) 373 (1.2%) 452 (1.4%) 296 (0.9%) 452 (1.4%) 5 (0.0%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) 308 (1.7%) 412 (2.3%) 270 (1.5%) 270 (1.5%) 279 (1.6%) 485 (1.0%) 279 (1.6%) 4 (0.0%) | 0.00 0.00 -0.03 -0.07 -0.06 -0.07 -0.08 -0.07 -0.08 -0.02 -0.03 -0.02 #DIV/0! | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 309 (0.5%) 436 (0.8%) 6.423 (11.1%) 6,535 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) 4,975 (8.6%) 3,131 (5.4%) 4,975 (8.6%) 53 (0.1%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,055 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) 3,762 (11.5%) 5,252 (16.1%) 3,679 (11.3%) 2,307 (7.1%) 3,679 (11.3%) 3,817 (11.7%) 2,397 (7.3%) 3,817 (11.7%) 45 (0.1%) | -0.07<br>-0.09<br>-0.01<br>-0.03<br>-0.01<br>-0.13<br>-0.14<br>-0.13<br>-0.14<br>-0.11<br>-0.08 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP; n (%) Lab values-BNP; n (%) Lab values-BNP (within 6 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BNN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) Lab values-NT-proBNP; n (%) Lab values-NT-proBNP; n (%) Lab values-NT-proBNP; n (%) Lab values-NT-proBNP; n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.8%) 4,168 (16.2%) 4,168 (16.2%) 4,306 (16.8%) 2,689 (10.5%) 4,306 (16.8%) 4,523 (17.6%) 2,835 (11.0%) 4,523 (17.6%) 37 (0.1%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) 3,409 (22.9%) 3,538 (23.8%) 2,212 (14.9%) 3,538 (23.8%) 41 (0.3%) 34 (0.2%) | -0.10 -0.13 -0.02 -0.04 -0.02 -0.18 -0.16 -0.18 -0.20 -0.18 -0.21 -0.15 -0.12 -0.15 -0.12 -0.15 -0.12 -0.15 -0.10 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) 293 (0.9%) 423 (1.3%) 373 (1.2%) 452 (1.4%) 296 (0.9%) 452 (1.4%) 5 (0.0%) 2 (0.0%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) 308 (1.7%) 412 (2.3%) 270 (1.5%) 279 (1.6%) 185 (1.0%) 279 (1.6%) 4 (0.0%) 3 (0.0%) | 0.00 0.00 -0.03 -0.07 -0.08 -0.07 -0.08 -0.02 -0.01 -0.02 #DIV/0! | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 309 (0.5%) 436 (0.8%) 6,423 (11.1%) 6,523 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) 2,940 (5.1%) 4,975 (8.6%) 3,131 (5.4%) 4,975 (8.6%) 53 (0.1%) 39 (0.1%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) 3,672 (11.5%) 2,307 (7.1%) 3,679 (11.3%) 3,817 (11.7%) 45 (0.1%) 37 (0.1%) | -0.07 -0.09 -0.01 -0.03 -0.01 -0.13 -0.12 -0.13 -0.14 -0.13 -0.14 -0.11 -0.08 -0.10 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP, n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNN (mg/dl); n (%) Lab values-BNN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-LDL level (mg/dl) (within 6 months); n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) Lab values-NT-proBNP; n (%) Lab values-NT-proBNP; n (%) Lab values-NT-proBNP (within 3 months); n (%) Lab values-NT-proBNP (within 3 months); n (%) Lab values-NT-proBNP (within 6 months); n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 6,112 (23.8%) 4,168 (16.2%) 6,112 (23.8%) 4,306 (16.8%) 2,689 (10.5%) 4,306 (16.8%) 4,523 (17.6%) 4,802 (17.6%) 48 (0.2%) 37 (0.1%) 48 (0.2%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) 3,409 (22.9%) 2,126 (14.3%) 3,409 (22.9%) 3,538 (23.8%) 4,1 (0.3%) 34 (0.2%) 41 (0.3%) | -0.10 -0.13 -0.02 -0.04 -0.02 -0.18 -0.16 -0.18 -0.20 -0.18 -0.20 -0.15 -0.12 -0.15 -0.12 -0.15 -0.12 -0.15 -0.12 -0.15 -0.10 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) 293 (0.9%) 423 (1.3%) 373 (1.2%) 251 (0.8%) 373 (1.2%) 452 (1.4%) 5 (0.0%) 5 (0.0%) 5 (0.0%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 330 (2.2%) 412 (2.3%) 308 (1.7%) 412 (2.3%) 270 (1.5%) 270 (1.5%) 279 (1.6%) 485 (1.0%) 279 (1.6%) 4 (0.0%) 3 (0.0%) 4 (0.0%) | 0.00 0.00 -0.03 -0.07 -0.08 -0.07 -0.08 -0.07 -0.08 -0.01 -0.02 #DIV/0! #DIV/0! | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 399 (0.5%) 436 (0.8%) 6,423 (11.1%) 6,535 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) 2,940 (5.1%) 4,975 (8.6%) 3,131 (5.4%) 4,975 (8.6%) 53 (0.1%) 39 (0.1%) 53 (0.1%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) 3,762 (11.5%) 5,252 (16.1%) 3,679 (11.3%) 2,307 (7.1%) 3,817 (11.7%) 45 (0.1%) 37 (0.1%) 45 (0.1%) | -0.07 -0.09 -0.01 -0.03 -0.01 -0.13 -0.14 -0.13 -0.14 -0.11 -0.08 -0.10 -0.08 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP; n (%) Lab values-BNP; n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 6 months); n (%) Lab values-BUN (mg/dl); n (%) Lab values-BUN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-LDL level (mg/dl) (vithin 6 months); n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) Lab values-NDL level (mg/dl) (within 6 months); n (%) Lab values-NT-proBNP; n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (1.6%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 4,107 (16.0%) 6,014 (23.8%) 4,168 (16.2%) 4,168 (16.2%) 4,306 (16.8%) 2,689 (10.5%) 4,306 (16.8%) 4,523 (17.6%) 2,835 (11.0%) 4,523 (17.6%) 37 (0.1%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) 3,409 (22.9%) 3,538 (23.8%) 2,212 (14.9%) 3,538 (23.8%) 41 (0.3%) 34 (0.2%) | -0.10 -0.13 -0.02 -0.04 -0.02 -0.18 -0.16 -0.18 -0.20 -0.18 -0.21 -0.15 -0.12 -0.15 -0.12 -0.15 -0.12 -0.15 -0.10 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) 293 (0.9%) 423 (1.3%) 373 (1.2%) 452 (1.4%) 296 (0.9%) 452 (1.4%) 5 (0.0%) 2 (0.0%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 390 (2.2%) 412 (2.3%) 308 (1.7%) 412 (2.3%) 270 (1.5%) 279 (1.6%) 185 (1.0%) 279 (1.6%) 4 (0.0%) 3 (0.0%) | 0.00 0.00 -0.03 -0.07 -0.08 -0.07 -0.08 -0.02 -0.01 -0.02 #DIV/0! | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 309 (0.5%) 436 (0.8%) 6,423 (11.1%) 6,523 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) 2,940 (5.1%) 4,975 (8.6%) 3,131 (5.4%) 4,975 (8.6%) 53 (0.1%) 39 (0.1%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) 3,672 (11.5%) 2,307 (7.1%) 3,679 (11.3%) 3,817 (11.7%) 45 (0.1%) 37 (0.1%) | -0.07 -0.09 -0.01 -0.03 -0.01 -0.13 -0.12 -0.13 -0.14 -0.13 -0.14 -0.11 -0.08 -0.10 |
| Lab values-HbA1c (%) v3; n (%) Lab values-HbA1c (%) (within 3 months) v3; n (%) Lab values-BhP, n (%) Lab values-BNP; n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNP (within 3 months); n (%) Lab values-BNN (mg/dl); n (%) Lab values-BNN (mg/dl) (within 3 months); n (%) Lab values-BUN (mg/dl) (within 6 months); n (%) Lab values-Creatinine (mg/dl) v2; n (%) Lab values-Creatinine (mg/dl) (within 3 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-HDL level (mg/dl) (within 6 months); n (%) Lab values-LDL level (mg/dl) (within 6 months); n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) Lab values-NT-proBNP; n (%) Lab values-NT-proBNP; n (%) Lab values-NT-proBNP (within 3 months); n (%) Lab values-NT-proBNP (within 3 months); n (%) Lab values-NT-proBNP (within 6 months); n (%) | 2,217 (8.6%) 3,444 (13.4%) 401 (1.6%) 281 (1.1%) 401 (23.4%) 4,107 (16.0%) 6,014 (23.4%) 6,112 (23.8%) 4,168 (16.2%) 6,112 (23.8%) 4,306 (16.8%) 2,689 (10.5%) 4,306 (16.8%) 4,523 (17.6%) 4,802 (17.6%) 48 (0.2%) 37 (0.1%) 48 (0.2%) | 1,747 (11.7%) 2,695 (18.1%) 281 (1.9%) 224 (1.5%) 281 (1.9%) 4,675 (31.4%) 3,320 (22.3%) 4,675 (31.4%) 4,840 (32.6%) 3,454 (23.2%) 4,840 (32.6%) 3,409 (22.9%) 2,126 (14.3%) 3,409 (22.9%) 2,126 (14.3%) 3,409 (22.9%) 3,538 (23.8%) 4,1 (0.3%) 34 (0.2%) 41 (0.3%) | -0.10 -0.13 -0.02 -0.04 -0.02 -0.18 -0.16 -0.18 -0.20 -0.18 -0.20 -0.15 -0.12 -0.15 -0.12 -0.15 -0.12 -0.15 -0.12 -0.15 -0.10 | 321 (1.0%) 456 (1.4%) 35 (0.1%) 28 (0.1%) 35 (0.1%) 409 (1.3%) 282 (0.9%) 409 (1.3%) 423 (1.3%) 293 (0.9%) 423 (1.3%) 373 (1.2%) 251 (0.8%) 373 (1.2%) 452 (1.4%) 5 (0.0%) 5 (0.0%) 5 (0.0%) | 170 (1.0%) 242 (1.4%) 28 (0.2%) 18 (0.1%) 28 (0.2%) 390 (2.2%) 290 (1.6%) 330 (2.2%) 412 (2.3%) 308 (1.7%) 412 (2.3%) 270 (1.5%) 270 (1.5%) 279 (1.6%) 485 (1.0%) 279 (1.6%) 4 (0.0%) 3 (0.0%) 4 (0.0%) | 0.00 0.00 -0.03 -0.07 -0.08 -0.07 -0.08 -0.07 -0.08 -0.01 -0.02 #DIV/0! #DIV/0! | N/A | N/A | #VALUEI | 3,900 (6.7%) 2,538 (4.4%) 3,900 (6.7%) 436 (0.8%) 399 (0.5%) 436 (0.8%) 6,423 (11.1%) 6,535 (11.3%) 4,461 (7.7%) 6,535 (11.3%) 4,679 (8.1%) 2,940 (5.1%) 4,975 (8.6%) 3,131 (5.4%) 4,975 (8.6%) 53 (0.1%) 39 (0.1%) 53 (0.1%) | 2,937 (9.0%) 1,917 (5.9%) 2,937 (9.0%) 309 (0.9%) 242 (0.7%) 309 (0.9%) 5,065 (15.5%) 3,610 (11.1%) 5,065 (15.5%) 5,252 (16.1%) 3,762 (11.5%) 5,252 (16.1%) 3,679 (11.3%) 2,307 (7.1%) 3,817 (11.7%) 45 (0.1%) 37 (0.1%) 45 (0.1%) | -0.07 -0.09 -0.01 -0.03 -0.01 -0.13 -0.12 -0.13 -0.14 -0.11 -0.08 -0.10 -0.08 -0.10 -0.00 |

| Lab values-Total cholesterol (mg/dl) (within 6 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| months) v2; n (%) | 4,382 (17.0%) | 3,446 (23.2%) | -0.16 | 372 (1.2%) | 269 (1.5%) | -0.03 | N/A | N/A | #VALUE! | 4,754 (8.2%) | 3,715 (11.4%) | -0.11 |
| Lab values-Triglyceride level (mg/dl); n (%) | 4,300 (16.7%) | 3,427 (23.0%) | -0.16 | 358 (1.1%) | 271 (1.5%) | -0.04 | N/A | N/A | #VALUE! | 4,658 (8.0%) | 3,698 (11.3%) | -0.11 |
| Lab values-Triglyceride level (mg/dl) (within 3 | | | | | | | | | | | | |
| months); n (%) | 2,685 (10.4%) | 2,139 (14.4%) | -0.12 | 240 (0.7%) | 182 (1.0%) | -0.03 | N/A | N/A | #VALUE! | 2,925 (5.0%) | 2,321 (7.1%) | -0.09 |
| Lab values-Triglyceride level (mg/dl) (within 6 | | | | | | | | | | | | |
| months); n (%) | 4,300 (16.7%) | 3,427 (23.0%) | -0.16 | 358 (1.1%) | 271 (1.5%) | -0.04 | N/A | N/A | #VALUE! | 4,658 (8.0%) | 3,698 (11.3%) | -0.11 |
| Lab result number-HbA1c (%) mean (only 2 to 20 | | | | | | | | | | | | |
| included) v4 | 3,412 | 2,685 | | 365 | 233 | | N/A | N/A | | 3,777 | 2,918 | |
| mean (sd) | 6.57 (1.15) | 6.43 (1.14) | 0.12 | 6.95 (1.39) | 6.74 (1.22) | 0.16 | N/A | N/A | #VALUE! | 6.61 (1.18) | 6.45 (1.15) | 0.14 |
| median [IQR] | 6.30 [5.90, 7.00] | 6.20 [5.70, 6.80] | 0.09 | 6.55 [6.05, 7.50] | 6.50 [6.00, 7.20] | 0.04 | N/A | N/A | #VALUE! | 6.32 (1.18) | 6.22 (1.15) | 0.09 |
| Missing; n (%) | 22,289 (86.7%) | 12,184 (81.9%) | 0.13 | 31,930 (98.9%) | 17,515 (98.7%) | 0.02 | N/A | N/A | #VALUE! | 54,219 (93.5%) | 29,699 (91.1%) | 0.09 |
| Lab result number-BNP mean v2 | 401 | 281 | | 35 | 28 | | N/A | N/A | | 436 | 309 | |
| mean (sd) | 321.38 (381.79) | 308.78 (481.63) | 0.03 | 534.56 (854.48) | 412.18 (586.24) | 0.17 | N/A | N/A | #VALUE! | 338.49 (438.16) | 318.15 (492.53) | 0.04 |
| median [IQR] | 217.00 [123.80, 376.80] | 197.00 [93.20, 325.50] | 0.05 | 187.50 [119.00, 531.25] | 148.90 [93.00, 375.75] | 0.05 | N/A | N/A | #VALUE! | 214.63 (438.16) | 192.64 (492.53) | 0.05 |
| Missing; n (%) | 25,300 (98.4%) | 14,588 (98.1%) | 0.02 | 32,260 (99.9%) | 17,720 (99.8%) | 0.03 | N/A | N/A | #VALUE! | 57,560 (99.2%) | 32,308 (99.1%) | 0.01 |
| Lab result number-BUN (mg/dl) mean v2 | 6,014 | 4,675 | | 409 | 390 | | N/A | N/A | | 6,423 | 5,065 | |
| mean (sd) | 18.98 (7.10) | 17.84 (5.88) | 0.17 | 19.26 (8.32) | 1,005.73 (11,839.99) | -0.12 | N/A | N/A | #VALUE! | 19.00 (7.18) | 93.91 (3282.21) | -0.03 |
| median [IQR] | 18.00 [14.33, 22.00] | 17.00 [14.00, 21.00] | 0.15 | 18.00 [15.00, 22.00] | 17.90 [15.00, 22.50] | 0.00 | N/A | N/A | #VALUE! | 18.00 (7.18) | #VALUE! | #VALUE! |
| Missing; n (%) | 19,687 (76.6%) | 10,194 (68.6%) | 0.18 | 31,886 (98.7%) | 17,358 (97.8%) | 0.07 | N/A | N/A | #VALUE! | 51,573 (88.9%) | 27,552 (84.5%) | 0.13 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 | | | | | | | | | | | | |
| to 15 included) v3 | 6,060 | 4,790 | | 413 | 403 | | N/A | N/A | | 6,473 | 5,193 | |
| mean (sd) | 1.00 (0.26) | 0.95 (0.23) | 0.20 | 1.03 (0.29) | 0.97 (0.23) | 0.23 | N/A | N/A | #VALUE! | 1.00 (0.26) | 0.95 (0.23) | 0.20 |
| median [IQR] | 0.96 [0.82, 1.12] | 0.93 [0.80, 1.07] | 0.12 | 0.99 [0.84, 1.17] | 0.96 [0.81, 1.10] | 0.11 | N/A | N/A | #VALUE! | 0.96 (0.26) | 0.93 (0.23) | 0.12 |
| Missing; n (%) | 19,641 (76.4%) | 10,079 (67.8%) | 0.19 | 31,882 (98.7%) | 17,345 (97.7%) | 0.08 | N/A | N/A | #VALUE! | 51,523 (88.8%) | 27,424 (84.1%) | 0.14 |
| Lab result number- HDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 4,306 | 3,409 | | 373 | 269 | | N/A | N/A | | 4,679 | 3,678 | |
| mean (sd) | 51.05 (16.15) | 52.83 (16.13) | -0.11 | 44.36 (16.11) | 46.29 (16.99) | -0.12 | N/A | N/A | #VALUE! | 50.52 (16.15) | 52.35 (16.20) | -0.11 |
| median [IQR] | 48.50 [40.00, 60.00] | 50.00 [41.67, 62.00] | -0.09 | 44.00 [34.75, 52.00] | 45.00 [37.00, 55.00] | -0.06 | N/A | N/A | #VALUE! | 48.14 (16.15) | 49.63 (16.20) | -0.09 |
| Missing; n (%) | 21,395 (83.2%) | 11,460 (77.1%) | 0.15 | 31,922 (98.8%) | 17,479 (98.5%) | 0.03 | N/A | N/A | #VALUE! | 53,317 (91.9%) | 28,939 (88.7%) | 0.11 |
| Lab result number-LDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 4,420 | 3,473 | | 367 | 269 | | N/A | N/A | | 4,787 | 3,742 | |
| mean (sd) | 85.74 (33.20) | 87.86 (33.40) | -0.06 | 81.43 (33.48) | 87.95 (39.03) | -0.18 | N/A | N/A | #VALUE! | 85.41 (33.22) | 87.87 (33.84) | -0.07 |
| median [IQR] | 81.00 [64.00, 104.00] | 84.00 [64.00, 106.00] | -0.09 | 79.00 [62.00, 101.00] | 86.00 [64.00, 110.25] | -0.19 | N/A | N/A | #VALUE! | 80.85 (33.22) | 84.14 (33.84) | -0.10 |
| Missing; n (%) | 21,281 (82.8%) | 11,396 (76.6%) | 0.15 | 31,928 (98.9%) | 17,479 (98.5%) | 0.04 | N/A | N/A | #VALUE! | 53,209 (91.7%) | 28,875 (88.5%) | 0.11 |
| Lab result number-Total cholesterol (mg/dl) mean | | | | | | | | | | | | |
| (only =<5000 included) v2 | 4,379 | 3,443 | | 372 | 267 | | N/A | N/A | | 4,751 | 3,710 | |
| mean (sd) | 162.98 (40.62) | 166.15 (40.57) | -0.08 | 153.52 (43.84) | 161.18 (52.03) | -0.16 | N/A | N/A | #VALUE! | 162.24 (40.88) | 165.79 (41.50) | -0.09 |
| median [IQR] | 158.50 [135.50, 186.00] | 162.00 [138.00, 189.00] | -0.09 | 154.00 [133.00, 176.00] | 159.00 [131.00, 191.00] | -0.10 | N/A | N/A | #VALUE! | 158.15 (40.88) | 161.78 (41.50) | -0.09 |
| Missing; n (%) | 21,322 (83.0%) | 11,426 (76.8%) | 0.16 | 31,923 (98.8%) | 17,481 (98.5%) | 0.03 | N/A | N/A | #VALUE! | 53,245 (91.8%) | 28,907 (88.6%) | 0.11 |
| Lab result number-Triglyceride level (mg/dl) mean | | | | | | | | | | | . , , | |
| (only =<5000 included) v2 | 4,300 | 3,427 | | 358 | 270 | | N/A | N/A | | 4,658 | 3,697 | |
| mean (sd) | 130.55 (80.73) | 125.44 (72.65) | 0.07 | 143.25 (85.57) | 128.35 (78.86) | 0.18 | N/A | N/A | #VALUE! | 131.53 (81.12) | 125.65 (73.13) | 0.08 |
| median [IQR] | 113.00 [82.00, 154.00] | 107.00 [80.00, 152.00] | 0.08 | 126.00 [88.00, 179.00] | 117.50 [79.75, 157.50] | 0.10 | N/A | N/A | #VALUE! | 114.00 (81.12) | 107.77 (73.13) | 0.08 |
| Missing; n (%) | 21,401 (83.3%) | 11,442 (77.0%) | 0.16 | 31,937 (98.9%) | 17,478 (98.5%) | 0.04 | N/A | N/A | #VALUE! | 53,338 (92.0%) | 28,920 (88.7%) | 0.11 |
| Lab result number- Hemoglobin mean (only >0 | . , , | . , , | | | , , , | | • | • | | . , , | | |
| included) | 4,383 | 3,561 | | 284 | 285 | | N/A | N/A | | 4,667 | 3,846 | |
| mean (sd) | 13.66 (1.55) | 13.78 (1.61) | -0.08 | 13.12 (2.32) | 815.42 (10,013.02) | -0.11 | N/A | N/A | #VALUE! | 13.63 (1.61) | 73.18 (2722.01) | -0.03 |
| median [IQR] | 13.60 [12.70, 14.70] | 13.80 [12.76, 14.82] | -0.13 | 13.40 [12.30, 14.47] | 14.00 [12.80, 14.90] | 0.00 | N/A | N/A | #VALUE! | 13.59 (1.61) | #VALUE! | #VALUE! |
| Missing; n (%) | 21,318 (82.9%) | 11,308 (76.1%) | 0.17 | 32,011 (99.1%) | 17,463 (98.4%) | 0.06 | N/A | N/A | #VALUE! | 53,329 (92.0%) | 28,771 (88.2%) | 0.13 |
| Lab result number- Serum sodium mean (only > 90 | . , | . , | | | . , | | | | | . , | | |
| and < 190 included) | 5,895 | 4,582 | | 341 | 365 | | N/A | N/A | | 6,236 | 4,947 | |
| mean (sd) | 140.05 (2.96) | 140.27 (2.94) | -0.07 | 139.62 (3.02) | 139.71 (2.77) | -0.03 | N/A | N/A | #VALUE! | 140.03 (2.96) | 140.23 (2.93) | -0.07 |
| median [IQR] | 140.00 [138.50, 142.00] | 140.50 [139.00, 142.00] | -0.17 | 140.00 [138.00, 141.00] | 140.00 [138.00, 142.00] | 0.00 | N/A | N/A | #VALUE! | 140.00 (2.96) | 140.46 (2.93) | -0.16 |
| Missing; n (%) | 19,806 (77.1%) | 10,287 (69.2%) | 0.18 | 31,954 (98.9%) | 17,383 (97.9%) | 0.08 | N/A | N/A | #VALUE! | 51,760 (89.2%) | 27,670 (84.8%) | 0.13 |
| Lab result number- Albumin mean (only >0 and <=10 | | | | | | | | | | | | |
| included) | 5,206 | 4,061 | | 263 | 286 | | N/A | N/A | | 5,469 | 4,347 | |
| mean (sd) | 4.14 (0.32) | 4.19 (0.33) | -0.15 | 4.01 (0.70) | 4.09 (0.59) | -0.12 | N/A | N/A | #VALUE! | 4.13 (0.35) | 4.18 (0.35) | -0.14 |
| median [IQR] | 4.15 [3.95, 4.35] | 4.20 [4.00, 4.40] | -0.15 | 4.10 [3.83, 4.35] | 4.20 [4.00, 4.40] | -0.15 | N/A | N/A | #VALUE! | 4.15 (0.35) | 4.20 (0.35) | -0.14 |
| Missing; n (%) | 20,495 (79.7%) | 10,808 (72.7%) | 0.16 | 32,032 (99.2%) | 17,462 (98.4%) | 0.07 | N/A | N/A | #VALUE! | 52,527 (90.6%) | 28,270 (86.7%) | 0.12 |
| Lab result number-Glucose (fasting or random) mean | , , | | | , | | | • | • | | / | | |
| (only 10-1000 included) | 5,816 | 4,563 | | 336 | 362 | | N/A | N/A | | 6,152 | 4,925 | |
| mean (sd) | 113.88 (37.92) | 112.94 (36.12) | 0.03 | 128.18 (55.83) | 129.74 (45.68) | -0.03 | N/A | N/A | #VALUE! | 114.66 (39.11) | 114.17 (36.91) | 0.01 |
| median [IQR] | 103.00 [92.00, 122.00] | 103.00 [93.00, 121.00] | 0.00 | 114.00 [97.00, 138.94] | 117.00 [100.00, 143.08] | -0.06 | N/A | N/A | #VALUE! | 103.60 (39.11) | 104.03 (36.91) | -0.01 |
| Missing; n (%) | 19,885 (77.4%) | 10,306 (69.3%) | 0.18 | 31,959 (99.0%) | 17,386 (98.0%) | 0.08 | N/A | N/A | #VALUE! | 51,844 (89.4%) | 27,692 (84.9%) | 0.13 |
| Lab result number- Potassium mean (only 1-7 | | , | | ,, | , , | | • | • | | . , | , | |
| included) | 6,075 | 4,778 | | 402 | 377 | | N/A | N/A | | 6,477 | 5,155 | |

| mean (sd) | 4.35 (0.44) | 4.38 (0.44) | -0.07 | 4.33 (0.42) | 4.34 (0.41) | -0.02 | N/A | N/A | #VALUE! | 4.35 (0.44) | 4.38 (0.44) | -0.07 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| median [IQR] | 4.30 [4.10, 4.60] | 4.40 [4.10, 4.65] | -0.23 | 4.30 [4.10, 4.60] | 4.30 [4.10, 4.60] | 0.00 | N/A | N/A | #VALUE! | 4.30 (0.44) | 4.39 (0.44) | -0.20 |
| Missing; n (%) | 19,626 (76.4%) | 10,091 (67.9%) | 0.19 | 31,893 (98.8%) | 17,371 (97.9%) | 0.07 | N/A | N/A | #VALUE! | 51,519 (88.8%) | 27,462 (84.2%) | 0.13 |
| Comorbidity Scores | | | | | | | | | | | | |
| CCI (180 days)- ICD9 and ICD10 v2 | 2 27 (4 72) | 2 44 (4 74) | | 2.04 (4.67) | 2.00 (4.55) | | 2.07 (2.40) | 2 00 (2 00) | 0.04 | 2.00 (4.05) | 2.05 (4.00) | 0.00 |
| mean (sd) | 3.37 (1.73) | 3.44 (1.71) | -0.04 | 3.01 (1.67) | 3.08 (1.56) | -0.04 | 2.87 (2.10) | 2.90 (2.09) | -0.01 | 2.99 (1.95) | 3.05 (1.90) | -0.03 |
| median [IQR] | 3.00 [2.00, 4.00] | 3.00 [2.00, 5.00] | 0.00 | 3.00 [2.00, 4.00] | 3.00 [2.00, 4.00] | 0.00 | 3.00 [1.00, 4.00] | | 0.00 | 3.00 (1.95) | 3.00 (1.90) | 0.00 |
| Non-Frailty; n (%) | 13,921 (54.2%) | 8,405 (56.5%) | -0.05 | 16,295 (50.5%) | 9,068 (51.1%) | -0.01 | 2,130 (2.3%) | 887 (2.2%) | 0.01 | 32,346 (21.5%) | 18,360 (25.1%) | -0.09 |
| Frailty Score (mean): Empirical Version 365 days, v2 | 0.10 (0.05) | 0.19 (0.06) | 0.00 | 0.19 (0.05) | 0.18 (0.05) | 0.20 | 18.75 (12.79) | 47 47 (42 70) | 0.12 | 44 50 (40 02) | 9.61 (9.52) | 0.20 |
| mean (sd) | 0.19 (0.06) | | 0.00 | | | 0.20 | | 17.17 (12.78) | 0.12 | 11.59 (10.03) | 8.13 (9.52) | 0.20 |
| median [IQR]<br>Healthcare Utilization | 0.18 [0.15, 0.22] | 0.18 [0.15, 0.21] | 0.00 | 0.18 [0.15, 0.21] | 0.17 [0.15, 0.20] | 0.20 | 16.16 [9.68, 25.10] [ | 4.51 [8.15, 23.26] | 0.13 | 10.00 (10.03) | 8.13 (9.52) | 0.19 |
| Any hospitalization; n (%) | 5,289 (20.6%) | 3,814 (25.7%) | -0.12 | 7,942 (24.6%) | 5,601 (31.6%) | -0.16 | 35,792 (38.7%) | 20,776 (51.1%) | -0.25 | 49,023 (32.6%) | 30,191 (41.2%) | -0.18 |
| Any hospitalization, in (%) Any hospitalization within prior 30 days; n (%) | 3,558 (13.8%) | 2,423 (16.3%) | -0.12 | 4,737 (14.7%) | 3,876 (21.8%) | -0.18 | 21,828 (23.6%) | 13,998 (34.4%) | -0.24 | 30123 (20.0%) | 20297 (27.7%) | -0.18 |
| Any hospitalization during prior 31-180 days; n (%) | 2,003 (7.8%) | 1,604 (10.8%) | -0.10 | 3,530 (10.9%) | 1,982 (11.2%) | -0.01 | 16,767 (18.1%) | 8,551 (21.0%) | -0.07 | 22300 (14.8%) | 12137 (16.6%) | -0.05 |
| Endocrinologist Visit; n (%) | 745 (2.9%) | 496 (3.3%) | -0.02 | 1,051 (3.3%) | 737 (4.2%) | -0.01 | 4,770 (5.2%) | 2,301 (5.7%) | -0.02 | 6566 (4.4%) | 3534 (4.8%) | -0.02 |
| Endocrinologist Visit, ii (/8) Endocrinologist Visit (30 days prior); n (%) | 254 (1.0%) | 165 (1.1%) | -0.02 | 343 (1.1%) | 253 (1.4%) | -0.03 | 1,441 (1.6%) | 779 (1.9%) | -0.02 | 2038 (1.4%) | 1197 (1.6%) | -0.02 |
| Endocrinologist Visit (30 days prior); n (%) | 614 (2.4%) | 412 (2.8%) | -0.03 | 903 (2.8%) | 621 (3.5%) | -0.04 | 4,153 (4.5%) | 1,951 (4.8%) | -0.01 | 5670 (3.8%) | 2984 (4.1%) | -0.02 |
| Internal medicine/family medicine visits; n (%) | 22,697 (88.3%) | 12,893 (86.7%) | 0.05 | 25,755 (79.7%) | 14,625 (82.4%) | -0.07 | 79,393 (85.9%) | 36,147 (88.9%) | -0.09 | 127845 (85.0%) | 63665 (86.9%) | -0.05 |
| Internal medicine/family medicine visits (30 days | 22,037 (00.370) | 12,055 (00.770) | 0.03 | 23,733 (73.770) | 11,023 (021170) | 0.07 | 73,333 (03.370) | 30,117 (00.370) | 0.03 | 127013 (03.070) | 03003 (00:370) | 0.03 |
| prior) v2; n (%) | 16,026 (62.4%) | 8,775 (59.0%) | 0.07 | 16,896 (52.3%) | 10,186 (57.4%) | -0.10 | 53,989 (58.4%) | 26,439 (65.0%) | -0.14 | 86911 (57.8%) | 45400 (62.0%) | -0.09 |
| Internal medicine/family medicine visits (31 to 180 | . , , | . , , | | . , , | , | | | , | | , , | , , | |
| days prior) v2; n (%) | 20,181 (78.5%) | 11,309 (76.1%) | 0.06 | 23,468 (72.7%) | 12,754 (71.9%) | 0.02 | 70,359 (76.1%) | 31,172 (76.7%) | -0.01 | 114008 (75.8%) | 55235 (75.4%) | 0.01 |
| Cardiologist visit; n (%) | 17,320 (67.4%) | 12,047 (81.0%) | -0.31 | 17,116 (53.0%) | 11,195 (63.1%) | -0.21 | 71,688 (77.6%) | 35,047 (86.2%) | -0.22 | 106124 (70.6%) | 58289 (79.6%) | -0.21 |
| Number of Cardiologist visits (30 days prior); n (%) | 12,102 (47.1%) | 9,678 (65.1%) | -0.37 | 10,270 (31.8%) | 9,109 (51.3%) | -0.40 | 46,370 (50.2%) | 27,902 (68.6%) | -0.38 | 68742 (45.7%) | 46689 (63.7%) | -0.37 |
| Number of Cardiologist visits (31 to 180 days prior); | | | | | | | | | | | | |
| n (%) | 11,899 (46.3%) | 7,468 (50.2%) | -0.08 | 13,333 (41.3%) | 6,899 (38.9%) | 0.05 | 52,530 (56.8%) | 21,981 (54.1%) | 0.05 | 77762 (51.7%) | 36348 (49.6%) | 0.04 |
| Electrocardiogram v2; n (%) | 16,445 (64.0%) | 12,125 (81.5%) | -0.40 | 19,397 (60.1%) | 14,074 (79.3%) | -0.43 | 66,036 (71.5%) | 35,363 (87.0%) | -0.39 | 101878 (67.7%) | 61562 (84.0%) | -0.39 |
| Use of glucose test strips; n (%) | 348 (1.4%) | 227 (1.5%) | -0.01 | 334 (1.0%) | 217 (1.2%) | -0.02 | 1,863 (2.0%) | 1,006 (2.5%) | -0.03 | 2545 (1.7%) | 1450 (2.0%) | -0.02 |
| Dialysis; n (%) | 3 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| number of different/distinct medication | | | | | | | | | | | | |
| prescriptions | | | | | | | | | | | | |
| mean (sd) | 8.98 (4.25) | 9.52 (4.58) | -0.12 | 9.50 (4.46) | 9.73 (4.60) | -0.05 | 10.36 (4.52) | 11.16 (4.98) | -0.17 | 9.94 (4.46) | 10.48 (4.81) | 0.00 |
| median [IQR] | 8.00 [6.00, 11.00] | 9.00 [6.00, 12.00] | -0.23 | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 0.00 | 10.00 [7.00, 13.00] [ | 0.00 [8.00, 14.00] | 0.00 | 5.45 (5.28) | 6.43 (5.46) | 0.00 |
| Number of Hospitalizations | | | | | | | | | | | | |
| mean (sd) | 0.23 (0.50) | 0.29 (0.55) | -0.11 | 0.27 (0.50) | 0.35 (0.54) | -0.15 | 0.49 (0.72) | 0.64 (0.76) | -0.20 | 0.40 (0.64) | 0.50 (0.67) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | -1.35 | 0.00 (0.72) | 0.24 (0.74) | 0.00 |
| Number of hospital days | | | | | | | | | | | | |
| mean (sd) | 1.17 (3.39) | 1.27 (3.31) | -0.03 | 1.47 (4.58) | 1.48 (3.36) | 0.00 | 2.99 (6.48) | 3.45 (6.68) | -0.07 | 2.35 (5.68) | 2.53 (5.45) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 [0.00, 4.00] | 2.00 [0.00, 5.00] | -0.30 | 0.00 (6.38) | 0.48 (5.77) | 0.00 |
| Number of Emergency Department (ED) visits v3 | 0.50(4.20) | 0.04 (4.47) | 0.45 | 0.40 (4.70) | 0.50 (0.05) | 0.40 | 4 00 (4 75) | 4 20 (4 00) | 0.46 | 0.05 (4.55) | 4 40 (4 00) | |
| mean (sd) | 0.60 (1.20) | 0.81 (1.47) | -0.16 | 0.43 (1.72) | 0.69 (2.35) | -0.13 | 1.08 (1.75) | 1.38 (1.98) | -0.16 | 0.86 (1.66) | 1.10 (1.99) | 0.00 |
| median [IQR]<br>Number of Office visits | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | -0.54 | 0.00 (1.99) | 0.24 (2.38) | 0.00 |
| | F FC (4.20) | F 72 (2.00) | 0.04 | C 45 (5 00) | F 00 /4 44) | 0.13 | 12.00 (12.00) | 42.04/42.20) | 0.00 | 40.02 (44.20) | 40.22 (40.20) | 0.00 |
| mean (sd) | 5.56 (4.39)<br>5.00 [2.00, 8.00] | 5.73 (3.98)<br>5.00 [3.00, 8.00] | -0.04<br>0.00 | 6.45 (5.08) | 5.89 (4.11) | 0.12<br>0.00 | 13.98 (13.90)<br>10.00 [5.00, 19.00] I | 13.94 (13.20) | 0.00<br>-0.07 | 10.92 (11.29)<br>4.08 (11.74) | 10.32 (10.20)<br>4.89 (10.45) | 0.00<br>0.00 |
| median [IQR]<br>Number of Endocrinologist visits | 5.00 [2.00, 8.00] | 5.00 [3.00, 8.00] | 0.00 | 5.00 [3.00, 9.00] | 5.00 [3.00, 8.00] | 0.00 | 10.00 [5.00, 19.00] | 1.00 [5.00, 18.00] | -0.07 | 4.08 (11.74) | 4.89 (10.45) | 0.00 |
| mean (sd) | 0.11 (1.11) | 0.13 (1.11) | -0.02 | 0.12 (1.01) | 0.16 (1.25) | -0.04 | 0.26 (1.93) | 0.27 (1.84) | -0.01 | 0.20 (1.65) | 0.21 (1.58) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | - ( - , | 0.00 | 0.00 (1.77) | 0.00 (1.73) | 0.00 |
| Number of internal medicine/family medicine visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.77) | 0.00 (1.73) | 0.00 |
| mean (sd) | 10.42 (12.51) | 9.05 (11.93) | 0.11 | 8.01 (11.59) | 7.29 (10.23) | 0.07 | 9.70 (11.61) | 9.63 (10.82) | 0.01 | 9.46 (11.76) | 8.95 (10.92) | 0.00 |
| median [IQR] | 7.00 [2.00, 14.00] | 6.00 [2.00, 12.00] | 0.08 | 4.00 [1.00, 10.00] | 4.00 [1.00, 9.00] | 0.00 | 6.00 [2.00, 13.00] | | -0.09 | 3.34 (13.86) | 3.88 (12.32) | 0.00 |
| Number of Cardiologist visits | 7.00 [2.00, 2.1.00] | 0.00 (2.00, 12.00) | 0.00 | 1.00 [1.00, 10.00] | 1.00 [2.00, 5.00] | 0.00 | 0.00 (2.00, 25.00) | 7.00 [5.00, 15.00] | 0.03 | 3.3 (13.00) | 3.00 (12.32) | 0.00 |
| mean (sd) | 4.23 (5.80) | 5.24 (5.92) | -0.17 | 3.14 (5.45) | 3.46 (4.82) | -0.06 | 5.69 (7.71) | 6.37 (7.97) | -0.09 | 4.89 (6.97) | 5.44 (6.93) | 0.00 |
| median [IQR] | 2.00 [0.00, 6.00] | 4.00 [1.00, 7.00] | -0.34 | 1.00 [0.00, 4.00] | 2.00 [0.00, 5.00] | -0.19 | 3.00 [1.00, 8.00] | | -0.13 | 1.20 (7.78) | 2.27 (7.43) | 0.00 |
| Number electrocardiograms received v2 | | , | | | | | | | | - ( - , | , -, | |
| mean (sd) | 1.62 (2.18) | 2.42 (2.58) | -0.33 | 1.36 (1.88) | 1.99 (2.05) | -0.32 | 2.05 (2.35) | 2.85 (2.57) | -0.32 | 1.83 (2.23) | 2.55 (2.46) | 0.00 |
| median [IQR] | 1.00 [0.00, 2.00] | 2.00 [1.00, 3.00] | -0.42 | 1.00 [0.00, 2.00] | 1.00 [1.00, 3.00] | 0.00 | 1.00 [0.00, 3.00] | | -0.41 | 0.60 (2.53) | 1.13 (2.71) | 0.00 |
| Number of HbA1c tests ordered | , | ,, | | | | | | | | | 7 | |
| mean (sd) | 0.46 (0.73) | 0.49 (0.73) | -0.04 | 0.21 (0.54) | 0.27 (0.59) | -0.11 | 0.57 (0.81) | 0.59 (0.82) | -0.02 | 0.47 (0.75) | 0.49 (0.75) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (0.82) | 0.00 (0.82) | 0.00 |
| Number of glucose tests ordered | | | | | | | | • | | . , | | |
| mean (sd) | 0.19 (1.94) | 0.20 (0.86) | -0.01 | 0.13 (0.81) | 0.15 (0.84) | -0.02 | 0.20 (0.94) | 0.23 (0.75) | -0.04 | 0.18 (1.15) | 0.20 (0.80) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.26) | 0.00 (0.92) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.63 (0.82) | 0.71 (0.84) | -0.10 | 0.27 (0.68) | 0.40 (0.88) | -0.17 | 0.66 (0.77) | 0.72 (0.80) | -0.08 | 0.57 (0.76) | 0.64 (0.83) | 0.00 |

| median [IQR] | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | -1.20 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 0.21 (0.87) | 0.45 (0.96) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number of creatinine tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.07 (0.39) | 0.07 (0.34) | 0.00 | 0.06 (0.36) | 0.05 (0.29) | 0.03 | 0.12 (0.49) | 0.11 (0.43) | 0.02 | 0.10 (0.45) | 0.09 (0.38) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.50) | 0.00 (0.42) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.04 (0.32) | 0.04 (0.26) | 0.00 | 0.04 (0.27) | 0.03 (0.23) | 0.04 | 0.08 (0.40) | 0.07 (0.33) | 0.03 | 0.06 (0.36) | 0.05 (0.29) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.40) | 0.00 (0.32) | 0.00 |
| Number of tests for microalbuminuria | | | | | | | | | | | | |
| mean (sd) | 0.22 (0.66) | 0.22 (0.66) | 0.00 | 0.09 (0.42) | 0.11 (0.47) | -0.04 | 0.16 (0.48) | 0.17 (0.49) | -0.02 | 0.16 (0.50) | 0.17 (0.52) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.57) | 0.00 (0.59) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | | | | | | | | | | , , | , , | |
| digit level Copy | | | | | | | | | | | | |
| mean (sd) | 5.69 (7.91) | 8.77 (9.30) | -0.36 | 2.78 (5.59) | 4.42 (6.78) | -0.26 | 9.07 (11.13) | 11.98 (12.28) | -0.25 | 7.14 (9.67) | 9.50 (10.60) | 0.00 |
| median [IQR] | 3.00 [0.00, 9.00] | 7.00 [0.00, 13.00] | -0.46 | 0.00 [0.00, 3.00] | 1.00 [0.00, 7.00] | -0.16 | 5.00 [0.00, 15.00] | 9.00 [0.00, 19.00] | -0.34 | 1.59 (10.30) | 3.84 (11.26) | 0.00 |
| For PS | | | | | | | | | | , , | , , | |
| Hemorrhagic stroke+Other cerebrovascular | | | | | | | | | | | | |
| disease+Cerebrovascular procedure (for PS); n (%) | 912 (3.5%) | 691 (4.6%) | -0.06 | 986 (3.1%) | 607 (3.4%) | -0.02 | 4,474 (4.8%) | 2,233 (5.5%) | -0.03 | 6372 (4.2%) | 3531 (4.8%) | -0.03 |
| Occurrence of creatinine tests ordered (for PS); n (%) | 1,338 (5.2%) | 824 (5.5%) | -0.01 | 1,445 (4.5%) | 732 (4.1%) | 0.02 | 8,254 (8.9%) | 3,521 (8.7%) | 0.01 | 11037 (7.3%) | 5077 (6.9%) | 0.02 |
| Occurrence of BUN tests ordered (for PS); n (%) | 824 (3.2%) | 492 (3.3%) | -0.01 | 873 (2.7%) | 479 (2.7%) | 0.00 | 5,372 (5.8%) | 2,228 (5.5%) | 0.01 | 7069 (4.7%) | 3199 (4.4%) | 0.01 |
| Occurrence of chronic renal insufficiency w/o CKD | | | | | | | | | | | | |
| (for PS) v2; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 682 (0.7%) | 243 (0.6%) | 0.01 | 682 (0.5%) | 243 (0.3%) | 0.03 |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 | 0 | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Chronic kidney disease Stage 3-6 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1,912 (2.1%) | 547 (1.3%) | 0.06 | 1912 (1.3%) | 547 (0.7%) | 0.06 |
| Bladder stones+Kidney stones (for PS); n (%) | 210 (0.8%) | 179 (1.2%) | -0.04 | 313 (1.0%) | 209 (1.2%) | -0.02 | 1,291 (1.4%) | 685 (1.7%) | -0.02 | 1814 (1.2%) | 1073 (1.5%) | -0.03 |
| Diabetes with peripheral circulatory | | | | | | | | | | | | |
| disorders+Gangrene+Osteomyelitis(for PS) v3 with | | | | | | | | | | | | |
| ICD10 Copy; n (%) | 943 (3.7%) | 452 (3.0%) | 0.04 | 939 (2.9%) | 397 (2.2%) | 0.04 | 5,228 (5.7%) | 2,132 (5.2%) | 0.02 | 7110 (4.7%) | 2981 (4.1%) | 0.03 |
| Alcohol abuse or dependence+Drug abuse or | | | | | | | | | | | | |
| dependence (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 173 (0.2%) | 139 (0.3%) | -0.02 | 173 (0.1%) | 139 (0.2%) | -0.03 |
| Diabetes with other ophthalmic | | | | | | | | | | | | |
| manifestations+Retinal detachment, vitreous | | | | | | | | | | | | |
| hemorrhage, vitrectomy+Retinal laser coagulation | | | | | | | | | | | | |
| therapy (for PS); n (%) | 115 (0.4%) | 84 (0.6%) | -0.03 | 555 (1.7%) | 220 (1.2%) | 0.04 | 1,437 (1.6%) | 593 (1.5%) | 0.01 | 2107 (1.4%) | 897 (1.2%) | 0.02 |
| Other atherosclerosis+Cardiac conduction | | | | | | | | | | | | |
| disorders+Other CVD (for PS) v2 Copy; n (%) | 10,167 (39.6%) | 6,504 (43.7%) | -0.08 | 11,709 (36.3%) | 6,953 (39.2%) | -0.06 | 37,639 (40.7%) | 18,343 (45.1%) | -0.09 | 59515 (39.6%) | 31800 (43.4%) | -0.08 |
| Previous cardiac procedure (CABG or PTCA or Stent) + | | | | | | | | | | | | |
| History of CABG or PTCA (for PS) v3; n (%) | 2,140 (8.3%) | 1,535 (10.3%) | -0.07 | 1,558 (4.8%) | 947 (5.3%) | -0.02 | 12,496 (13.5%) | 6,545 (16.1%) | -0.07 | 16194 (10.8%) | 9027 (12.3%) | -0.05 |
| Hyperthyroidism + Hypothyroidism + Other disorders | 5 404 (20 20) | 2 200 (22 20() | 0.05 | 4.5.44.(4.4.40() | 2.050 (47.20) | 0.00 | 46 704 (40 40() | C 004 (47 00() | 0.00 | 255 45 (47 70/) | 42250 (40.40() | 0.04 |
| of thyroid gland (for PS); n (%) | 5,181 (20.2%) | 3,309 (22.3%) | -0.05 | 4,641 (14.4%) | 3,058 (17.2%) | -0.08 | 16,724 (18.1%) | 6,901 (17.0%) | 0.03 | 26546 (17.7%) | 13268 (18.1%) | -0.01 |
| Delirium + Psychosis (for PS); n (%) | 679 (2.6%) | 400 (2.7%) | -0.01 | 861 (2.7%) | 369 (2.1%) | 0.04 | 4,298 (4.7%) | 2,093 (5.1%) | -0.02 | 5838 (3.9%) | 2862 (3.9%) | 0.00 |
| Any use of Meglitinides (for PS); n (%) | 56 (0.2%) | 43 (0.3%) | -0.02 | 166 (0.5%) | 80 (0.5%) | 0.00 | 460 (0.5%) | 200 (0.5%) | 0.00 | 682 (0.5%) | 323 (0.4%) | 0.01 |
| Any use of AGIs (for PS); n (%) | 24 (0.1%) | 10 (0.1%) | 0.00 | 46 (0.1%) | 12 (0.1%) | 0.00 | 139 (0.2%) | 57 (0.1%) | 0.03 | 209 (0.1%) | 79 (0.1%) | 0.00 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 3 (0.0%) | 1 (0.0%) | #DIV/0! | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 1,917 (2.1%) | 549 (1.4%) | 0.05 | 1921 (1.3%) | 550 (0.8%) | 0.05 |
| Use of thiazide- United; n (%) | 3,246 (12.6%) | 1,792 (12.1%) | 0.02 | 3,732 (11.6%) | 2,078 (11.7%) | 0.00 | 11,852 (12.8%) | 5,583 (13.7%) | -0.03 | 18830 (12.5%) | 9453 (12.9%) | -0.01 |
| Use of beta blockers; n (%) | 17,651 (68.7%) | 10,352 (69.6%) | -0.02 | 22,255 (68.9%) | 12,673 (71.4%) | -0.05 | 67,017 (72.5%) | 30,360 (74.7%) | -0.05 | 106923 (71.1%) | 53385 (72.9%) | -0.04 |
| Use of calcium channel blockers; n (%) | 9,670 (37.6%) | 6,047 (40.7%) | -0.06 | 12,176 (37.7%) | 7,379 (41.6%) | -0.08 | 37,046 (40.1%) | 18,250 (44.9%) | -0.10 | 58892 (39.2%) | 31676 (43.2%) | -0.08 |
| All antidiabetic medications except Insulin; n (%) | 6,249 (24.3%) | 3,472 (23.4%) | 0.02 | 7,734 (23.9%) | 4,459 (25.1%) | -0.03 | 26,614 (28.8%) | 12,216 (30.1%) | -0.03 | 40597 (27.0%) | 20147 (27.5%) | -0.01 |
| DM Medications - Insulin Copy; n (%) | 1,395 (5.4%) | 653 (4.4%) | 0.05 | 2,314 (7.2%) | 1,089 (6.1%) | 0.04 | 6,547 (7.1%) | 2,810 (6.9%) | 0.01 | 10256 (6.8%) | 4552 (6.2%) | 0.02 |
| Use of Low Intensity Statins; n (%) | 9,654 (37.6%) | 4,898 (32.9%) | 0.10 | 11,758 (36.4%) | 5,834 (32.9%) | 0.07 | 35,863 (38.8%) | 14,698 (36.2%) | 0.05 | 57275 (38.1%) | 25430 (34.7%) | 0.07 |
| Use of High Intensity Statins; n (%) | 5,758 (22.4%) | 4,335 (29.2%) | -0.16 | 7,351 (22.8%) | 4,764 (26.8%) | -0.09 | 21,260 (23.0%) | 11,124 (27.4%) | -0.10 | 34369 (22.9%) | 20223 (27.6%) | -0.11 |
| Malignant hypertension; n (%) | 1,402 (5.5%) | 605 (4.1%) | 0.07 | 14,434 (44.7%) | 7,875 (44.4%) | 0.01 | 24,773 (26.8%) | 11,920 (29.3%) | -0.06 | 40609 (27.0%) | 20400 (27.8%) | -0.02 |
| Cardiovascular stress test; n (%) | 119 (0.5%) | 72 (0.5%) | 0.00 | 232 (0.7%) | 126 (0.7%) | 0.00 | 901 (1.0%) | 384 (0.9%) | 0.01 | 1252 (0.8%) | 582 (0.8%) | 0.00 |
| Echocardiogram; n (%) | 9,046 (35.2%) | 7,241 (48.7%) | -0.28 | 11,883 (36.8%) | 9,419 (53.1%) | -0.33 | 41,768 (45.2%) | 25,031 (61.6%) | -0.33 | 62697 (41.7%) | 41691 (56.9%) | -0.31 |
| Number of BNP tests | | | | | | | | | | | | |
| mean (sd) | 0.13 (0.49) | 0.16 (0.53) | -0.06 | 0.08 (0.45) | 0.10 (0.40) | -0.05 | 0.24 (0.66) | 0.27 (0.66) | -0.05 | 0.19 (0.59) | 0.21 (0.58) | -0.03 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.66) | 0.00 (0.62) | 0.00 |
| Number of Cardiac biomarkers tests (tropnin, CK-MBs, Myo | oglobin CDV) | | | | | | | | | | | |
| mean (sd) | 0.37 (1.26) | 0.57 (1.61) | -0.14 | 0.27 (1.17) | 0.47 (1.53) | -0.15 | 0.31 (0.65) | 0.42 (0.75) | -0.16 | 0.31 (0.91) | 0.46 (1.19) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.14 | 0.27 (1.17) | 0.47 (1.53) | 0.00 | 0.00 [0.00, 0.00] | | 0.00 | 0.31 (0.91) | 0.46 (1.19) | 0.00 |
| incular [/Qh] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.17) | 0.00 (1.46) | 0.00 |
| Number of Ambulatory Blood pressure monitoring tests | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.03) | 0.00 (0.03) | 0.00 | 0.00 (0.04) | 0.00 (0.05) | 0.00 | 0.00 (0.03) | 0.00 (0.04) | 0.00 | 0.00 (0.03) | 0.00 (0.04) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.04) | 0.00 (0.05) | 0.00 |
| N of days on antihypertensive medications during baseline | 2 | | | | | | 0 | 0 | | | | |

| mean (sd) | 138.54 (63.34) | 137.54 (63.50) | 0.02 | 140.38 (63.02) | 137.96 (64.23) | 0.04 | 147.39 (56.03) | 147.97 (55.26) | -0.01 | 144.37 (58.88) | 143.43 (59.26) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| median [IQR] | 174.00 [120.00, 181.00] | 173.00 [116.00, 181.00] | 0.02 | 177.00 [126.00, 181.00] | 174.00 [119.00, 181.00] | 0.05 | 177.00 [144.00, 181.00] | 0 [145.00, 181.00] | 0.02 | 105.75 (71.09) | 119.89 (69.29) | 0.00 |
| N of days in database anytime prior | | | | | | | 0 | 0 | | | | |
| mean (sd) | 1,959.27 (1,297.23) | 2,058.84 (1,433.06) | -0.07 | 2,420.20 (1,291.48) | 2,541.09 (1,409.03) | -0.09 | 953 45 (634 65) | 823.51 (522.94) | 0.22 | 1440.28 (945.08) | 1490.25 (1024.40) | 0.00 |
| ·····cair (sa) | 1,776.00 [827.00, | 1,720.00 [832.00, | 0.07 | 2,120.20 (1,231.10) | 2,3 (2.03 (1, 103.03) | 0.03 | 333.13 (031.03) | 023.31 (322.31) | 0.22 | 1110.20 (313.00) | 1130.23 (1021110) | 0.00 |
| modian [IOR] | 2,836.00] | | 0.045 | 00 [1 353 00 3 470 00] | .1.00 [1,278.00, 3,708.75] | 0.0471 | 16.00 [478.00, 1,286.00] ( | 0 [400 00 061 00] | 0.09 | 1008.23 (1248.91) | 1117 65 (1202 20) | 0.00 |
| median [IQR] | 2,836.00] | 3,097.00] | 0.04 30 | 3.00 [1,232.00, 3,479.00] | .1.00 [1,278.00, 3,708.73] | 0.047 | 16.00 [478.00, 1,286.00] | 0 [490.00, 961.00] | 0.09 | 1008.23 (1248.91) | 1117.65 (1292.30) | 0.00 |
| | | | | | | | _ | _ | | | | |
| Mean Copay for per prescription cost (charges in | | | | | | | 0 | 0 | | | | |
| mean (sd) | 28.47 (41.39) | 29.22 (39.66) | -0.02 | 19.16 (19.36) | 18.88 (20.59) | 0.01 | | 117.02 (103.79) | 0.04 | 83.63 (91.22) | 75.43 (79.99) | 0.00 |
| median [IQR] | 17.87 [8.00, 34.79] | 18.85 [7.82, 36.19] | -0.02 | 15.00 [7.40, 25.46] | 14.01 [6.55, 25.02] | 0.05 | 99.09 [70.50, 141.51] | 40 [68.67, 135.00] | 0.03 | 27.55 (92.04) | 30.33 (80.82) | 0.00 |
| Missing; n (%) | 697 (2.7%) | 299 (2.0%) | 0.05 | 831 (2.6%) | 341 (1.9%) | 0.05 | 1,655 (1.8%) | 476 (1.2%) | 0.05 | 3183 (2.1%) | 1116 (1.5%) | 0.05 |
| Colonoscopy; n (%) | 640 (2.5%) | 432 (2.9%) | -0.02 | 868 (2.7%) | 644 (3.6%) | -0.05 | 2,623 (2.8%) | 1,364 (3.4%) | -0.03 | 4131 (2.7%) | 2440 (3.3%) | -0.04 |
| Fecal occult blood (FOB) test; n (%) | 754 (2.9%) | 493 (3.3%) | -0.02 | 598 (1.9%) | 404 (2.3%) | -0.03 | 2,177 (2.4%) | 1,058 (2.6%) | -0.01 | 3529 (2.3%) | 1955 (2.7%) | -0.03 |
| Flu vaccine; n (%) | 5,240 (20.4%) | 2,802 (18.8%) | 0.04 | 4,338 (13.4%) | 2,190 (12.3%) | 0.03 | 30,438 (32.9%) | 13,288 (32.7%) | 0.00 | 40016 (26.6%) | 18280 (24.9%) | 0.04 |
| Mammogram; n (%) | 2,062 (8.0%) | 1,374 (9.2%) | -0.04 | 1,495 (4.6%) | 1,054 (5.9%) | -0.06 | 8,045 (8.7%) | 3,965 (9.8%) | -0.04 | 11602 (7.7%) | 6393 (8.7%) | -0.04 |
| Pap smear; n (%) | 305 (1.2%) | 250 (1.7%) | -0.04 | 405 (1.3%) | 358 (2.0%) | -0.05 | 1,287 (1.4%) | 814 (2.0%) | -0.05 | 1997 (1.3%) | 1422 (1.9%) | -0.05 |
| Pneumonia vaccine; n (%) | 3,034 (11.8%) | 2,543 (17.1%) | -0.15 | 1,406 (4.4%) | 1,266 (7.1%) | -0.12 | 14,621 (15.8%) | 8,703 (21.4%) | -0.14 | 19061 (12.7%) | 12512 (17.1%) | -0.12 |
| PSA test or Prostate exam for DRE; n (%) | 2,967 (11.5%) | 2,054 (13.8%) | -0.07 | 1,970 (6.1%) | 1,552 (8.7%) | -0.10 | 9,178 (9.9%) | 4,445 (10.9%) | -0.03 | 14115 (9.4%) | 8051 (11.0%) | -0.05 |
| Bone mineral density; n (%) | 805 (3.1%) | 532 (3.6%) | -0.03 | 452 (1.4%) | 276 (1.6%) | -0.02 | 3,027 (3.3%) | 1,480 (3.6%) | -0.02 | 4284 (2.8%) | 2288 (3.1%) | -0.02 |
| Use of Sympatomimetic agents; n (%) | 51 (0.2%) | 60 (0.4%) | -0.04 | 104 (0.3%) | 95 (0.5%) | -0.03 | 205 (0.2%) | 119 (0.3%) | -0.02 | 360 (0.2%) | 274 (0.4%) | -0.04 |
| Use of CNS stimulants; n (%) | 48 (0.2%) | 45 (0.3%) | -0.02 | 111 (0.3%) | 93 (0.5%) | -0.03 | 163 (0.2%) | 109 (0.3%) | -0.02 | 322 (0.2%) | 247 (0.3%) | -0.02 |
| Use of estrogens, progestins, androgens; n (%) | 559 (2.2%) | 471 (3.2%) | -0.06 | 1,035 (3.2%) | 806 (4.5%) | -0.07 | 2,155 (2.3%) | 1,280 (3.1%) | -0.05 | 3749 (2.5%) | 2557 (3.5%) | -0.06 |
| Use of Angiogenesis inhibitors; n (%) | 6 (0.0%) | , , | #DIV/0! | 10 (0.0%) | 5 (0.0%) | #DIV/0! | 24 (0.0%) | 14 (0.0%) | #DIV/0! | 40 (0.0%) | 23 (0.0%) | #DIV/0! |
| Use of Oral Immunosuppressants; n (%) | 5 (0.0%) | 1 (0.0%) | #DIV/0! | 21 (0.1%) | 7 (0.0%) | 0.04 | 24 (0.0%) | ** | #VALUE! | 50 (0.0%) | #VALUE! | #VALUE! |
| | | | | | | | | 44 (0.00() | | | | |
| Use of fondaparinux or Bivalirudin; n (%) | 13 (0.1%) | 1 (0.0%) | 0.04 | 14 (0.0%) | 3 (0.0%) | #DIV/0! | 43 (0.0%) | 11 (0.0%) | #DIV/0! | 70 (0.0%) | 15 (0.0%) | #DIV/0! |
| Use of other direct thrombin inhibitors (lepirudi | | | | | | | | | | | | 4 |
| desirudin, argatroban); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of Ticagrelor ON CED; n (%) | 18 (0.1%) | 40 (0.3%) | -0.04 | 29 (0.1%) | 29 (0.2%) | -0.03 | 30 (0.0%) | 19 (0.0%) | #DIV/0! | 77 (0.1%) | 88 (0.1%) | 0.00 |
| Use of Ticagrelor; n (%) | 33 (0.1%) | 68 (0.5%) | -0.07 | 38 (0.1%) | 48 (0.3%) | -0.04 | 208 (0.2%) | 143 (0.4%) | -0.04 | 279 (0.2%) | 259 (0.4%) | -0.04 |
| Number of D-dimer tests | | | | | | | | | | | | |
| mean (sd) | 0.02 (0.17) | 0.03 (0.21) | -0.05 | 0.01 (0.13) | 0.03 (0.20) | -0.12 | 0.03 (0.19) | 0.05 (0.23) | -0.09 | 0.02 (0.18) | 0.04 (0.22) | 0.00 |
| median [IQR] | 0.00,00.0,0.00 | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.19) | 0.00 (0.25) | 0.00 |
| Numbe of CRP, high-sensitivity CRP tests | (,, | (,) | | (,, | () | | (,, | (,, | | () | **** (**=*) | |
| = | 0.05 (0.33) | 0.07 (0.36) | -0.06 | 0.03 (0.33) | 0.04 (0.37) | -0.04 | 0.08 (0.42) | 0.10 (0.47) | -0.04 | 0.06 (0.37) | 0.09 (0.41) | 0.00 |
| mean (sd) | , , | , , | | 0.03 (0.23) | 0.04 (0.27) | | , , | , , | | 0.06 (0.37) | 0.08 (0.41) | |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.40) | 0.00 (0.44) | 0.00 |
| Number of PT or aPTTt tests | | | | | | | | | | | | |
| mean (sd) | 2.81 (4.00) | 0.46 (1.30) | 0.79 | 2.00 (3.43) | 0.37 (1.15) | 0.64 | 3.70 (4.84) | 0.42 (1.13) | 0.93 | 3.18 (4.43) | 0.42 (1.17) | 0.01 |
| median [IQR] | 1.00 [0.00, 5.00] | 0.00 [0.00, 0.00] | 0.34 | 0.00 [0.00, 3.00] | 0.00 [0.00, 0.00] | 0.00 | 1.00 [0.00, 6.00] | 0.00 [0.00, 1.00] | 0.28 | 0.39 (4.94) | 0.00 (1.34) | 0.00 |
| Number of Bleeding time tests | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.01) | 0.00 (0.00) | 0.00 | 0.00 (0.00) | 0.00 (0.02) | 0.00 | 0.00 (0.01) | 0.00 (0.01) | 0.00 | 0.00 (0.01) | 0.00 (0.01) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.01) | 0.00 (0.02) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | | | | | | | | | | , | , | |
| mean (sd) | 3.32 (0.71) | 3.41 (0.80) | -0.12 | 3.23 (0.72) | 3.24 (0.80) | -0.01 | 3.49 (0.71) | 3.58 (0.74) | -0.12 | 3.41 (0.71) | 3.46 (0.77) | 0.00 |
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | | 3.00 [3.00, 4.00] | 0.00 | 1.80 (0.85) | 2.06 (0.89) | 0.00 |
| • • • | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 1.80 (0.85) | 2.06 (0.89) | 0.00 |
| N of Generic name drugs | | | | | | | | | | | | |
| mean (sd) | 18.50 (14.88) | 18.50 (15.49) | 0.00 | 14.58 (9.95) | 14.60 (10.87) | 0.00 | 19.40 (13.61) | | -0.07 | 18.21 (13.15) | 18.63 (14.47) | 0.00 |
| median [IQR] | 15.00 [9.00, 23.00] | 15.00 [8.00, 24.00] | 0.00 | 13.00 [8.00, 19.00] | 12.00 [7.00, 19.00] | 0.10 | 16.00 [10.00, 25.00] 7 | 7.00 [10.00, 26.00] | -0.07 | 8.79 (14.58) | 10.07 (15.70) | 0.00 |
| N of Brand name drugs | | | | | | | | | | | | |
| mean (sd) | 3.32 (4.93) | 4.72 (5.32) | -0.27 | 4.08 (4.53) | 5.12 (4.82) | -0.22 | 3.85 (5.03) | 5.57 (6.03) | -0.31 | 3.81 (4.91) | 5.29 (5.62) | 0.00 |
| median [IQR] | 2.00 [0.00, 5.00] | 3.00 [1.00, 6.00] | -0.19 | 3.00 [1.00, 6.00] | 4.00 [2.00, 7.00] | -0.21 | 2.00 [0.00, 6.00] | 4.00 [2.00, 7.00] | -0.36 | 1.42 (5.68) | 2.55 (6.23) | 0.00 |
| Use of clopidogrel; n (%) | 2,022 (7.9%) | 1,719 (11.6%) | -0.12 | 2,811 (8.7%) | 2,115 (11.9%) | -0.11 | 9,421 (10.2%) | 5,719 (14.1%) | -0.12 | 14254 (9.5%) | 9553 (13.0%) | -0.11 |
| Systemic embolism; n (%) | 223 (0.9%) | 121 (0.8%) | 0.01 | 237 (0.7%) | 128 (0.7%) | 0.00 | 1,013 (1.1%) | 386 (0.9%) | 0.02 | 1473 (1.0%) | 635 (0.9%) | 0.01 |
| DVT; n (%) | 93 (0.4%) | 40 (0.3%) | 0.02 | 90 (0.3%) | 33 (0.2%) | 0.02 | 1,966 (2.1%) | 738 (1.8%) | 0.02 | 2149 (1.4%) | 811 (1.1%) | 0.03 |
| PE; n (%) | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 481 (0.5%) | | 0.00 | 482 (0.3%) | 187 (0.3%) | 0.00 |
| | | 1 (0.0%) | #DIV/U! | 0 (0.0%) | 0 (0.0%) | #010/01 | 461 (0.5%) | 186 (0.5%) | 0.00 | 462 (0.5%) | 107 (0.5%) | 0.00 |
| Diabetes: 1 inpatient or 2 outpatient claims with | | 4.070 (22.50() | 0.05 | 40.555 (00.70) | 5 505 (22 00) | 0.04 | 44 545 (45 00/) | 40.250 (44.00() | 0.00 | 54244 (40.00() | 20024 (20 50() | 0.00 |
| 183 days ; n (%) | 9,210 (35.8%) | 4,979 (33.5%) | 0.05 | 10,556 (32.7%) | 5,685 (32.0%) | 0.01 | 41,545 (45.0%) | 18,260 (44.9%) | 0.00 | 61311 (40.8%) | 28924 (39.5%) | 0.03 |
| Intracranial or retroperitoneal hemorrhage: 1 | | | | | | | | | | | | |
| inpatient or 2 outpatient claims within 183 days | | | | | | | | | | | | |
| (%) | 42 (0.2%) | 20 (0.1%) | 0.03 | 72 (0.2%) | 20 (0.1%) | 0.03 | 326 (0.4%) | 114 (0.3%) | 0.02 | 440 (0.3%) | 154 (0.2%) | 0.02 |
| Peptic Ulcer Disease; n (%) | 3,489 (13.6%) | 2,703 (18.2%) | -0.13 | 2,889 (8.9%) | 2,207 (12.4%) | -0.11 | 16,513 (17.9%) | 9,656 (23.8%) | -0.15 | 22891 (15.2%) | 14566 (19.9%) | -0.12 |
| Upper GI bleed; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 86 (0.1%) | 31 (0.1%) | 0.00 | 86 (0.1%) | 31 (0.0%) | 0.04 |
| Lower/unspecified GI bleed; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1,049 (1.1%) | 509 (1.3%) | -0.02 | 1049 (0.7%) | 509 (0.7%) | 0.00 |
| Urogenital bleed; n (%) | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1,725 (1.9%) | 729 (1.8%) | 0.01 | 1725 (1.1%) | 730 (1.0%) | 0.01 |
| Other bleeds; n (%) | 4 (0.0%) | 3 (0.0%) | #DIV/0! | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 969 (1.0%) | 399 (1.0%) | 0.00 | 973 (0.6%) | 403 (0.6%) | 0.00 |
| Prior cancer; n (%) | 2,927 (11.4%) | 2,127 (14.3%) | -0.09 | 3,033 (9.4%) | 1,750 (9.9%) | -0.02 | 11,109 (12.0%) | 5,640 (13.9%) | -0.06 | 17069 (11.3%) | 9517 (13.0%) | -0.05 |
| Aspirin; n (%) | 139 (0.5%) | 154 (1.0%) | -0.06 | 357 (1.1%) | 314 (1.8%) | -0.06 | 418 (0.5%) | 266 (0.7%) | -0.03 | 914 (0.6%) | 734 (1.0%) | -0.04 |

| / ! / | 72 (0.20() | 55 (0.40() | 0.00 | 450 (0.50() | 440 (0.70() | 0.00 | 274 (0.40() | 227 (2.50() | 0.00 | 505 (0.40() | 440 (0.50() | 0.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Aspirin/dipyridamole; n (%) | 73 (0.3%) | 55 (0.4%) | -0.02 | 159 (0.5%) | 118 (0.7%) | -0.03 | 374 (0.4%) | 237 (0.6%) | -0.03 | 606 (0.4%) | 410 (0.6%) | -0.03 |
| Other antiplatelet agents; n (%) | 151 (0.6%) | 69 (0.5%) | 0.01 | 182 (0.6%) | 103 (0.6%) | 0.00 | 601 (0.7%) | 289 (0.7%) | 0.00 | 934 (0.6%) | 461 (0.6%) | 0.00 |
| PGP inhibitors; n (%) | 10,770 (41.9%) | 6,482 (43.6%) | -0.03 | 14,437 (44.7%) | 8,199 (46.2%) | -0.03 | 44,650 (48.3%) | 20,953 (51.5%) | -0.06 | 69857 (46.4%) | 35634 (48.6%) | -0.04 |
| Other gastroprotective agents; n (%) | 182 (0.7%) | 140 (0.9%) | -0.02 | 301 (0.9%) | 204 (1.1%) | -0.02 | 1,082 (1.2%) | 671 (1.7%) | -0.04 | 1565 (1.0%) | 1015 (1.4%) | -0.04 |
| Number of lipid tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.63 (0.82) | 0.71 (0.84) | -0.10 | 0.27 (0.68) | 0.40 (0.88) | -0.17 | 0.69 (0.83) | 0.76 (0.89) | -0.08 | 0.59 (0.80) | 0.66 (0.88) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | -1.20 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 0.21 (0.91) | 0.45 (1.01) | 0.00 |
| Proton pump inhibitor; n (%) | 4,768 (18.6%) | 3,236 (21.8%) | -0.08 | 6,352 (19.7%) | 3,979 (22.4%) | -0.07 | 23,264 (25.2%) | 11,663 (28.7%) | -0.08 | 34384 (22.9%) | 18878 (25.8%) | -0.07 |
| H2 receptor antagonist; n (%) | 1,060 (4.1%) | 632 (4.3%) | -0.01 | 1,125 (3.5%) | 684 (3.9%) | -0.02 | 5,503 (6.0%) | 2,836 (7.0%) | -0.04 | 7688 (5.1%) | 4152 (5.7%) | -0.03 |
| Vitamin K therapy; n (%) | 20 (0.1%) | 4 (0.0%) | 0.04 | 57 (0.2%) | 4 (0.0%) | 0.06 | 119 (0.1%) | ** | #VALUE! | 196 (0.1%) | #VALUE! | #VALUE! |
| Number of neurologist visits | | | | | | | | | | | | |
| mean (sd) | 0.29 (1.48) | 0.36 (1.49) | -0.05 | 0.23 (1.34) | 0.27 (1.34) | -0.03 | 0.49 (2.00) | 0.54 (2.01) | -0.02 | 0.40 (1.79) | 0.44 (1.77) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.98) | 0.00 (1.92) | 0.00 |
| Number of INR (prothrombin) tests ordered | | | | | | | | | | | | |
| mean (sd) | 2.68 (3.90) | 0.29 (0.92) | 0.84 | 1.90 (3.33) | 0.23 (0.81) | 0.69 | 3.68 (4.80) | 0.39 (1.09) | 0.95 | 3.13 (4.37) | 0.33 (0.99) | 0.01 |
| median [IQR] | 1.00 [0.00, 5.00] | 0.00 [0.00, 0.00] | 0.35 | 0.00 [0.00, 2.00] | 0.00 [0.00, 0.00] | 0.00 | 1.00 [0.00, 6.00] | , , | 0.29 | 0.39 (4.85) | 0.00 (1.09) | 0.00 |
| Treating prescriber - Cardiologist; n (%) | 12,149 (47.3%) | 9,745 (65.5%) | -0.37 | 12,028 (37.2%) | 10,681 (60.2%) | -0.47 | 46,370 (50.2%) | 27,902 (68.6%) | -0.38 | 70547 (46.9%) | 48328 (66.0%) | -0.39 |
| Treating prescriber - Primary Care Physician; n (%) | 16,835 (65.5%) | 9,464 (63.6%) | 0.04 | 9,639 (29.8%) | 5,942 (33.5%) | -0.08 | 25,268 (27,3%) | 12.084 (29.7%) | -0.05 | 51742 (34.4%) | 27490 (37.5%) | -0.06 |
| Treating prescriber - Other; n (%) | 21,098 (82.1%) | 12,821 (86.2%) | -0.11 | 24,503 (75.9%) | 14,433 (81.3%) | -0.13 | 77,468 (83.8%) | 36,185 (89.0%) | -0.15 | 123069 (81.8%) | 63439 (86.6%) | -0.13 |
| Alpha blockers; n (%) | 3,114 (12.1%) | 1,816 (12.2%) | 0.00 | 4,170 (12.9%) | 2,035 (11.5%) | 0.04 | 11,524 (12.5%) | 5,009 (12.3%) | 0.01 | 18808 (12.5%) | 8860 (12.1%) | 0.01 |
| CHADS2 score, 180 days, V | 3,111(1211/0) | 1,010 (12.270) | 0.00 | 1,170 (12.570) | 2,000 (11.070) | 0.01 | 11,52 (12.5%) | 3,003 (12.570) | 0.01 | 10000 (12.570) | 0000 (12.170) | 0.01 |
| mean (sd) | 2.22 (1.17) | 1.98 (1.19) | 0.20 | 2.23 (1.18) | 2.05 (1.20) | 0.15 | 3.80 (1.61) | 3.62 (1.65) | 0.11 | 3.19 (1.46) | 2.91 (1.47) | 0.00 |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.00 | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.00 | | 3.00 [2.00, 5.00] | 0.61 | 1.63 (1.64) | 1.62 (1.61) | 0.00 |
| Use of Prasugrel; n (%) | 43 (0.2%) | | -0.04 | 69 (0.2%) | 88 (0.5%) | -0.05 | 4.00 [5.00, 5.00] | 3.00 [2.00, 3.00] | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Use of Loop Diuretics+other diuretics+other | 43 (0.2%) | 58 (0.4%) | -0.04 | 69 (0.2%) | 88 (0.5%) | -0.05 | | | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| hypertension drugs; n (%) | 9,459 (36.8%) | 4,643 (31.2%) | 0.12 | 12,825 (39.7%) | 5,131 (28.9%) | 0.23 | 45,778 (49.5%) | 17,784 (43.7%) | 0.12 | 68062 (45.3%) | 27558 (37.6%) | 0.16 |
| - · | 9,459 (50.6%) | 4,043 (31.2%) | 0.12 | 12,023 (39.7%) | 3,131 (20.9%) | 0.23 | 43,776 (49.3%) | 17,764 (43.7%) | 0.12 | 00002 (43.3%) | 2/336 (37.0%) | 0.16 |
| Commercial vs Medicare Advantage- Business Type Code - CORRECT ONE - OPTUM | | | | | | | | | | | | |
| Commercial: n (%) | 3,292 (12.8%) | 3244 (21.8%) | -0.24 | 27,877 (86.3%) | 13,057 (73.6%) | 0.32 | | | #VALUE! | 31,169 (53.7%) | 16,301 (50.0%) | 0.07 |
| | | , , | | | | | - | - | | . , , | | |
| Medicare Advantage; n (%) | 22,409 (87.2%) | 11625 (78.2%) | 0.24 | 4,418 (13.7%) | 4,691 (26.4%) | -0.32 | - | - | #VALUE! | 26,827 (46.3%) | 16,316 (50.0%) | -0.07 |
| Commercial vs Medicare Advantage- Business Type<br>Code | | | | | | | | | | | | |
| | 2 202 (42 00/) | 2 244 (24 20() | | | | | | | | 2 202 (42 20) | 2 244 (24 20() | 0.24 |
| COM = COMMERCIAL; n (%) | 3,292 (12.8%) | 3,244 (21.8%) | -0.24 | - | - | | - | - | #VALUE! | 3,292 (12.8%) | 3,244 (21.8%) | -0.24 |
| MCR = MEDICARE; n (%) | 22,409 (87.2%) | 11,625 (78.2%) | 0.24 | - | - | | - | - | #VALUE! | 22,409 (87.2%) | 11,625 (78.2%) | 0.24 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added in 2015); n | | | 4 | | | | | | | | | 4 |
| (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data Type | | | | | | | | | | | | |
| 1 - Fee For Service; n (%) | - | = | | 3,872 (12.0%) | 4,189 (23.6%) | -0.31 | - | = | | 3,872 (12.0%) | 4,189 (23.6%) | -0.31 |
| 2 - Encounter; n (%) | - | - | | 546 (1.7%) | 502 (2.8%) | -0.07 | - | - | | 546 (1.7%) | 502 (2.8%) | -0.07 |
| 3 - Medicare; n (%) | - | - | | 25,005 (77.4%) | 12,039 (67.8%) | 0.22 | - | - | | 25,005 (77.4%) | 12,039 (67.8%) | 0.22 |
| 4 - Medicare Encounter; n (%) | - | - | | 2,872 (8.9%) | 1,018 (5.7%) | 0.12 | - | - | | 2,872 (8.9%) | 1,018 (5.7%) | 0.12 |
| Metropolitan Statistical Area - Urban (any MSA) vs | | | | | | | | | | | | |
| Rural (non-MSA) | | | | | | | | | | 0 | 0 | 0.00 |
| Urban; n (%) | - | - | | 24,996 (77.4%) | 12,798 (72.1%) | 0.12 | - | - | | 24,996 (77.4%) | 12,798 (72.1%) | 0.12 |
| Rural; n (%) | - | - | | 490 (1.5%) | 680 (3.8%) | -0.14 | - | - | | 490 (1.5%) | 680 (3.8%) | -0.14 |
| Unknown/Missing; n (%) | - | - | | 6,809 (21.1%) | 4,270 (24.1%) | -0.07 | - | - | | 6,809 (21.1%) | 4,270 (24.1%) | -0.07 |
| | | | | | | Di | ue to CMS cell suppress | ion policy, all values le | ss than 11 are | | | |

Due to CMS cell suppression policy, all values less than 11 are denoted with \*\*

| | | | | | PS-matched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Optur | | | MarketS | | | Medic | | | | POOLED | |
| Variable | Reference-warfarin | Exposure - rivaroxaban<br>(15 or 20 mg) | St. Diff. | Reference- warfarin | Exposure - rivaroxaban<br>(15 or 20 mg) | St. Diff. | Reference-warfarin | Exposure - rivaroxaban<br>(15 or 20 mg) | St. Diff. | Reference- warfarin | Exposure - rivaroxaban<br>(15 or 20 mg) | St. Diff |
| Number of patients | 8,950 | 8,950 | St. Dill. | 11,300 | 11,300 | 3t. Dill. | 31,068 | 31,068 | Jt. Dill. | 51,318 | 51,318 | Jt. Dili |
| Age | 0,550 | 0,550 | | 11,500 | 11,500 | | 51,000 | 32,000 | | 51,515 | 31,310 | |
| mean (sd) | 75.84 (8.34) | 75.85 (8.57) | 0.00 | 75.02 (10.73) | 75.15 (10.38) | -0.01 | 78.73 (8.21) | 78.77 (8.02) | 0.00 | 77.41 (8.85) | 77.46 (8.69) | -0.01 |
| median [IQR] | 77.00 [71.00, 82.00] | 77.00 [71.00, 82.00] | 0.00 | 77.00 [68.00, 83.00] | 77.00 [68.00, 83.00] | 0.00 | 79.00 [74.00, 84.00] | 79.00 [74.00, 84.00] | 0.00 | 78.21 (8.85) | 78.21 (8.69) | 0.00 |
| Age categories without zero category | | | | | | | | | | , , | , , | |
| 18 - 54; n (%) | 198 (2.2%) | 212 (2.4%) | -0.01 | 484 (4.3%) | 371 (3.3%) | 0.05 | 310 (1.0%) | 298 (1.0%) | 0.00 | 992 (1.9%) | 881 (1.7%) | 0.0 |
| 55 - 64; n (%) | 682 (7.6%) | 723 (8.1%) | -0.02 | 1,629 (14.4%) | 1,717 (15.2%) | -0.02 | 998 (3.2%) | 923 (3.0%) | 0.01 | 3,309 (6.4%) | 3,363 (6.6%) | -0.0 |
| 65 - 74; n (%) | 2,239 (25.0%) | 2,150 (24.0%) | 0.02 | 2,325 (20.6%) | 2,352 (20.8%) | 0.00 | 6,715 (21.6%) | 6,584 (21.2%) | 0.01 | 11,279 (22.0%) | 11,086 (21.6%) | 0.0 |
| >= 75; n (%) | 5,831 (65.2%) | 5,865 (65.5%) | -0.01 | 6,862 (60.7%) | 6,860 (60.7%) | 0.00 | 23,045 (74.2%) | 23,263 (74.9%) | -0.02 | 35,738 (69.6%) | 35,988 (70.1%) | -0.0 |
| Gender without zero category- United | 4 472 (50 00/) | 4 525 (50 70() | 0.04 | C 022 (F2 40() | C 020 (F2 40) | 0.00 | 42 627 (40 70) | 42 722 (40 00() | 0.00 | 22 442 (45 40() | 22 207 (45 40) | 0.0 |
| Males; n (%)<br>Females; n (%) | 4,473 (50.0%)<br>4,477 (50.0%) | 4,535 (50.7%)<br>4,415 (49.3%) | -0.01<br>0.01 | 6,033 (53.4%)<br>5,267 (46.6%) | 6,030 (53.4%)<br>5,270 (46.6%) | 0.00 | 12,637 (40.7%)<br>18,431 (59.3%) | 12,722 (40.9%)<br>18,346 (59.1%) | 0.00 | 23,143 (45.1%)<br>28,175 (54.9%) | 23,287 (45.4%)<br>28,031 (54.6%) | -0.0:<br>0.0: |
| Race | 4,477 (50.0%) | 4,415 (49.5%) | 0.01 | 3,267 (46.6%) | 3,270 (46.6%) | 0.00 | 16,431 (39.3%) | 16,546 (59.1%) | 0.00 | 26,173 (34.9%) | 26,031 (34.6%) | 0.0. |
| White; n (%) | | | | | | | 28,382 (91.4%) | 28,419 (91.5%) | | 28,382 (91.4%) | 28,419 (91.5%) | 0.00 |
| Black: n (%) | | | | | | | 1,389 (4.5%) | 1,354 (4.4%) | | 1,389 (4.5%) | 1,354 (4.4%) | 0.00 |
| Asian; n (%) | | | | | | | 339 (1.1%) | 333 (1.1%) | | 339 (1.1%) | 333 (1.1%) | 0.00 |
| Hispanic; n (%) | | | | | | | 433 (1.4%) | 421 (1.4%) | | 433 (1.4%) | 421 (1.4%) | 0.00 |
| North American Native; n (%) | | | | | | | 133 (0.4%) | 136 (0.4%) | | 133 (0.4%) | 136 (0.4%) | 0.00 |
| Other/Unknown; n (%) | | | | | | | 392 (1.3%) | 405 (1.3%) | | 392 (1.3%) | 405 (1.3%) | 0.00 |
| Region without zero category- United v3 (lumping | | | | | | | | | | | | |
| missing&other category with West)Northeast; n (%) | 1,313 (14.7%) | 1,310 (14.6%) | 0.00 | 2,698 (23.9%) | 2,762 (24.4%) | -0.01 | 6,528 (21.0%) | 6,476 (20.8%) | 0.00 | 10,539 (20.5%) | 10,548 (20.6%) | 0.00 |
| South; n (%) | 3,278 (36.6%) | 3,242 (36.2%) | 0.01 | 3,425 (30.3%) | 3,431 (30.4%) | 0.00 | 11,305 (36.4%) | 11,225 (36.1%) | 0.01 | 18,008 (35.1%) | 17,898 (34.9%) | 0.00 |
| Midwest; n (%) | 1,900 (21.2%) | 1,902 (21.3%) | 0.00 | 3,502 (31.0%) | 3,436 (30.4%) | 0.01 | 8,521 (27.4%) | 8,630 (27.8%) | -0.01 | 13,923 (27.1%) | 13,968 (27.2%) | 0.00 |
| West; n (%) | 2,459 (27.5%) | 2,496 (27.9%) | -0.01 | 1,619 (14.3%) | 1,608 (14.2%) | 0.00 | 4,714 (15.2%) | 4,737 (15.2%) | 0.00 | 8,792 (17.1%) | 8,841 (17.2%) | 0.00 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 56 (0.5%) | 63 (0.6%) | -0.01 | N/A | N/A | #VALUE! | 56 (0.5%) | 63 (0.6%) | -0.01 |
| CV Covariates | | | | | | | | | | | | |
| Ischemic heart disease; n (%) | 3,345 (37.4%) | 3,391 (37.9%) | -0.01 | 4,174 (36.9%) | 4,143 (36.7%) | 0.00 | 13,673 (44.0%) | 13,547 (43.6%) | 0.01 | 21,192 (41.3%) | 21,081 (41.1%) | 0.00 |
| Acute MI; n (%) | 283 (3.2%) | 286 (3.2%) | 0.00 | 335 (3.0%) | 321 (2.8%) | 0.01 | 1,279 (4.1%) | 1,279 (4.1%) | 0.00 | 1897 (3.7%) | 1886 (3.7%) | 0.00 |
| ACS/unstable angina; n (%) | 260 (2.9%) | 272 (3.0%) | -0.01 | 329 (2.9%) | 314 (2.8%) | 0.01 | 1,247 (4.0%) | 1,204 (3.9%) | 0.01 | 1836 (3.6%) | 1790 (3.5%) | 0.01 |
| Old MI; n (%) | 511 (5.7%) | 520 (5.8%) | 0.00 | 367 (3.2%) | 368 (3.3%) | -0.01 | 2,737 (8.8%) | 2,639 (8.5%) | 0.01 | 3615 (7.0%) | 3527 (6.9%) | 0.00 |
| Stable angina; n (%) Coronary atherosclerosis and other forms of chronic | 482 (5.4%) | 502 (5.6%) | -0.01 | 456 (4.0%) | 438 (3.9%) | 0.01 | 1,541 (5.0%) | 1,478 (4.8%) | 0.01 | 2,479 (4.8%) | 2,418 (4.7%) | 0.00 |
| ischemic heart disease: n (%) | 3,067 (34.3%) | 3,086 (34.5%) | 0.00 | 3,851 (34.1%) | 3,793 (33.6%) | 0.01 | 12,563 (40.4%) | 12,456 (40.1%) | 0.01 | 19,481 (38.0%) | 19,335 (37.7%) | 0.01 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) | 142 (1.6%) | 152 (1.7%) | -0.01 | 210 (1.9%) | 212 (1.9%) | 0.00 | 545 (1.8%) | 561 (1.8%) | 0.00 | 897 (1.7%) | 925 (1.8%) | -0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent) | ,, | . , . , | | , , , , | , , | | , | | | . , | , | |
| v4; n (%) | 119 (1.3%) | 70 (0.8%) | 0.05 | 164 (1.5%) | 94 (0.8%) | 0.07 | 581 (1.9%) | 386 (1.2%) | 0.06 | 864 (1.7%) | 550 (1.1%) | 0.05 |
| History of CABG or PTCA; n (%) | 862 (9.6%) | 877 (9.8%) | -0.01 | 539 (4.8%) | 614 (5.4%) | -0.03 | 4,822 (15.5%) | 4,833 (15.6%) | 0.00 | 6,223 (12.1%) | 6,324 (12.3%) | -0.01 |
| Any stroke; n (%) | 1,763 (19.7%) | 1,721 (19.2%) | 0.01 | 2,030 (18.0%) | 2,018 (17.9%) | 0.00 | 6,768 (21.8%) | 6,728 (21.7%) | 0.00 | 10,561 (20.6%) | 10,467 (20.4%) | 0.00 |
| Ischemic stroke (w and w/o mention of cerebral | | | | | | | | | | | | |
| infarction); n (%) | 1,763 (19.7%) | 1,721 (19.2%) | 0.01 | 2,030 (18.0%) | 2,018 (17.9%) | 0.00 | 6,754 (21.7%) | 6,712 (21.6%) | 0.00 | 10,547 (20.6%) | 10,451 (20.4%) | 0.00 |
| Hemorrhagic stroke; n (%) | 0 (0.0%)<br>691 (7.7%) | 0 (0.0%)<br>671 (7.5%) | #DIV/0!<br>0.01 | 0 (0.0%) | 0 (0.0%) | #DIV/0!<br>0.00 | 84 (0.3%) | 82 (0.3%) | 0.00 | 084 (0.2%)<br>3614 (7.0%) | 82 (0.2%)<br>3587 (7.0%) | 0.00 |
| TIA; n (%) Other cerebrovascular disease; n (%) | 373 (4.2%) | 358 (4.0%) | 0.01 | 830 (7.3%)<br>361 (3.2%) | 826 (7.3%)<br>359 (3.2%) | 0.00 | 2,093 (6.7%)<br>1,630 (5.2%) | 2,090 (6.7%)<br>1,585 (5.1%) | 0.00 | 2364 (4.6%) | 2302 (4.5%) | 0.00 |
| Late effects of cerebrovascular disease; n (%) | 364 (4.1%) | 365 (4.1%) | 0.00 | 300 (2.7%) | 293 (2.6%) | 0.01 | 1,876 (6.0%) | 1,871 (6.0%) | 0.00 | 2540 (4.9%) | 2529 (4.9%) | 0.00 |
| Cerebrovascular procedure; n (%) | 14 (0.2%) | 11 (0.1%) | 0.03 | 20 (0.2%) | 22 (0.2%) | 0.00 | 100 (0.3%) | 89 (0.3%) | 0.00 | 134 (0.3%) | 122 (0.2%) | 0.02 |
| Heart failure (CHF); n (%) | 2,372 (26.5%) | 2,375 (26.5%) | 0.00 | 2,676 (23.7%) | 2,699 (23.9%) | 0.00 | 11,720 (37.7%) | 11,670 (37.6%) | 0.00 | 16,768 (32.7%) | 16,744 (32.6%) | 0.00 |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2; | . , , | . , , | | . , , | , | | , | . , , | | . , , | | |
| n (%) | 912 (10.2%) | 920 (10.3%) | 0.00 | 1,016 (9.0%) | 1,004 (8.9%) | 0.00 | 3,753 (12.1%) | 3,694 (11.9%) | 0.01 | 5,681 (11.1%) | 5,618 (10.9%) | 0.01 |
| Atrial fibrillation; n (%) | 8,698 (97.2%) | 8,704 (97.3%) | -0.01 | 11,051 (97.8%) | 11,001 (97.4%) | 0.03 | 30,164 (97.1%) | 30,159 (97.1%) | 0.00 | 49,913 (97.3%) | 49,864 (97.2%) | 0.01 |
| Other cardiac dysrhythmia; n (%) | 5,962 (66.6%) | 5,864 (65.5%) | 0.02 | 4,868 (43.1%) | 4,794 (42.4%) | 0.01 | 17,844 (57.4%) | 17,748 (57.1%) | 0.01 | 28,674 (55.9%) | 28,406 (55.4%) | 0.01 |
| Cardiac conduction disorders; n (%) | 923 (10.3%) | 893 (10.0%) | 0.01 | 908 (8.0%) | 884 (7.8%) | 0.01 | 3,351 (10.8%) | 3,266 (10.5%) | 0.01 | 5182 (10.1%) | 5043 (9.8%) | 0.01 |
| Other CVD; n (%) | 3,376 (37.7%) | 3,320 (37.1%) | 0.01 | 3,973 (35.2%) | 3,931 (34.8%) | 0.01 | 12,375 (39.8%) | 12,267 (39.5%) | 0.01 | 19,724 (38.4%) | 19,518 (38.0%) | 0.01 |
| Diabetes-related complications Diabetic retinopathy; n (%) | 147 (1.6%) | 162 (1.8%) | -0.02 | 161 (1.4%) | 170 (1.5%) | -0.01 | 537 (1.7%) | 554 (1.8%) | -0.01 | #VALUE! | 886 (1.7%) | #VALUE |
| Diabetic retinopatny; n (%) Diabetes with other ophthalmic manifestations; n | 147 (1.6%) | 102 (1.6%) | -0.02 | 101 (1.4%) | 1/0(1.3%) | -0.01 | 337 (1.7%) | 334 (1.6%) | -0.01 | #VALUE! | 000 (1./%) | #VALUE |
| (%) | 15 (0.2%) | 19 (0.2%) | 0.00 | 139 (1.2%) | 123 (1.1%) | 0.01 | 356 (1.1%) | 355 (1.1%) | 0.00 | 510 (1.0%) | 497 (1.0%) | 0.00 |
| Retinal detachment, vitreous hemorrhage, | (2.79) | (/0) | 2.20 | (-12/0) | (-:-/9) | | (1-/0) | (/9) | | (0/0) | (0/0) | 5.00 |
| vitrectomy; n (%) | 16 (0.2%) | 21 (0.2%) | 0.00 | 26 (0.2%) | 21 (0.2%) | 0.00 | 55 (0.2%) | 65 (0.2%) | 0.00 | 097 (0.2%) | 107 (0.2%) | 0.00 |
| Retinal laser coagulation therapy; n (%) | 12 (0.1%) | 7 (0.1%) | 0.00 | 27 (0.2%) | 21 (0.2%) | 0.00 | 61 (0.2%) | 60 (0.2%) | 0.00 | 100 (0.2%) | 88 (0.2%) | 0.00 |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 558 (6.2%) | 583 (6.5%) | -0.01 | 534 (4.7%) | 551 (4.9%) | -0.01 | 2,148 (6.9%) | 2,163 (7.0%) | 0.00 | 3240 (6.3%) | 3297 (6.4%) | 0.00 |
| Occurrence of diabetic nephropathy V3 with ICD10 | | | | | | | | | | | | |
| Copy; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 401 (1.3%) | 415 (1.3%) | 0.00 | 401 (0.8%) | 415 (0.8%) | 0.00 |
| Hypoglycemia v2; n (%) | 68 (0.8%) | 85 (0.9%) | -0.01 | 146 (1.3%) | 140 (1.2%) | 0.01 | 850 (2.7%) | 854 (2.7%) | 0.00 | 1064 (2.1%) | 1079 (2.1%) | 0.00 |

| Harmonia a (64) | FOC /F 70/) | 400 (F. FR() | 0.01 | 200 (2 70() | 204 (2.6%) | 0.01 | 2 020 (6 50) | 4.000 (6.30() | 0.04 | 2025 (5.50() | 2744 (5.20() | 0.01 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Hyperglycemia; n (%) Disorders of fluid electrolyte and acid-base balance; n | 506 (5.7%) | 490 (5.5%) | 0.01 | 309 (2.7%) | 294 (2.6%) | 0.01 | 2,020 (6.5%) | 1,960 (6.3%) | 0.01 | 2835 (5.5%) | 2744 (5.3%) | 0.01 |
| (%) | 1,013 (11.3%) | 976 (10.9%) | 0.01 | 959 (8.5%) | 934 (8.3%) | 0.01 | 4,247 (13.7%) | 4,163 (13.4%) | 0.01 | 6219 (12.1%) | 6073 (11.8%) | 0.01 |
| Diabetic ketoacidosis; n (%) | 12 (0.1%) | 15 (0.2%) | -0.03 | 18 (0.2%) | 16 (0.1%) | 0.03 | 67 (0.2%) | 61 (0.2%) | 0.00 | 97 (0.2%) | 92 (0.2%) | 0.00 |
| Hyperosmolar hyperglycemic nonketotic syndrome | () | (, | | () | () | | () | () | | () | () | |
| (HONK); n (%) | 7 (0.1%) | 15 (0.2%) | -0.03 | 11 (0.1%) | 9 (0.1%) | 0.00 | 55 (0.2%) | 58 (0.2%) | 0.00 | 73 (0.1%) | 82 (0.2%) | -0.03 |
| Diabetes with peripheral circulatory disorders with | . , | , , | | , , | , , | | , , | , , | | , , | , , | |
| ICD-10 v2 Copy; n (%) | 290 (3.2%) | 248 (2.8%) | 0.02 | 248 (2.2%) | 241 (2.1%) | 0.01 | 1,408 (4.5%) | 1,448 (4.7%) | -0.01 | 1946 (3.8%) | 1937 (3.8%) | 0.00 |
| Diabetic Foot; n (%) | 199 (2.2%) | 181 (2.0%) | 0.01 | 245 (2.2%) | 242 (2.1%) | 0.01 | 1,221 (3.9%) | 1,196 (3.8%) | 0.01 | 1665 (3.2%) | 1619 (3.2%) | 0.00 |
| Gangrene v2; n (%) | 10 (0.1%) | 18 (0.2%) | -0.03 | 15 (0.1%) | 9 (0.1%) | 0.00 | 73 (0.2%) | 66 (0.2%) | 0.00 | 098 (0.2%) | 93 (0.2%) | 0.00 |
| Lower extremity amputation; n (%) | 40 (0.4%) | 36 (0.4%) | 0.00 | 16 (0.1%) | 21 (0.2%) | -0.03 | 193 (0.6%) | 163 (0.5%) | 0.01 | 249 (0.5%) | 220 (0.4%) | 0.01 |
| Osteomyelitis; n (%) | 31 (0.3%) | 29 (0.3%) | 0.00 | 42 (0.4%) | 47 (0.4%) | 0.00 | 194 (0.6%) | 207 (0.7%) | -0.01 | 267 (0.5%) | 283 (0.6%) | -0.01 |
| Skin infections v2; n (%) | 480 (5.4%) | 496 (5.5%) | 0.00 | 706 (6.2%) | 697 (6.2%) | 0.00 | 2,223 (7.2%) | 2,259 (7.3%) | 0.00 | 3409 (6.6%) | 3452 (6.7%) | 0.00 |
| Erectile dysfunction; n (%) | 161 (1.8%) | 156 (1.7%) | 0.01 | 172 (1.5%) | 179 (1.6%) | -0.01 | 238 (0.8%) | 233 (0.7%) | 0.01 | 571 (1.1%) | 568 (1.1%) | 0.00 |
| Diabetes with unspecified complication; n (%) | 144 (1.6%) | 150 (1.7%) | -0.01 | 137 (1.2%) | 137 (1.2%) | 0.00 | 545 (1.8%) | 515 (1.7%) | 0.01 | 826 (1.6%) | 802 (1.6%) | 0.00 |
| Diabetes mellitus without mention of complications; | | | | | | | | | | | | |
| n (%) | 3,162 (35.3%) | 3,150 (35.2%) | 0.00 | 3,738 (33.1%) | 3,747 (33.2%) | 0.00 | 13,515 (43.5%) | 13,644 (43.9%) | -0.01 | 20,415 (39.8%) | 20,541 (40.0%) | 0.00 |
| Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) | 7,782 (86.9%) | 7,761 (86.7%) | 0.01 | 8,716 (77.1%) | 8,716 (77.1%) | 0.00 | 29,357 (94.5%) | 29,270 (94.2%) | 0.01 | 45,855 (89.4%) | 45,747 (89.1%) | 0.01 |
| Hyperlipidemia v2; n (%) | 5,766 (64.4%) | 5,800 (64.8%) | -0.01 | 5,868 (51.9%) | 5,812 (51.4%) | 0.01 | 19,778 (63.7%) | 19,631 (63.2%) | 0.01 | 31,412 (61.2%) | 31,243 (60.9%) | 0.01 |
| Edema; n (%) | 1,034 (11.6%) | 1,057 (11.8%) | -0.01 | 1,013 (9.0%) | 960 (8.5%) | 0.02 | 3,510 (11.3%) | 3,503 (11.3%) | 0.00 | 5557 (10.8%) | 5520 (10.8%) | 0.00 |
| Renal Dysfunction (non-diabetic) v2; n (%) | 4 (0.0%) | 4 (0.0%) | #DIV/0! | 11 (0.1%) | 12 (0.1%) | 0.00 | 1,202 (3.9%) | 1,189 (3.8%) | 0.01 | 1217 (2.4%) | 1205 (2.3%) | 0.01 |
| Occurrence of acute renal disease v2; n (%) | 3 (0.0%) | 3 (0.0%) | #DIV/0! | 11 (0.1%) | 12 (0.1%) | 0.00 | 162 (0.5%) | 150 (0.5%) | 0.00 | 176 (0.3%) | 165 (0.3%) | 0.00 |
| Occurrence of chronic renal insufficiency; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 666 (2.1%) | 671 (2.2%) | -0.01 | 666 (1.3%) | 671 (1.3%) | 0.00 |
| Chronic kidney disease v2; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 629 (2.0%) | 629 (2.0%) | 0.00 | 629 (1.2%) | 629 (1.2%) | 0.00 |
| CKD Stage 3-4; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 458 (1.5%) | 438 (1.4%) | 0.01 | 458 (0.9%) | 438 (0.9%) | 0.00 |
| Occurrence of hypertensive nephropathy; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 184 (0.6%) | 174 (0.6%) | 0.00 | 184 (0.4%) | 174 (0.3%) | 0.02 |
| Occurrence of miscellaneous renal insufficiency v2; n | | | | | | | | | | | | |
| (%) | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 470 (1.5%) | 471 (1.5%) | 0.00 | 471 (0.9%) | 472 (0.9%) | 0.00 |
| Glaucoma or cataracts v2; n (%) | 1,894 (21.2%) | 1,900 (21.2%) | 0.00 | 2,536 (22.4%) | 2,439 (21.6%) | 0.02 | 6,537 (21.0%) | 6,644 (21.4%) | -0.01 | 10,967 (21.4%) | 10,983 (21.4%) | 0.00 |
| Cellulitis or abscess of toe; n (%) | 118 (1.3%) | 139 (1.6%) | -0.03 | 108 (1.0%) | 111 (1.0%) | 0.00 | 576 (1.9%) | 566 (1.8%) | 0.01 | 802 (1.6%) | 816 (1.6%) | 0.00 |
| Foot ulcer; n (%) | 202 (2.3%) | 183 (2.0%) | 0.02 | 254 (2.2%) | 247 (2.2%) | 0.00 | 1,089 (3.5%) | 1,063 (3.4%) | 0.01 | 1545 (3.0%) | 1493 (2.9%) | 0.01 |
| Bladder stones; n (%) | 4 (0.0%) | 8 (0.1%) | -0.04 | 10 (0.1%) | 11 (0.1%) | 0.00 | 32 (0.1%) | 38 (0.1%) | 0.00 | 46 (0.1%) | 57 (0.1%) | 0.00 |
| Kidney stones; n (%) | 82 (0.9%) | 90 (1.0%) | -0.01 | 115 (1.0%) | 120 (1.1%) | -0.01 | 471 (1.5%) | 470 (1.5%) | 0.00 | 668 (1.3%) | 680 (1.3%) | 0.00 |
| Urinary tract infections (UTIs); n (%) | 863 (9.6%) | 811 (9.1%) | 0.02 | 866 (7.7%) | 893 (7.9%) | -0.01 | 5,140 (16.5%) | 5,099 (16.4%) | 0.00 | 6,869 (13.4%) | 6,803 (13.3%) | 0.00 |
| Dipstick urinalysis; n (%) | 2,549 (28.5%) | 2,577 (28.8%) | -0.01 | 2,309 (20.4%) | 2,468 (21.8%) | -0.03 | 11,599 (37.3%) | 12,095 (38.9%) | -0.03 | 16,457 (32.1%) | 17,140 (33.4%) | -0.03 |
| Non-dipstick urinalysis; n (%) | 1,254 (14.0%) | 1,189 (13.3%) | 0.02 | 693 (6.1%) | 660 (5.8%) | 0.01 | 4,879 (15.7%) | 4,740 (15.3%) | 0.01 | 6,826 (13.3%) | 6,589 (12.8%) | 0.01 |
| Urine function test; n (%) | 241 (2.7%) | 209 (2.3%) | 0.03 | 443 (3.9%) | 383 (3.4%) | 0.03 | 1,175 (3.8%) | 1,210 (3.9%) | -0.01 | 1859 (3.6%) | 1802 (3.5%) | 0.01 |
| Cytology; n (%) | 75 (0.8%)<br>88 (1.0%) | 105 (1.2%)<br>77 (0.9%) | -0.04<br>0.01 | 128 (1.1%) | 111 (1.0%)<br>136 (1.2%) | 0.01<br>0.03 | 613 (2.0%)<br>622 (2.0%) | 709 (2.3%)<br>648 (2.1%) | -0.02<br>-0.01 | 816 (1.6%)<br>892 (1.7%) | 925 (1.8%)<br>861 (1.7%) | -0.02<br>0.00 |
| Cystoscopy; n (%) Other Covariates | 00 (1.0%) | 77 (0.9%) | 0.01 | 182 (1.6%) | 130 (1.2%) | 0.03 | 022 (2.0%) | 046 (2.1%) | -0.01 | 892 (1.7%) | 001 (1.7%) | 0.00 |
| Liver disease: n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 366 (1.2%) | 348 (1.1%) | 0.01 | 366 (0.7%) | 348 (0.7%) | 0.00 |
| Osteoarthritis: n (%) | 1,847 (20.6%) | 1,844 (20.6%) | 0.00 | 1,933 (17.1%) | 1,954 (17.3%) | -0.01 | 7,796 (25.1%) | 7,776 (25.0%) | 0.00 | 11576 (22.6%) | 11574 (22.6%) | 0.00 |
| Other arthritis, arthropathies and musculoskeletal | 2,017 (20.070) | 2,011 (20.070) | 0.00 | 1,555 (17.170) | 1,551 (17.570) | 0.01 | 7,730 (23.270) | 7,770 (23.070) | 0.00 | 11370 (22.070) | 11374 (22.070) | 0.00 |
| pain; n (%) | 3,488 (39.0%) | 3,487 (39.0%) | 0.00 | 4,219 (37.3%) | 4,209 (37.2%) | 0.00 | 13,347 (43.0%) | 13,256 (42.7%) | 0.01 | 21054 (41.0%) | 20952 (40.8%) | 0.00 |
| Dorsopathies; n (%) | 1,992 (22.3%) | 2,023 (22.6%) | -0.01 | 2,342 (20.7%) | 2,342 (20.7%) | 0.00 | 7,506 (24.2%) | 7,495 (24.1%) | 0.00 | 11840 (23.1%) | 11860 (23.1%) | 0.00 |
| Fractures; n (%) | 349 (3.9%) | 340 (3.8%) | 0.01 | 447 (4.0%) | 480 (4.2%) | -0.01 | 1,787 (5.8%) | 1,785 (5.7%) | 0.00 | 2583 (5.0%) | 2605 (5.1%) | 0.00 |
| Falls v2; n (%) | 473 (5.3%) | 478 (5.3%) | 0.00 | 232 (2.1%) | 227 (2.0%) | 0.01 | 992 (3.2%) | 1,011 (3.3%) | -0.01 | 1697 (3.3%) | 1716 (3.3%) | 0.00 |
| Osteoporosis; n (%) | 768 (8.6%) | 746 (8.3%) | 0.01 | 702 (6.2%) | 709 (6.3%) | 0.00 | 3,282 (10.6%) | 3,320 (10.7%) | 0.00 | 4752 (9.3%) | 4775 (9.3%) | 0.00 |
| Hyperthyroidism; n (%) | 124 (1.4%) | 103 (1.2%) | 0.02 | 109 (1.0%) | 111 (1.0%) | 0.00 | 430 (1.4%) | 440 (1.4%) | 0.00 | 663 (1.3%) | 654 (1.3%) | 0.00 |
| Hypothyroidism v2; n (%) | 1,709 (19.1%) | 1,709 (19.1%) | 0.00 | 1,606 (14.2%) | 1,556 (13.8%) | 0.01 | 4,788 (15.4%) | 4,787 (15.4%) | 0.00 | 8103 (15.8%) | 8052 (15.7%) | 0.00 |
| Other disorders of thyroid gland V2; n (%) | 334 (3.7%) | 325 (3.6%) | 0.01 | 373 (3.3%) | 400 (3.5%) | -0.01 | 1,184 (3.8%) | 1,157 (3.7%) | 0.01 | 1891 (3.7%) | 1882 (3.7%) | 0.00 |
| Depression; n (%) | 753 (8.4%) | 771 (8.6%) | -0.01 | 695 (6.2%) | 716 (6.3%) | 0.00 | 3,844 (12.4%) | 3,846 (12.4%) | 0.00 | 5292 (10.3%) | 5333 (10.4%) | 0.00 |
| Anxiety; n (%) | 874 (9.8%) | 866 (9.7%) | 0.00 | 659 (5.8%) | 673 (6.0%) | -0.01 | 3,598 (11.6%) | 3,556 (11.4%) | 0.01 | 5131 (10.0%) | 5095 (9.9%) | 0.00 |
| Sleep_Disorder; n (%) | 726 (8.1%) | 736 (8.2%) | 0.00 | 1,294 (11.5%) | 1,277 (11.3%) | 0.01 | 2,776 (8.9%) | 2,753 (8.9%) | 0.00 | 4796 (9.3%) | 4766 (9.3%) | 0.00 |
| Dementia; n (%) | 684 (7.6%) | 653 (7.3%) | 0.01 | 618 (5.5%) | 610 (5.4%) | 0.00 | 3,305 (10.6%) | 3,289 (10.6%) | 0.00 | 4607 (9.0%) | 4552 (8.9%) | 0.00 |
| Delirium; n (%) | 171 (1.9%) | 170 (1.9%) | 0.00 | 164 (1.5%) | 174 (1.5%) | 0.00 | 1,074 (3.5%) | 1,042 (3.4%) | 0.01 | 1409 (2.7%) | 1386 (2.7%) | 0.00 |
| Psychosis; n (%) | 126 (1.4%) | 117 (1.3%) | 0.01 | 136 (1.2%) | 142 (1.3%) | -0.01 | 734 (2.4%) | 737 (2.4%) | 0.00 | 996 (1.9%) | 996 (1.9%) | 0.00 |
| Obesity; n (%) Overweight; n (%) | 1,384 (15.5%)<br>423 (4.7%) | 1,388 (15.5%)<br>421 (4.7%) | 0.00 | 1,122 (9.9%)<br>190 (1.7%) | 1,195 (10.6%)<br>179 (1.6%) | -0.02<br>0.01 | 5,082 (16.4%)<br>988 (3.2%) | 4,996 (16.1%)<br>1,015 (3.3%) | 0.01<br>-0.01 | 7588 (14.8%)<br>1601 (3.1%) | 7579 (14.8%)<br>1615 (3.1%) | 0.00 |
| Smoking; n (%) | 1,515 (16.9%) | 1,472 (16.4%) | 0.01 | 801 (7.1%) | 817 (7.2%) | 0.00 | 8,813 (28.4%) | 8,655 (27.9%) | 0.01 | 11129 (21.7%) | 10944 (21.3%) | 0.01 |
| Alcohol abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 24 (0.1%) | 22 (0.1%) | 0.00 | 24 (0.0%) | 22 (0.0%) | #DIV/0! |
| Drug abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 72 (0.2%) | 62 (0.2%) | 0.00 | 72 (0.1%) | 62 (0.1%) | 0.00 |
| COPD; n (%) | 1,561 (17.4%) | 1,567 (17.5%) | 0.00 | 1,692 (15.0%) | 1,671 (14.8%) | 0.01 | 6,895 (22.2%) | 6,863 (22.1%) | 0.00 | 10148 (19.8%) | 10101 (19.7%) | 0.00 |
| Asthma; n (%) | 627 (7.0%) | 613 (6.8%) | 0.01 | 701 (6.2%) | 692 (6.1%) | 0.00 | 2,585 (8.3%) | 2,551 (8.2%) | 0.00 | 3913 (7.6%) | 3856 (7.5%) | 0.00 |
| Obstructive sleep apnea; n (%) | 1,002 (11.2%) | 991 (11.1%) | 0.00 | 1,245 (11.0%) | 1,186 (10.5%) | 0.02 | 3,001 (9.7%) | 2,961 (9.5%) | 0.01 | 5248 (10.2%) | 5138 (10.0%) | 0.01 |
| Pneumonia; n (%) | 583 (6.5%) | 564 (6.3%) | 0.01 | 757 (6.7%) | 774 (6.8%) | 0.00 | 3,435 (11.1%) | 3,386 (10.9%) | 0.01 | 4775 (9.3%) | 4724 (9.2%) | 0.00 |
| Imaging; n (%) | 13 (0.1%) | 12 (0.1%) | 0.00 | 17 (0.2%) | 14 (0.1%) | 0.03 | 166 (0.5%) | 132 (0.4%) | 0.01 | 196 (0.4%) | 158 (0.3%) | 0.02 |
| Other Medications | , , | , , | | , , | | | , , | , , | | , , | . , | |

| Use of ACE inhibitors; n (%) | 3,302 (36.9%) | 3.351 (37.4%) | -0.01 | 4.037 (35.7%) | 4,053 (35.9%) | 0.00 | 12.056 (38.8%) | 12,104 (39.0%) | 0.00 | 19395 (37.8%) | 19508 (38.0%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Use of ARBs; n (%) | 2,148 (24.0%) | 2,097 (23.4%) | 0.01 | 2,946 (26.1%) | 2,929 (25.9%) | 0.00 | 7,885 (25.4%) | 7,901 (25.4%) | 0.00 | 12979 (25.3%) | 12927 (25.2%) | 0.00 |
| Use of Loop Diuretics - United; n (%) | 2,452 (27.4%) | 2,457 (27.5%) | 0.00 | 3,074 (27.2%) | 2,962 (26.2%) | 0.02 | 12,075 (38.9%) | 12,145 (39.1%) | 0.00 | 17601 (34.3%) | 17564 (34.2%) | 0.00 |
| Use of other diuretics - United; If (%) | 499 (5.6%) | 452 (5.1%) | 0.00 | 678 (6.0%) | , | 0.02 | 2,204 (7.1%) | | 0.00 | 3381 (6.6%) | 3286 (6.4%) | 0.00 |
| , | | | 0.02 | | 628 (5.6%) | 0.02 | | 2,206 (7.1%) | 0.00 | | | 0.01 |
| Use of nitrates-United; n (%) | 721 (8.1%) | 639 (7.1%) | | 1,067 (9.4%) | 937 (8.3%) | | 3,909 (12.6%) | 3,522 (11.3%) | | 5697 (11.1%) | 5098 (9.9%) | |
| Use of other hypertension drugs; n (%) | 658 (7.4%) | 690 (7.7%) | -0.01 | 798 (7.1%) | 953 (8.4%) | -0.05 | 2,616 (8.4%) | 2,741 (8.8%) | -0.01 | 4072 (7.9%) | 4384 (8.5%) | -0.02 |
| Use of digoxin- United; n (%) | 1,060 (11.8%) | 907 (10.1%) | 0.05 | 1,932 (17.1%) | 1,413 (12.5%) | 0.13 | 4,898 (15.8%) | 4,232 (13.6%) | 0.06 | 7890 (15.4%) | 6552 (12.8%) | 0.07 |
| Use of Anti-arrhythmics; n (%) | 1,039 (11.6%) | 1,022 (11.4%) | 0.01 | 1,549 (13.7%) | 1,578 (14.0%) | -0.01 | 3,969 (12.8%) | 4,042 (13.0%) | -0.01 | 6557 (12.8%) | 6642 (12.9%) | 0.00 |
| Use of COPD/asthma meds- United; n (%) | 1,652 (18.5%) | 1,660 (18.5%) | 0.00 | 2,257 (20.0%) | 2,211 (19.6%) | 0.01 | 7,164 (23.1%) | 6,884 (22.2%) | 0.02 | 11073 (21.6%) | 10755 (21.0%) | 0.01 |
| Use of statins; n (%) | 5,403 (60.4%) | 5,381 (60.1%) | 0.01 | 6,725 (59.5%) | 6,779 (60.0%) | -0.01 | 18,970 (61.1%) | 19,049 (61.3%) | 0.00 | 31098 (60.6%) | 31209 (60.8%) | 0.00 |
| Use of other lipid-lowering drugs; n (%) | 561 (6.3%) | 570 (6.4%) | 0.00 | 1,042 (9.2%) | 1,077 (9.5%) | -0.01 | 2,197 (7.1%) | 2,209 (7.1%) | 0.00 | 3800 (7.4%) | 3856 (7.5%) | 0.00 |
| Use of antiplatelet agents; n (%) | 1,266 (14.1%) | 1,275 (14.2%) | 0.00 | 1,925 (17.0%) | 1,862 (16.5%) | 0.01 | 5,449 (17.5%) | 5,400 (17.4%) | 0.00 | 8640 (16.8%) | 8537 (16.6%) | 0.01 |
| Use of heparin and other low-molecular weight | | | | | | | | | | | | |
| heparins; n (%) | 28 (0.3%) | 48 (0.5%) | -0.03 | 1 (0.0%) | 2 (0.0%) | #DIV/0! | 191 (0.6%) | 270 (0.9%) | -0.03 | 220 (0.4%) | 320 (0.6%) | -0.03 |
| Use of NSAIDs; n (%) | 1,022 (11.4%) | 1,003 (11.2%) | 0.01 | 1,228 (10.9%) | 1,245 (11.0%) | 0.00 | 3,906 (12.6%) | 3,909 (12.6%) | 0.00 | 6156 (12.0%) | 6157 (12.0%) | 0.00 |
| Use of oral corticosteroids; n (%) | 1,770 (19.8%) | 1,758 (19.6%) | 0.01 | 2,198 (19.5%) | 2,216 (19.6%) | 0.00 | 7,748 (24.9%) | 7,700 (24.8%) | 0.00 | 11716 (22.8%) | 11674 (22.7%) | 0.00 |
| Use of bisphosphonate (United); n (%) | 341 (3.8%) | 337 (3.8%) | 0.00 | 381 (3.4%) | 380 (3.4%) | 0.00 | 1,209 (3.9%) | 1,234 (4.0%) | -0.01 | 1931 (3.8%) | 1951 (3.8%) | 0.00 |
| | . , | | | | | | | | | 13747 (26.8%) | | |
| Use of opioids- United; n (%) | 2,033 (22.7%) | 2,065 (23.1%) | -0.01 | 2,709 (24.0%) | 2,735 (24.2%) | 0.00 | 9,005 (29.0%) | 8,989 (28.9%) | 0.00 | | 13789 (26.9%) | 0.00 |
| Use of antidepressants; n (%) | 1,849 (20.7%) | 1,855 (20.7%) | 0.00 | 2,139 (18.9%) | 2,136 (18.9%) | 0.00 | 8,280 (26.7%) | 8,229 (26.5%) | 0.00 | 12268 (23.9%) | 12220 (23.8%) | 0.00 |
| Use of antipsychotics; n (%) | 157 (1.8%) | 157 (1.8%) | 0.00 | 161 (1.4%) | 157 (1.4%) | 0.00 | 956 (3.1%) | 931 (3.0%) | 0.01 | 1274 (2.5%) | 1245 (2.4%) | 0.01 |
| Use of anticonvulsants; n (%) | 1,091 (12.2%) | 1,112 (12.4%) | -0.01 | 1,164 (10.3%) | 1,145 (10.1%) | 0.01 | 4,966 (16.0%) | 4,964 (16.0%) | 0.00 | 7221 (14.1%) | 7221 (14.1%) | 0.00 |
| Use of lithium- United; n (%) | 4 (0.0%) | 6 (0.1%) | -0.04 | 10 (0.1%) | 12 (0.1%) | 0.00 | ** | 23 (0.1%) | #VALUE! | #VALUE! | 41 (0.1%) | #VALUE! |
| Use of Benzos- United; n (%) | 1,012 (11.3%) | 1,061 (11.9%) | -0.02 | 1,532 (13.6%) | 1,498 (13.3%) | 0.01 | 4,482 (14.4%) | 4,481 (14.4%) | 0.00 | 7026 (13.7%) | 7040 (13.7%) | 0.00 |
| Use of anxiolytics/hypnotics- United; n (%) | 479 (5.4%) | 469 (5.2%) | 0.01 | 743 (6.6%) | 762 (6.7%) | 0.00 | 2,166 (7.0%) | 2,139 (6.9%) | 0.00 | 3388 (6.6%) | 3370 (6.6%) | 0.00 |
| Use of dementia meds- United; n (%) | 340 (3.8%) | 346 (3.9%) | -0.01 | 407 (3.6%) | 409 (3.6%) | 0.00 | 1,688 (5.4%) | 1,700 (5.5%) | 0.00 | 2435 (4.7%) | 2455 (4.8%) | 0.00 |
| Use of antiparkinsonian meds- United; n (%) | 236 (2.6%) | 245 (2.7%) | -0.01 | 317 (2.8%) | 306 (2.7%) | 0.01 | 1,223 (3.9%) | 1,253 (4.0%) | -0.01 | 1776 (3.5%) | 1804 (3.5%) | 0.00 |
| Any use of pramlintide; n (%) | 1 (0.0%) | 3 (0.0%) | #DIV/0! | 2 (0.0%) | 1 (0.0%) | #DIV/0! | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Any use of 1st generation sulfonylureas; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.0%) | 0 (0.0%) | #DIV/0! | ** | ** | #VALUE! | #VALUE! | #VALUE! | 0.00 |
| Entresto (sacubitril/valsartan); n (%) | 38 (0.4%) | 22 (0.2%) | 0.04 | 15 (0.1%) | 6 (0.1%) | 0.00 | 35 (0.1%) | 43 (0.1%) | 0.00 | 88 (0.2%) | 71 (0.1%) | 0.00 |
| Labs | 36 (0.4%) | 22 (0.270) | 0.04 | 13 (0.170) | 0 (0.170) | 0.00 | 33 (0.170) | 45 (0.170) | 0.00 | 20,250 | 20,250 | 0.00 |
| Lab values- HbA1c (%) v3; n (%) | 1,433 (16.0%) | 1,474 (16.5%) | -0.01 | 137 (1.2%) | 124 (1.1%) | 0.01 | N/A | N/A | #VALUE! | 1,570 (7.8%) | 1,598 (7.9%) | 0.00 |
| Lab values- HbA1c (%) (within 3 months) v3; n (%) | 941 (10.5%) | 955 (10.7%) | -0.01 | 98 (0.9%) | 89 (0.8%) | 0.01 | N/A | N/A<br>N/A | #VALUE! | | | 0.00 |
| | , , | . , | | , , | , , | | , | | | 1,039 (5.1%) | 1,044 (5.2%) | |
| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 1,433 (16.0%) | 1,474 (16.5%) | -0.01 | 137 (1.2%) | 124 (1.1%) | 0.01 | N/A | N/A | #VALUE! | 1,570 (7.8%) | 1,598 (7.9%) | 0.00 |
| Lab values- BNP; n (%) | 154 (1.7%) | 168 (1.9%) | -0.02 | 18 (0.2%) | 16 (0.1%) | 0.03 | N/A | N/A | #VALUE! | 172 (0.8%) | 184 (0.9%) | -0.01 |
| Lab values- BNP (within 3 months); n (%) | 114 (1.3%) | 132 (1.5%) | -0.02 | 16 (0.1%) | 11 (0.1%) | 0.00 | N/A | N/A | #VALUE! | 130 (0.6%) | 143 (0.7%) | -0.01 |
| Lab values- BNP (within 6 months); n (%) | 154 (1.7%) | 168 (1.9%) | -0.02 | 18 (0.2%) | 16 (0.1%) | 0.03 | N/A | N/A | #VALUE! | 172 (0.8%) | 184 (0.9%) | -0.01 |
| Lab values- BUN (mg/dl); n (%) | 2,374 (26.5%) | 2,650 (29.6%) | -0.07 | 167 (1.5%) | 206 (1.8%) | -0.02 | N/A | N/A | #VALUE! | 2,541 (12.5%) | 2,856 (14.1%) | -0.05 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 1,640 (18.3%) | 1,900 (21.2%) | -0.07 | 121 (1.1%) | 156 (1.4%) | -0.03 | N/A | N/A | #VALUE! | 1,761 (8.7%) | 2,056 (10.2%) | -0.05 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 2,374 (26.5%) | 2,650 (29.6%) | -0.07 | 167 (1.5%) | 206 (1.8%) | -0.02 | N/A | N/A | #VALUE! | 2,541 (12.5%) | 2,856 (14.1%) | -0.05 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 2,429 (27.1%) | 2,743 (30.6%) | -0.08 | 171 (1.5%) | 220 (1.9%) | -0.03 | N/A | N/A | #VALUE! | 2,600 (12.8%) | 2,963 (14.6%) | -0.05 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2; | | | | , , | , , | | • | · | | | | |
| n (%) | 1,676 (18.7%) | 1,980 (22.1%) | -0.08 | 124 (1.1%) | 168 (1.5%) | -0.04 | N/A | N/A | #VALUE! | 1,800 (8.9%) | 2,148 (10.6%) | -0.06 |
| Lab values- Creatinine (mg/dl) (within 6 months) v2; | , , , , , , , | ,, | | | , | | • | • | | , ( , | , . , , | |
| n (%) | 2,429 (27.1%) | 2,743 (30.6%) | -0.08 | 171 (1.5%) | 220 (1.9%) | -0.03 | N/A | N/A | #VALUE! | 2,600 (12.8%) | 2,963 (14.6%) | -0.05 |
| Lab values- HDL level (mg/dl); n (%) | 1,739 (19.4%) | 1,872 (20.9%) | -0.04 | 123 (1.1%) | 132 (1.2%) | -0.01 | N/A | N/A | #VALUE! | 1,862 (9.2%) | 2,004 (9.9%) | -0.02 |
| | _,, | _, (, | | () | () | | | | | _,(, | _,, | |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 1,100 (12.3%) | 1,168 (13.1%) | -0.02 | 87 (0.8%) | 90 (0.8%) | 0.00 | N/A | N/A | #VALUE! | 1,187 (5.9%) | 1,258 (6.2%) | -0.01 |
| ( | -, (, | -, (, | | a. (a.a) | () | | | | | _, (0.07.7) | | |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 1,739 (19.4%) | 1,872 (20.9%) | -0.04 | 123 (1.1%) | 132 (1.2%) | -0.01 | N/A | N/A | #VALUE! | 1,862 (9.2%) | 2,004 (9.9%) | -0.02 |
| Lab values- LDL level (mg/dl) v2; n (%) | 1,819 (20.3%) | 1,948 (21.8%) | -0.04 | 146 (1.3%) | 140 (1.2%) | 0.01 | N/A | N/A | #VALUE! | 1,965 (9.7%) | 2,088 (10.3%) | -0.02 |
| Lab values- LDL level (mg/dl) (within 3 months) v2; n | 1,819 (20.3%) | 1,540 (21.070) | -0.04 | 140 (1.3%) | 140 (1.270) | 0.01 | N/A | IV/A | #VALUE: | 1,903 (9.7%) | 2,000 (10.370) | -0.02 |
| | 1 160 (13 0%) | 1 220 (12 60/) | -0.02 | 104 (0.0%) | 04 (0.00/) | 0.01 | N/A | N/A | #VALUE! | 1 364 (6 3%) | 1 214 (6 50/) | -0.01 |
| (%) | 1,160 (13.0%) | 1,220 (13.6%) | -0.02 | 104 (0.9%) | 94 (0.8%) | 0.01 | N/A | IV/A | #VALUE: | 1,264 (6.2%) | 1,314 (6.5%) | -0.01 |
| Lab values- LDL level (mg/dl) (within 6 months) v2; n<br>(%) | 1,819 (20.3%) | 1,948 (21.8%) | -0.04 | 146 (1.3%) | 140 (1.2%) | 0.01 | N/A | N/A | #VALUE! | 1,965 (9.7%) | 2,088 (10.3%) | -0.02 |
| Lab values- NT-proBNP; n (%) | 15 (0.2%) | 22 (0.2%) | 0.00 | 5 (0.0%) | 2 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 20 (0.1%) | 24 (0.1%) | 0.00 |
| Lab values- NT-proBNP (within 3 months); n (%) | 13 (0.1%) | 19 (0.2%) | -0.03 | 2 (0.0%) | 1 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 15 (0.1%) | 20 (0.1%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 15 (0.2%) | 22 (0.2%) | 0.00 | 5 (0.0%) | 2 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 20 (0.1%) | 24 (0.1%) | - |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 1,765 (19.7%) | 1,886 (21.1%) | -0.03 | 119 (1.1%) | 131 (1.2%) | -0.01 | N/A | N/A | #VALUE! | 1,884 (9.3%) | 2,017 (10.0%) | -0.02 |
| Lab values-Total cholesterol (mg/dl) (within 3 | | | | | | | | | | | | |
| months) v2; n (%) | 1,122 (12.5%) | 1,179 (13.2%) | -0.02 | 83 (0.7%) | 89 (0.8%) | -0.01 | N/A | N/A | #VALUE! | 1,205 (6.0%) | 1,268 (6.3%) | -0.01 |
| Lab values-Total cholesterol (mg/dl) (within 6 | | | | | | | | | | | | |
| months) v2; n (%) | 1,765 (19.7%) | 1,886 (21.1%) | -0.03 | 119 (1.1%) | 131 (1.2%) | -0.01 | N/A | N/A | #VALUE! | 1,884 (9.3%) | 2,017 (10.0%) | -0.02 |
| Lab values-Triglyceride level (mg/dl); n (%) | 1,734 (19.4%) | 1,874 (20.9%) | -0.04 | 121 (1.1%) | 132 (1.2%) | -0.01 | N/A | N/A | #VALUE! | 1,855 (9.2%) | 2,006 (9.9%) | -0.02 |
| Lab values- Triglyceride level (mg/dl) (within 3 | | | | | | | | | | | | |
| months); n (%) | 1,100 (12.3%) | 1,170 (13.1%) | -0.02 | 86 (0.8%) | 90 (0.8%) | 0.00 | N/A | N/A | #VALUE! | 1,186 (5.9%) | 1,260 (6.2%) | -0.01 |
| Lab values-Triglyceride level (mg/dl) (within 6 | | | | | | | | | | | | |
| months); n (%) | 1,734 (19.4%) | 1,874 (20.9%) | -0.04 | 121 (1.1%) | 132 (1.2%) | -0.01 | N/A | N/A | #VALUE! | 1,855 (9.2%) | 2,006 (9.9%) | -0.02 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | | | | | | | | | | | | |
| included) v4 | 1,416 | 1,466 | | 122 | 122 | | N/A | N/A | | 1,538 | 1,588 | |

| mean (sd) | 6.48 (1.08) | 6.51 (1.20) | -0.03 | 6.91 (1.38) | 6.62 (1.12) | 0.23 | N/A | N/A | #VALUE! | 6.51 (1.11) | 6.52 (1.19) | -0.01 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| median [IQR] | 6.20 [5.80, 6.90] | 6.20 [5.80, 6.90] | 0.00 | 6.50 [6.00, 7.53] | 6.50 [6.00, 7.20] | 0.00 | N/A | N/A | #VALUE! | 6.22 (1.11) | 6.22 (1.19) | 0.00 |
| Missing; n (%) | 7,534 (84.2%) | 7,484 (83.6%) | 0.02 | 11,178 (98.9%) | 11,178 (98.9%) | 0.00 | N/A | N/A | #VALUE! | 18,712 (92.4%) | 18,662 (92.2%) | 0.01 |
| Lab result number- BNP mean v2 | 154 | 168 | | 18 | 16 | | N/A | N/A | | 172 | 184 | |
| mean (sd) | 341.80 (493.50) | 331.40 (517.59) | 0.02 | 513.00 (1,035.89) | 408.20 (481.08) | 0.13 | N/A | N/A | #VALUE! | 359.72 (573.09) | 338.08 (516.10) | 0.04 |
| median [IQR] | 208.70 [104.59, 362.50] | 225.62 [98.17, 371.25] | -0.03 | | 237.25 [100.00, 415.75] | -0.11 | N/A | N/A | #VALUE! | 202.40 (573.09) | 226.63 (516.10) | -0.04 |
| Missing; n (%) | 8,796 (98.3%) | 8,782 (98.1%) | 0.02 | 11,282 (99.8%) | 11,284 (99.9%) | -0.03 | N/A | N/A | #VALUE! | 20,078 (99.2%) | 20,066 (99.1%) | 0.01 |
| | | | 0.02 | | | -0.03 | | | #VALUE: | | | 0.01 |
| Lab result number-BUN (mg/dl) mean v2 | 2,374 | 2,650 | | 167 | 206 | | N/A | N/A | | 2,541 | 2,856 | |
| mean (sd) | 18.15 (6.34) | 18.15 (6.10) | 0.00 | 17.73 (6.63) | 20.03 (6.83) | -0.34 | N/A | N/A | #VALUE! | 18.12 (6.36) | 18.29 (6.16) | -0.03 |
| median [IQR] | 17.00 [14.00, 21.00] | 17.00 [14.00, 21.00] | 0.00 | 17.50 [14.00, 21.00] | 18.38 [16.00, 23.00] | -0.13 | N/A | N/A | #VALUE! | 17.03 (6.36) | 17.10 (6.16) | -0.01 |
| Missing; n (%) | 6,576 (73.5%) | 6,300 (70.4%) | 0.07 | 11,133 (98.5%) | 11,094 (98.2%) | 0.02 | N/A | N/A | #VALUE! | 17,709 (87.5%) | 17,394 (85.9%) | 0.05 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 | | | | | | | | | | | | |
| to 15 included) v3 | 2,407 | 2,715 | | 166 | 218 | | N/A | N/A | | 2,573 | 2,933 | |
| mean (sd) | 0.97 (0.24) | 0.96 (0.24) | 0.04 | 0.98 (0.22) | 1.00 (0.24) | -0.09 | N/A | N/A | #VALUE! | 0.97 (0.24) | 0.96 (0.24) | 0.04 |
| median [IQR] | 0.94 [0.80, 1.10] | 0.94 [0.81, 1.09] | 0.00 | 0.98 [0.82, 1.11] | 0.99 [0.81, 1.14] | -0.04 | N/A | N/A | #VALUE! | 0.94 (0.24) | 0.94 (0.24) | 0.00 |
| Missing; n (%) | 6,543 (73.1%) | 6,235 (69.7%) | 0.08 | 11,134 (98.5%) | 11,082 (98.1%) | 0.03 | N/A | N/A | #VALUE! | 17,677 (87.3%) | 17,317 (85.5%) | 0.05 |
| Lab result number- HDL level (mg/dl) mean (only | 0,3 13 (7 3.170) | 0,233 (03.770) | 0.00 | 11,131 (30.370) | 11,002 (50.170) | 0.03 | , | 14/11 | WAY LOC. | 17,077 (07.570) | 17,517 (65.576) | 0.05 |
| | 1 720 | 1,872 | | 123 | 132 | | N/A | N/A | | 1.862 | 2,004 | |
| =<5000 included) v2 | 1,739 | | | | | | | | | *** | | |
| mean (sd) | 51.74 (16.26) | 52.61 (16.33) | -0.05 | 44.07 (17.47) | 48.84 (15.34) | -0.29 | N/A | N/A | #VALUE! | 51.23 (16.35) | 52.36 (16.27) | -0.07 |
| median [IQR] | 49.50 [40.00, 60.00] | 50.00 [41.00, 62.00] | -0.03 | 43.00 [34.00, 52.00] | 48.75 [37.00, 57.00] | -0.35 | N/A | N/A | #VALUE! | 49.07 (16.35) | 49.92 (16.27) | -0.05 |
| Missing; n (%) | 7,211 (80.6%) | 7,078 (79.1%) | 0.04 | 11,177 (98.9%) | 11,168 (98.8%) | 0.01 | N/A | N/A | #VALUE! | 18,388 (90.8%) | 18,246 (90.1%) | 0.02 |
| Lab result number- LDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 1,776 | 1,911 | | 120 | 137 | | N/A | N/A | | 1,896 | 2,048 | |
| mean (sd) | 88.73 (32.54) | 86.79 (32.88) | 0.06 | 83.58 (33.64) | 88.09 (35.90) | -0.13 | N/A | N/A | #VALUE! | 88.40 (32.62) | 86.88 (33.10) | 0.05 |
| median [IQR] | 85.00 [67.00, 108.00] | 83.00 [64.00, 104.00] | 0.06 | 81.00 [62.25, 103.38] | 84.00 [64.00, 113.00] | -0.09 | N/A | N/A | #VALUE! | 84.75 (32.62) | 83.07 (33.10) | 0.05 |
| Missing; n (%) | 7,174 (80.2%) | 7,039 (78.6%) | 0.04 | 11,180 (98.9%) | 11,163 (98.8%) | 0.01 | N/A | N/A | #VALUE! | 18,354 (90.6%) | 18,202 (89.9%) | 0.02 |
| | 7,174 (00.270) | 7,033 (76.0%) | 0.04 | 11,100 (50.5%) | 11,103 (30.070) | 0.01 | 11/1 | 19/5 | #VALUE: | 10,554 (50.0%) | 10,202 (03.570) | 0.02 |
| Lab result number-Total cholesterol (mg/dl) mean<br>(only =<5000 included) v2 | 1,763 | 1,884 | | 119 | 131 | | N/A | N/A | | 1,882 | 2,015 | |
| | | | | | | | · | • | | | | |
| mean (sd) | 165.93 (40.58) | 165.05 (40.64) | 0.02 | 155.14 (47.10) | 162.30 (41.22) | -0.16 | N/A | N/A | #VALUE! | 165.25 (41.03) | 164.87 (40.69) | 0.01 |
| median [IQR] | 161.00 [139.00, 190.00] | 161.00 [137.00, 188.00] | | 158.00 [134.00, 184.00] | 159.00 [131.00, 194.00] | -0.02 | N/A | N/A | #VALUE! | 160.81 (41.03) | 160.87 (40.69) | 0.00 |
| Missing; n (%) | 7,187 (80.3%) | 7,066 (78.9%) | 0.03 | 11,181 (98.9%) | 11,169 (98.8%) | 0.01 | N/A | N/A | #VALUE! | 18,368 (90.7%) | 18,235 (90.0%) | 0.02 |
| Lab result number-Triglyceride level (mg/dl) mean | | | | | | | | | | | | |
| (only =<5000 included) v2 | 1,734 | 1,874 | | 121 | 132 | | N/A | N/A | | 1,855 | 2,006 | |
| mean (sd) | 128.92 (81.96) | 125.55 (76.48) | 0.04 | 134.40 (74.12) | 124.14 (58.72) | 0.15 | N/A | N/A | #VALUE! | 129.28 (81.50) | 125.46 (75.47) | 0.05 |
| median [IQR] | 112.00 [82.38, 151.62] | 107.00 [79.00, 149.25] | 0.06 | 116.50 [84.50, 179.00] | 117.00 [78.25, 150.00] | -0.01 | N/A | N/A | #VALUE! | 112.29 (81.50) | 107.66 (75.47) | 0.06 |
| Missing; n (%) | 7,216 (80.6%) | 7,076 (79.1%) | 0.04 | 11,179 (98.9%) | 11,168 (98.8%) | 0.01 | N/A | N/A | #VALUE! | 18,395 (90.8%) | 18,244 (90.1%) | 0.02 |
| | 7,210 (80.0%) | 7,070 (73.1%) | 0.04 | 11,179 (98.9%) | 11,108 (56.6%) | 0.01 | N/A | N/A | #VALUE: | 18,393 (90.8%) | 18,244 (90.176) | 0.02 |
| Lab result number- Hemoglobin mean (only >0 | 1.772 | 2.002 | | 127 | 147 | | 21/2 | 11/0 | | 1.899 | 2.450 | |
| included) | -, | 2,003 | | | | | N/A | N/A | | -, | 2,150 | |
| mean (sd) | 13.68 (1.53) | 13.75 (1.63) | -0.04 | 13.23 (2.25) | 13.71 (1.67) | -0.24 | N/A | N/A | #VALUE! | 13.65 (1.59) | 13.75 (1.63) | -0.06 |
| median [IQR] | 13.65 [12.70, 14.70] | 13.80 [12.75, 14.80] | -0.09 | 13.40 [12.30, 14.60] | 13.80 [12.70, 14.70] | -0.20 | N/A | N/A | #VALUE! | 13.63 (1.59) | | |
| Missing; n (%) | 7,178 (80.2%) | | | | | 0.20 | | | | | 13.80 (1.63) | -0.11 |
| Lab result number-Serum sodium mean (only > 90 | | 6,947 (77.6%) | 0.06 | 11,173 (98.9%) | 11,153 (98.7%) | 0.02 | N/A | N/A | #VALUE! | 18,351 (90.6%) | 13.80 (1.63)<br>18,100 (89.4%) | -0.11<br>0.04 |
| and < 190 included) | | 6,947 (77.6%) | 0.06 | 11,173 (98.9%) | 11,153 (98.7%) | | N/A | N/A | #VALUE! | | | |
| mann (cd) | 2,338 | 6,947 (77.6%)<br>2,577 | 0.06 | 11,173 (98.9%)<br>154 | 11,153 (98.7%)<br>188 | | N/A<br>N/A | N/A<br>N/A | #VALUE! | | | |
| mean (sd) | 2,338<br>140.09 (3.01) | | -0.02 | | | | | • | #VALUE! | 18,351 (90.6%) | 18,100 (89.4%) | |
| | 140.09 (3.01) | 2,577<br>140.14 (2.99) | -0.02 | 154<br>139.54 (2.88) | 188<br>139.92 (2.69) | -0.14 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 18,351 (90.6%)<br>2,492<br>140.06 (3.00) | 18,100 (89.4%)<br>2,765<br>140.13 (2.97) | -0.02 |
| median [IQR] | 140.09 (3.01)<br>140.00 [138.50, 142.00] | 2,577<br>140.14 (2.99)<br>140.00 [139.00, 142.00] | -0.02<br>0.00 | 154<br>139.54 (2.88)<br>140.00 [138.00, 141.00] | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00] | 0.02<br>-0.14<br>0.00 | N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A | #VALUE! | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) | 18,100 (89.4%) 2,765 140.13 (2.97) 140.00 (2.97) | -0.02<br>0.00 |
| median [IQR]<br>Missing; n (%) | 140.09 (3.01) | 2,577<br>140.14 (2.99) | -0.02 | 154<br>139.54 (2.88) | 188<br>139.92 (2.69) | -0.14 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 18,351 (90.6%)<br>2,492<br>140.06 (3.00) | 18,100 (89.4%)<br>2,765<br>140.13 (2.97) | -0.02 |
| median [IQR]<br>Missing; n (%)<br>Lab result number-Albumin mean (only >0 and <=10 | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%) | 2,577<br>140.14 (2.99)<br>140.00 [139.00, 142.00]<br>6,373 (71.2%) | -0.02<br>0.00 | 154<br>139.54 (2.88)<br>140.00 [138.00, 141.00]<br>11,146 (98.6%) | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%) | 0.02<br>-0.14<br>0.00 | N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A | #VALUE! | 18,351 (90.6%)<br>2,492<br>140.06 (3.00)<br>140.00 (3.00)<br>17,758 (87.7%) | 18,100 (89.4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) | -0.02<br>0.00 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092 | 2,577<br>140.14 (2.99)<br>140.00 [139.00, 142.00]<br>6,373 (71.2%)<br>2,243 | -0.02<br>0.00<br>0.06 | 154<br>139.54 (2.88)<br>140.00 [138.00, 141.00]<br>11,146 (98.6%) | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%) | -0.14<br>0.00<br>0.02 | N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE!<br>#VALUE! | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) | 18,100 (89.4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 | -0.02<br>0.00<br>0.04 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32) | 2,577<br>140.14 (2.99)<br>140.00 [139.00, 142.00]<br>6,373 (71.2%)<br>2,243<br>4.18 (0.33) | -0.02<br>0.00<br>0.06 | 154<br>139.54 (2.88)<br>140.00 [138.00, 141.00]<br>11,146 (98.6%)<br>112<br>4.01 (0.84) | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%)<br>146<br>4.12 (0.36) | 0.02<br>-0.14<br>0.00<br>0.02 | N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE!<br>#VALUE! | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) | 18,100 (89.4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) | -0.02<br>0.00<br>0.04 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR] | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40] | 2,577<br>140.14 (2.99)<br>140.00 [139.00, 142.00]<br>6,373 (71.2%)<br>2,243<br>4.18 (0.33)<br>4.20 [4.00, 4.40] | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00 | 154<br>139.54 (2.88)<br>140.00 [138.00, 141.00]<br>11,146 (98.6%)<br>112<br>4.01 (0.84)<br>4.20 [3.90, 4.40] | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%)<br>146<br>4.12 (0.36)<br>4.10 (3.90, 4.40] | 0.02<br>-0.14<br>0.00<br>0.02<br>-0.17<br>0.15 | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE!<br>#VALUE!<br>#VALUE! | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) | -0.02<br>0.00<br>0.04<br>-0.06<br>0.03 |
| median [IQR]Missing; n (%) Lab result number- Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%) | 2,577<br>140.14 (2.99)<br>140.00 [139.00, 142.00]<br>6,373 (71.2%)<br>2,243<br>4.18 (0.33) | -0.02<br>0.00<br>0.06 | 154<br>139.54 (2.88)<br>140.00 [138.00, 141.00]<br>11,146 (98.6%)<br>112<br>4.01 (0.84) | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%)<br>146<br>4.12 (0.36) | 0.02<br>-0.14<br>0.00<br>0.02 | N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE!<br>#VALUE! | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) | 18,100 (89.4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) | -0.02<br>0.00<br>0.04 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only>0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%) | 2,577<br>140.14 (2.99)<br>140.00 [139.00, 142.00]<br>6,373 (71.2%)<br>2,243<br>4.18 (0.33)<br>4.20 [4.00, 4.40]<br>6,707 (74.9%) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00 | 154<br>139.54 (2.88)<br>140.00 (138.00, 141.00)<br>11,146 (98.6%)<br>112<br>4.01 (0.84)<br>4.20 (3.90, 4.40)<br>11,188 (99.0%) | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%)<br>146<br>4.12 (0.36)<br>4.10 [3.90, 4.40]<br>11,154 (98.7%) | 0.02<br>-0.14<br>0.00<br>0.02<br>-0.17<br>0.15 | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE!<br>#VALUE!<br>#VALUE! | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) | 18,100 (89.4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) | -0.02<br>0.00<br>0.04<br>-0.06<br>0.03 |
| median [IQR]Missing; n (%) Lab result number- Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%) | 2,577<br>140.14 (2.99)<br>140.00 [139.00, 142.00]<br>6,373 (71.2%)<br>2,243<br>4.18 (0.33)<br>4.20 [4.00, 4.40] | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00 | 154<br>139.54 (2.88)<br>140.00 [138.00, 141.00]<br>11,146 (98.6%)<br>112<br>4.01 (0.84)<br>4.20 [3.90, 4.40] | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%)<br>146<br>4.12 (0.36)<br>4.10 (3.90, 4.40] | 0.02<br>-0.14<br>0.00<br>0.02<br>-0.17<br>0.15 | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE!<br>#VALUE!<br>#VALUE! | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) | -0.02<br>0.00<br>0.04<br>-0.06<br>0.03 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only>0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%) | 2,577<br>140.14 (2.99)<br>140.00 [139.00, 142.00]<br>6,373 (71.2%)<br>2,243<br>4.18 (0.33)<br>4.20 [4.00, 4.40]<br>6,707 (74.9%) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00 | 154<br>139.54 (2.88)<br>140.00 (138.00, 141.00)<br>11,146 (98.6%)<br>112<br>4.01 (0.84)<br>4.20 (3.90, 4.40)<br>11,188 (99.0%) | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%)<br>146<br>4.12 (0.36)<br>4.10 [3.90, 4.40]<br>11,154 (98.7%) | 0.02<br>-0.14<br>0.00<br>0.02<br>-0.17<br>0.15 | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE!<br>#VALUE!<br>#VALUE! | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) | 18,100 (89.4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) | -0.02<br>0.00<br>0.04<br>-0.06<br>0.03 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309 | 2,577<br>140.14 (2.99)<br>140.00 (139.00, 142.00)<br>6,373 (71.2%)<br>2,243<br>4.18 (0.33)<br>4.20 (4.00, 4.40)<br>6,707 (74.9%) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04 | 154<br>139.54 (2.88)<br>140.00 (138.00, 141.00)<br>11,146 (98.6%)<br>112<br>4.01 (0.84)<br>4.20 (3.90, 4.40)<br>11,188 (99.0%)<br>153<br>126.15 (58.00) | 188<br>139.92 (2.69)<br>140.00 (138.00, 142.00)<br>11,112 (98.3%)<br>146<br>4.12 (0.36)<br>4.10 (3.90, 4.40)<br>11,154 (98.7%) | 0.02<br>-0.14<br>0.00<br>0.02<br>-0.17<br>0.15<br>0.03 | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) | -0.02<br>0.00<br>0.04<br>-0.06<br>0.03<br>0.03 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)mean (sd)meain [IQR] | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00] | 2,577<br>140.14 (2.99)<br>140.00 (139.00, 142.00)<br>6,373 (71.2%)<br>2,243<br>4.18 (0.33)<br>4.20 (4.00, 4.40)<br>6,707 (74.9%)<br>2,565<br>113.73 (37.41)<br>103.00 [93.00, 122.50] | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04 | 154<br>139.54 (2.88)<br>140.00 (138.00, 141.00)<br>11,146 (98.6%)<br>112<br>4.01 (0.84)<br>4.20 (3.90, 4.40)<br>11,188 (99.0%)<br>153<br>126.15 (58.00)<br>113.00 (95.00, 135.00) | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%)<br>146<br>4.12 (0.36)<br>4.10 (3.90, 4.40)<br>11,154 (98.7%)<br>186<br>126.78 (41.66)<br>116.00 [100.00, 142.00] | 0.02<br>-0.14<br>0.00<br>0.02<br>-0.17<br>0.15<br>0.03 | N/A | N/A | #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI | 2,492<br>140.06 (3.00)<br>140.00 (3.00)<br>17,758 (87.7%)<br>2,204<br>4.16 (0.36)<br>4.20 (0.36)<br>18,046 (89.1%)<br>2,462<br>114.24 (37.72)<br>103.62 (37.72) | 18,100 (89.4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) | -0.04<br>-0.02<br>-0.00<br>0.04<br>-0.06<br>0.03<br>0.03 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only>0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)mean (sd)mean (sd)median [IQR]Missing; n (%) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98) | 2,577<br>140.14 (2.99)<br>140.00 (139.00, 142.00)<br>6,373 (71.2%)<br>2,243<br>4.18 (0.33)<br>4.20 (4.00, 4.40)<br>6,707 (74.9%)<br>2,565<br>113.73 (37.41) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04 | 154<br>139.54 (2.88)<br>140.00 (138.00, 141.00)<br>11,146 (98.6%)<br>112<br>4.01 (0.84)<br>4.20 (3.90, 4.40)<br>11,188 (99.0%)<br>153<br>126.15 (58.00) | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%)<br>146<br>4.12 (0.36)<br>4.10 [3.90, 4.40]<br>11,154 (98.7%)<br>186<br>126.78 (41.66) | 0.02<br>-0.14<br>0.00<br>0.02<br>-0.17<br>0.15<br>0.03 | N/A | N/A | #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) | -0.02<br>0.00<br>0.04<br>-0.06<br>0.03<br>0.03 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)median [IQR]median [IQR]median [IQR]median [IQR]Missing; n (%) Lab result number-Potassium mean (only 1-7 | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%) | 2,577<br>140.14 (2.99)<br>140.00 [139.00, 142.00]<br>6,373 (71.2%)<br>2,243<br>4.18 (0.33)<br>4.20 [4.00, 4.40]<br>6,707 (74.9%)<br>2,565<br>113.73 (37.41)<br>103.00 [93.00, 122.50]<br>6,385 (71.3%) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04 | 154 139.54 (2.88) 140.00 (138.00, 141.00) 11,146 (98.6%) 112 4.01 (0.84) 4.20 (3.90, 4.40) 11,188 (99.0%) 153 126.15 (58.00) 113.00 [95.00, 135.00] 11,147 (98.6%) | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%)<br>146<br>4.12 (0.36)<br>4.10 [3.90, 4.40]<br>11,154 (98.7%)<br>186<br>126.78 (41.66)<br>116.00 [100.00, 142.00]<br>11,114 (98.4%) | 0.02<br>-0.14<br>0.00<br>0.02<br>-0.17<br>0.15<br>0.03 | N/A | N/A | #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 17,788 (87.8%) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 17,499 (86.4%) | -0.02<br>0.00<br>0.04<br>-0.06<br>0.03<br>0.03 |
| median [IQR]Missing; n (%) Lab result number- Albumin mean (only >0 and <=10 included)mean (sq)median [IQR]Missing; n (%) Lab result number- Glucose (fasting or random) mean (only 10-1000 included)mean (sq)median [IQR]Missing; n (%) Lab result number- Potassium mean (only 1-7 included) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403 | 2,577<br>140.14 (2.99)<br>140.00 [139.00, 142.00]<br>6,373 (71.2%)<br>2,243<br>4.18 (0.33)<br>4.20 [4.00, 4.40]<br>6,707 (74.9%)<br>2,565<br>113.73 (37.41)<br>103.00 [93.00, 122.50]<br>6,385 (71.3%) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.07 | 154 139.54 (2.88) 140.00 (138.00, 141.00) 11,146 (98.6%) 112 4.01 (0.84) 4.20 (3.90, 4.40) 11,188 (99.0%) 153 126.15 (58.00) 113.00 (95.00, 135.00) 11,147 (98.6%) | 188<br>139.92 (2.69)<br>140.00 [138.00, 142.00]<br>11,112 (98.3%)<br>146<br>4.12 (0.36)<br>4.10 (3.90, 4.40)<br>11,154 (98.7%)<br>186<br>126.78 (41.66)<br>116.00 [100.00, 142.00]<br>11,114 (98.4%) | 0.02<br>-0.14<br>0.00<br>0.02<br>-0.17<br>0.15<br>0.03<br>-0.01<br>-0.06<br>0.02 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 | -0.02<br>0.00<br>0.04<br>-0.06<br>0.03<br>0.03<br>-0.01<br>-0.01 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only>0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)mean (sd)mean (sd) Lab result number-Potassium mean (only 1-7 included) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403<br>4.37 (0.43) | 2,577 140.14 (2.99) 140.00 [139.00, 142.00] 6,373 (71.2%) 2,243 4.18 (0.33) 4.20 [4.00, 4.40] 6,707 (74.9%) 2,565 113.73 (37.41) 103.00 [93.00, 122.50] 6,385 (71.3%) 2,703 4.37 (0.46) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.07 | 154 139.54 (2.88) 140.00 (138.00,141.00) 11,146 (98.6%) 112 4.01 (0.84) 4.20 (3.90, 4.40) 11,188 (99.0%) 153 126.15 (58.00) 113.00 [95.00, 135.00] 11,147 (98.6%) 159 4.36 (0.45) | 188 139.92 (2.69) 140.00 [138.00, 142.00] 11,112 (98.3%) 146 4.12 (0.36) 4.10 [3.90, 4.40] 11,154 (98.7%) 186 126.78 (41.66) 116.00 [100.00, 142.00] 11,114 (98.4%) 203 4.36 (0.43) | 0.02<br>-0.14<br>0.00<br>0.02<br>-0.17<br>0.15<br>0.03<br>-0.01<br>-0.06<br>0.02 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 4.37 (0.43) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 4.37 (0.46) | -0.02<br>0.00<br>0.04<br>-0.06<br>0.03<br>0.03<br>-0.01<br>-0.01<br>0.04 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)median [IQR]median [IQR]median [IQR]Missing; n (%) Lab result number- Potassium mean (only 1-7 included)mean (sd)mean (sd)mean (sd)mean (sd) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403<br>4.37 (0.43)<br>4.40 [4.10, 4.60] | 2,577 140.14 (2.99) 140.00 [139.00, 142.00] 6,373 (71.2%) 2,243 4.18 (0.33) 4.20 [4.00, 4.40] 6,707 (74.9%) 2,565 113.73 (37.41) 103.00 [93.00, 122.50] 6,385 (71.3%) 2,703 4.37 (0.46) 4.40 [4.10, 4.60] | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.07 | 154 139.54 (2.88) 140.00 [138.00, 141.00] 11,146 [98.6%) 112 4.01 (0.84) 4.20 [3.90, 4.40] 11,188 (99.0%) 126.15 (58.00) 113.00 [95.00, 135.00] 11,147 (98.6%) 159 4.36 (0.45) 4.30 [4.10, 4.60] | 188 139.92 (2.69) 140.00 [138.00, 142.00] 11,112 (98.3%) 146 4.12 (0.36) 4.10 (3.90, 4.40) 11,154 (98.7%) 186 126.78 (41.66) 116.00 [100.00, 142.00] 11,114 (98.4%) 203 4.36 (0.43) 4.37 [4.10, 4.70] | 0.02 -0.14 0.00 0.02 -0.17 0.15 0.03 -0.01 -0.06 0.02 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 4.37 (0.43) 4.39 (0.43) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 4.37 (0.46) 4.40 (0.46) | -0.04 -0.02 0.00 0.04 -0.06 0.03 0.03 -0.01 -0.01 0.04 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Potassium mean (only 1-7 included)mean (sd)median [IQR]mean (sd)median [IQR]mean (sd) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403<br>4.37 (0.43) | 2,577 140.14 (2.99) 140.00 [139.00, 142.00] 6,373 (71.2%) 2,243 4.18 (0.33) 4.20 [4.00, 4.40] 6,707 (74.9%) 2,565 113.73 (37.41) 103.00 [93.00, 122.50] 6,385 (71.3%) 2,703 4.37 (0.46) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.07 | 154 139.54 (2.88) 140.00 (138.00,141.00) 11,146 (98.6%) 112 4.01 (0.84) 4.20 (3.90, 4.40) 11,188 (99.0%) 153 126.15 (58.00) 113.00 [95.00, 135.00] 11,147 (98.6%) 159 4.36 (0.45) | 188 139.92 (2.69) 140.00 [138.00, 142.00] 11,112 (98.3%) 146 4.12 (0.36) 4.10 [3.90, 4.40] 11,154 (98.7%) 186 126.78 (41.66) 116.00 [100.00, 142.00] 11,114 (98.4%) 203 4.36 (0.43) | 0.02<br>-0.14<br>0.00<br>0.02<br>-0.17<br>0.15<br>0.03<br>-0.01<br>-0.06<br>0.02 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 4.37 (0.43) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 4.37 (0.46) | -0.02<br>0.00<br>0.04<br>-0.06<br>0.03<br>0.03<br>-0.01<br>-0.01<br>0.04 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Potassium mean (only 1-7 included)median [IQR]median [IQR]median [IQR]median [IQR]median [IQR]median [IQR] | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403<br>4.37 (0.43)<br>4.40 [4.10, 4.60] | 2,577 140.14 (2.99) 140.00 [139.00, 142.00] 6,373 (71.2%) 2,243 4.18 (0.33) 4.20 [4.00, 4.40] 6,707 (74.9%) 2,565 113.73 (37.41) 103.00 [93.00, 122.50] 6,385 (71.3%) 2,703 4.37 (0.46) 4.40 [4.10, 4.60] | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.07 | 154 139.54 (2.88) 140.00 [138.00, 141.00] 11,146 [98.6%) 112 4.01 (0.84) 4.20 [3.90, 4.40] 11,188 (99.0%) 126.15 (58.00) 113.00 [95.00, 135.00] 11,147 (98.6%) 159 4.36 (0.45) 4.30 [4.10, 4.60] | 188 139.92 (2.69) 140.00 [138.00, 142.00] 11,112 (98.3%) 146 4.12 (0.36) 4.10 (3.90, 4.40) 11,154 (98.7%) 186 126.78 (41.66) 116.00 [100.00, 142.00] 11,114 (98.4%) 203 4.36 (0.43) 4.37 [4.10, 4.70] | 0.02 -0.14 0.00 0.02 -0.17 0.15 0.03 -0.01 -0.06 0.02 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 4.37 (0.43) 4.39 (0.43) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 4.37 (0.46) 4.40 (0.46) | -0.04 -0.02 0.00 0.04 -0.06 0.03 0.03 -0.01 -0.01 0.04 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Potassium mean (only 1-7 included)mean (sd)median [IQR]mean (sd)median [IQR]mean (sd) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403<br>4.37 (0.43)<br>4.40 [4.10, 4.60] | 2,577 140.14 (2.99) 140.00 [139.00, 142.00] 6,373 (71.2%) 2,243 4.18 (0.33) 4.20 [4.00, 4.40] 6,707 (74.9%) 2,565 113.73 (37.41) 103.00 [93.00, 122.50] 6,385 (71.3%) 2,703 4.37 (0.46) 4.40 [4.10, 4.60] | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.07 | 154 139.54 (2.88) 140.00 [138.00, 141.00] 11,146 [98.6%) 112 4.01 (0.84) 4.20 [3.90, 4.40] 11,188 (99.0%) 126.15 (58.00) 113.00 [95.00, 135.00] 11,147 (98.6%) 159 4.36 (0.45) 4.30 [4.10, 4.60] | 188 139.92 (2.69) 140.00 [138.00, 142.00] 11,112 (98.3%) 146 4.12 (0.36) 4.10 (3.90, 4.40) 11,154 (98.7%) 186 126.78 (41.66) 116.00 [100.00, 142.00] 11,114 (98.4%) 203 4.36 (0.43) 4.37 [4.10, 4.70] | 0.02 -0.14 0.00 0.02 -0.17 0.15 0.03 -0.01 -0.06 0.02 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 4.37 (0.43) 4.39 (0.43) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 4.37 (0.46) 4.40 (0.46) | -0.04 -0.02 0.00 0.04 -0.06 0.03 0.03 -0.01 -0.01 0.04 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Potassium mean (only 1-7 included)median [IQR]median [IQR]median [IQR]median [IQR]median [IQR]median [IQR] | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403<br>4.37 (0.43)<br>4.40 [4.10, 4.60] | 2,577 140.14 (2.99) 140.00 [139.00, 142.00] 6,373 (71.2%) 2,243 4.18 (0.33) 4.20 [4.00, 4.0] 6,707 (74.9%) 2,565 113.73 (37.41) 103.00 [93.00, 122.50] 6,385 (71.3%) 2,703 4.37 (0.46) 4.40 [4.10, 4.60] 6,247 (69.8%) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.07 | 154 139.54 (2.88) 140.00 [138.00, 141.00] 11,146 [98.6%) 112 4.01 (0.84) 4.20 [3.90, 4.40] 11,188 (99.0%) 126.15 (58.00) 113.00 [95.00, 135.00] 11,147 (98.6%) 159 4.36 (0.45) 4.30 [4.10, 4.60] | 188 139.92 (2.69) 140.00 [138.00, 142.00] 11,112 (98.3%) 146 4.12 (0.36) 4.10 (3.90, 4.40) 11,154 (98.7%) 186 126.78 (41.66) 116.00 [100.00, 142.00] 11,114 (98.4%) 203 4.36 (0.43) 4.37 [4.10, 4.70] | 0.02 -0.14 0.00 0.02 -0.17 0.15 0.03 -0.01 -0.06 0.02 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 4.37 (0.43) 4.39 (0.43) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 4.37 (0.46) 4.40 (0.46) | -0.04 -0.02 0.00 0.04 -0.06 0.03 0.03 -0.01 -0.01 0.04 |
| median [IQR]Missing; n (%) Lab result number- Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number- Glucose (fasting or random) mean (only 10-1000 included)median [IQR]median [IQR]missing; n (%) Lab result number- Potassium mean (only 1-7 included)mean (sd)mean (sd)median [IQR]Missing; n (%) Comorbidity Scores CCI (180 days)- ICD9 and ICD10 v2mean (sd) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.3.2)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403<br>4.37 (0.43)<br>4.40 [4.10, 4.60]<br>6,547 (73.2%) | 2,577 140.14 (2.99) 140.00 [139.00, 142.00] 6,373 (71.2%) 2,243 4.18 (0.33) 4.20 [4.00, 4.40] 6,707 (74.9%) 2,565 113.73 (37.41) 103.00 [93.00, 122.50] 6,385 (71.3%) 2,703 4.37 (0.46) 4.40 [4.10, 4.60] 6,247 (69.8%) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.07 | 154 139.54 (2.88) 140.00 (138.00, 141.00) 11,146 (98.6%) 112 4.01 (0.84) 4.20 (3.90, 4.40) 11,188 (99.0%) 153 126.15 (58.00) 113.00 (95.00, 135.00) 11,147 (98.6%) 4.36 (0.45) 4.30 (4.10, 4.60) 11,141 (98.6%) 3.15 (1.62) | 188 139.92 (2.69) 140.00 [138.00, 142.00] 11,112 [98.3%) 146 4.12 (0.36) 4.10 [3.90, 4.40] 11,154 (98.7%) 186 126.78 (41.66) 116.00 [100.00, 142.00] 11,114 (98.4%) 203 4.36 (0.43) 4.37 [4.10, 4.70] 11,097 (98.2%) | 0.02 -0.14 0.00 0.02 -0.17 0.15 0.03 -0.01 -0.06 0.02 -0.00 -0.16 0.03 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 4.37 (0.43) 4.39 (0.43) 17,688 (87.3%) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 4.37 (0.46) 4.40 (0.46) 17,344 (85.6%) | -0.02<br>0.00<br>0.04<br>-0.06<br>0.03<br>0.03<br>-0.01<br>-0.01<br>0.04<br>-0.00<br>-0.02<br>0.05 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Potassium mean (only 1-7 included)mean (sd)median [IQR]Missing; n (%) Comorbidity Scores CCI (180 days)-ICD9 and ICD10 v2mean (sd)median [IQR] | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403<br>4.37 (0.43)<br>4.40 [4.10, 4.60]<br>6,547 (73.2%) | 2,577 140.14 (2.99) 140.00 (139.00, 142.00) 6,373 (71.2%) 2,243 4.18 (0.33) 4.20 (4.00, 4.01) 6,707 (74.9%) 2,565 113.73 (37.41) 103.00 [93.00, 122.50] 6,385 (71.3%) 2,703 4.37 (0.46) 4.40 (4.10, 4.60] 6,247 (69.8%) 3.48 (1.74) 3.00 (2.00, 5.00) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.07 | 154 139.54 (2.88) 140.00 (138.00, 141.00) 11,146 (98.6%) 112 4.01 (0.84) 4.20 (3.90, 4.40) 11,188 (99.0%) 153 126.15 (58.00) 113.00 (95.00, 135.00) 11,147 (98.6%) 4.36 (0.45) 4.36 (0.45) 4.30 (4.10, 4.60) 11,141 (98.6%) 3.15 (1.62) 3.00 (2.00, 4.00) | 188 139.92 (2.69) 140.00 [138.00, 142.00] 11,112 (98.3%) 146 4.12 (0.36) 4.10 (3.90, 4.40) 11,154 (98.7%) 186 126.78 (41.66) 116.00 [100.00, 142.00] 11,114 (98.4%) 203 4.36 (0.43) 4.37 [4.10, 4.70] 11,097 (98.2%) 3.13 (1.62) 3.00 [2.00, 4.00] | 0.02 -0.14 0.00 0.02 -0.17 0.15 0.03 -0.01 -0.06 0.02 -0.00 -0.16 0.03 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 4.37 (0.43) 4.39 (0.43) 17,688 (87.3%) 3.07 (1.93) 3.00 (1.93) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 4.37 (0.46) 4.40 (0.46) 17,344 (85.6%) 3.06 (1.94) 3.00 (1.94) | 0.04 -0.02 0.00 0.04 -0.06 0.03 0.03 -0.01 -0.01 0.04 0.00 -0.02 0.05 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)median [IQR]median [IQR]Missing; n (%) Lab result number-Potassium mean (only 1-7 included)mean (sd)mean (sd)mean (sd)median [IQR]Missing; n (%) Comorbidity Scores CCI (180 days)-ICD9 and ICD10 v2mean (sd)mean (sd)median [IQR] Non-Frailty; n (%) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.3.2)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403<br>4.37 (0.43)<br>4.40 [4.10, 4.60]<br>6,547 (73.2%) | 2,577 140.14 (2.99) 140.00 [139.00, 142.00] 6,373 (71.2%) 2,243 4.18 (0.33) 4.20 [4.00, 4.40] 6,707 (74.9%) 2,565 113.73 (37.41) 103.00 [93.00, 122.50] 6,385 (71.3%) 2,703 4.37 (0.46) 4.40 [4.10, 4.60] 6,247 (69.8%) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.07 | 154 139.54 (2.88) 140.00 (138.00, 141.00) 11,146 (98.6%) 112 4.01 (0.84) 4.20 (3.90, 4.40) 11,188 (99.0%) 153 126.15 (58.00) 113.00 (95.00, 135.00) 11,147 (98.6%) 4.36 (0.45) 4.30 (4.10, 4.60) 11,141 (98.6%) 3.15 (1.62) | 188 139.92 (2.69) 140.00 [138.00, 142.00] 11,112 [98.3%) 146 4.12 (0.36) 4.10 [3.90, 4.40] 11,154 (98.7%) 186 126.78 (41.66) 116.00 [100.00, 142.00] 11,114 (98.4%) 203 4.36 (0.43) 4.37 [4.10, 4.70] 11,097 (98.2%) | 0.02 -0.14 0.00 0.02 -0.17 0.15 0.03 -0.01 -0.06 0.02 -0.00 -0.16 0.03 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 4.37 (0.43) 4.39 (0.43) 17,688 (87.3%) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 4.37 (0.46) 4.40 (0.46) 17,344 (85.6%) | 0.04 -0.02 0.00 0.04 -0.06 0.03 0.03 -0.01 -0.01 0.04 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)median [IQR]median [IQR]missing; n (%) Lab result number-Potassium mean (only 1-7 included)mean (sd)median [IQR]Missing; n (%) Comorbidity Scores CCI (180 days)-ICD9 and ICD10 v2median [IQR]median [IQR] Non-Frailty; n (%) Frailty Score (mean): Empirical Version 365 days, v2 | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403<br>4.37 (0.43)<br>4.40 [4.10, 4.60]<br>6,547 (73.2%)<br>3.47 (1.71)<br>3.00 [2.00, 5.00]<br>4,818 (53.8%) | 2,577 140.14 (2.99) 140.00 [139.00, 142.00] 6,373 (71.2%) 2,243 4.18 (0.33) 4.20 [4.00, 4.0] 6,707 (74.9%) 2,565 113.73 (37.41) 103.00 [93.00, 122.50] 6,385 (71.3%) 2,703 4.37 (0.46) 4.40 [4.10, 4.60] 6,247 (69.8%) 3.48 (1.74) 3.00 [2.00, 5.00] 4,943 (55.2%) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.00<br>0.08 | 154 139.54 (2.88) 140.00 (138.00, 141.00) 11,146 (98.6%) 112 4.01 (0.84) 4.20 (3.90, 4.40) 11,188 (99.0%) 153 126.15 (58.00) 113.00 [95.00, 135.00] 11,147 (98.6%) 159 4.36 (0.45) 4.30 (4.10, 4.60) 11,141 (98.6%) 3.15 (1.62) 3.00 (2.00, 4.00] 5,684 (50.3%) | 188 139.92 (2.69) 140.00 [138.00, 142.00] 11,112 [98.3%) 146 4.12 (0.36) 4.10 [3.90, 4.40] 11,154 [98.7%) 186 126.78 (41.66) 116.00 [100.00, 142.00] 11,114 (98.4%) 203 4.36 (0.43) 4.37 [4.10, 4.70] 11,097 (98.2%) 3.13 (1.62) 3.00 [2.00, 4.00] 5,645 (50.0%) | 0.02 -0.14 0.00 0.02 -0.17 0.15 0.03 -0.01 -0.06 0.02 0.00 -0.16 0.03 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 4.37 (0.43) 4.39 (0.43) 17,688 (87.3%) 3.07 (1.93) 3.00 (1.93) 11,336 (22.1%) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 4.37 (0.46) 4.40 (0.46) 17,344 (85.6%) 3.06 (1.94) 3.00 (1.94) 11,285 (22.0%) | 0.04 -0.02 0.00 0.04 -0.06 0.03 0.03 -0.01 -0.01 0.04 -0.02 0.05 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)median [IQR]median [IQR]Missing; n (%) Lab result number-Potassium mean (only 1-7 included)mean (sd)mean (sd)mean (sd)median [IQR]Missing; n (%) Comorbidity Scores CCI (180 days)-ICD9 and ICD10 v2mean (sd)mean (sd)median [IQR] Non-Frailty; n (%) | 140.09 (3.01)<br>140.00 [138.50, 142.00]<br>6,612 (73.9%)<br>2,092<br>4.17 (0.32)<br>4.20 [4.00, 4.40]<br>6,858 (76.6%)<br>2,309<br>113.45 (35.98)<br>103.00 [93.00, 121.00]<br>6,641 (74.2%)<br>2,403<br>4.37 (0.43)<br>4.40 [4.10, 4.60]<br>6,547 (73.2%) | 2,577 140.14 (2.99) 140.00 (139.00, 142.00) 6,373 (71.2%) 2,243 4.18 (0.33) 4.20 (4.00, 4.01) 6,707 (74.9%) 2,565 113.73 (37.41) 103.00 [93.00, 122.50] 6,385 (71.3%) 2,703 4.37 (0.46) 4.40 (4.10, 4.60] 6,247 (69.8%) 3.48 (1.74) 3.00 (2.00, 5.00) | -0.02<br>0.00<br>0.06<br>-0.03<br>0.00<br>0.04<br>-0.01<br>0.00<br>0.07 | 154 139.54 (2.88) 140.00 (138.00, 141.00) 11,146 (98.6%) 112 4.01 (0.84) 4.20 (3.90, 4.40) 11,188 (99.0%) 153 126.15 (58.00) 113.00 (95.00, 135.00) 11,147 (98.6%) 4.36 (0.45) 4.36 (0.45) 4.30 (4.10, 4.60) 11,141 (98.6%) 3.15 (1.62) 3.00 (2.00, 4.00) | 188 139.92 (2.69) 140.00 [138.00, 142.00] 11,112 (98.3%) 146 4.12 (0.36) 4.10 (3.90, 4.40) 11,154 (98.7%) 186 126.78 (41.66) 116.00 [100.00, 142.00] 11,114 (98.4%) 203 4.36 (0.43) 4.37 [4.10, 4.70] 11,097 (98.2%) 3.13 (1.62) 3.00 [2.00, 4.00] | 0.02 -0.14 0.00 0.02 -0.17 0.15 0.03 -0.01 -0.06 0.02 -0.00 -0.16 0.03 | N/A | N/A | #VALUEI | 18,351 (90.6%) 2,492 140.06 (3.00) 140.00 (3.00) 17,758 (87.7%) 2,204 4.16 (0.36) 4.20 (0.36) 18,046 (89.1%) 2,462 114.24 (37.72) 103.62 (37.72) 103.62 (37.72) 17,788 (87.8%) 2,562 4.37 (0.43) 4.39 (0.43) 17,688 (87.3%) 3.07 (1.93) 3.00 (1.93) | 18,100 (89,4%) 2,765 140.13 (2.97) 140.00 (2.97) 17,485 (86.3%) 2,389 4.18 (0.33) 4.19 (0.33) 17,861 (88.2%) 2,751 114.61 (37.72) 103.88 (37.72) 103.88 (37.72) 17,499 (86.4%) 2,906 4.37 (0.46) 4.40 (0.46) 17,344 (85.6%) 3.06 (1.94) 3.00 (1.94) | 0.04 -0.02 0.00 0.04 -0.06 0.03 0.03 -0.01 -0.01 0.04 0.00 -0.02 0.05 |

| Healthcare Utilization | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Any hospitalization; n (%) | 2,257 (25.2%) | 2,314 (25.9%) | -0.02 | 3,579 (31.7%) | 3,582 (31.7%) | 0.00 | 15,976 (51.4%) | 15,922 (51.2%) | 0.00 | 21,812 (42.5%) | 21,818 (42.5%) | 0.00 |
| Any hospitalization within prior 30 days; n (%) | 1,520 (17.0%) | 1,514 (16.9%) | 0.00 | 2,456 (21.7%) | 2,479 (21.9%) | 0.00 | 11,249 (36.2%) | 11,049 (35.6%) | 0.01 | 15225 (29.7%) | 15042 (29.3%) | 0.01 |
| Any hospitalization during prior 31-180 days; n (%) | 866 (9.7%) | 932 (10.4%) | -0.02 | 1,279 (11.3%) | 1,268 (11.2%) | 0.00 | 6,194 (19.9%) | 6,196 (19.9%) | 0.00 | 8339 (16.2%) | 8396 (16.4%) | -0.01 |
| Endocrinologist Visit; n (%) | 286 (3.2%) | 266 (3.0%) | 0.01 | 424 (3.8%) | 440 (3.9%) | -0.01 | 1,662 (5.3%) | 1,637 (5.3%) | 0.00 | 2372 (4.6%) | 2343 (4.6%) | 0.00 |
| Endocrinologist Visit (30 days prior); n (%) | 101 (1.1%) | 81 (0.9%) | 0.02 | 153 (1.4%) | 150 (1.3%) | 0.01 | 557 (1.8%) | 540 (1.7%) | 0.01 | 811 (1.6%) | 771 (1.5%) | 0.01 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 232 (2.6%) | 224 (2.5%) | 0.01 | 361 (3.2%) | 372 (3.3%) | -0.01 | 1,406 (4.5%) | 1,384 (4.5%) | 0.00 | 1999 (3.9%) | 1980 (3.9%) | 0.00 |
| Internal medicine/family medicine visits; n (%) | 7,789 (87.0%) | 7,872 (88.0%) | -0.03 | 9,294 (82.2%) | 9,180 (81.2%) | 0.03 | 27,136 (87.3%) | 27,571 (88.7%) | -0.04 | 44219 (86.2%) | 44623 (87.0%) | -0.02 |
| Internal medicine/family medicine visits (30 days | | | | | | | | | | | | |
| prior) v2; n (%) | 5,509 (61.6%) | 5,525 (61.7%) | 0.00 | 6,399 (56.6%) | 6,455 (57.1%) | -0.01 | 20,182 (65.0%) | 20,407 (65.7%) | -0.01 | 32090 (62.5%) | 32387 (63.1%) | -0.01 |
| Internal medicine/family medicine visits (31 to 180 | | | | | | | | | | | | |
| days prior) v2; n (%) | 6,784 (75.8%) | 6,904 (77.1%) | -0.03 | 8,254 (73.0%) | 8,060 (71.3%) | 0.04 | 23,086 (74.3%) | 23,526 (75.7%) | -0.03 | 38124 (74.3%) | 38490 (75.0%) | -0.02 |
| Cardiologist visit; n (%) | 6,799 (76.0%) | 6,934 (77.5%) | -0.04 | 6,695 (59.2%) | 6,471 (57.3%) | 0.04 | 26,281 (84.6%) | 26,471 (85.2%) | -0.02 | 39775 (77.5%) | 39876 (77.7%) | 0.00 |
| Number of Cardiologist visits (30 days prior); n (%) | 5,531 (61.8%) | 5,397 (60.3%) | 0.03 | 4,970 (44.0%) | 4,973 (44.0%) | 0.00 | 21,163 (68.1%) | 20,800 (66.9%) | 0.03 | 31664 (61.7%) | 31170 (60.7%) | 0.02 |
| Number of Cardiologist visits (31 to 180 days prior); | 4 400 (46 00/) | 4,233 (47.3%) | -0.01 | 4,502 (39.8%) | 4,157 (36.8%) | 0.06 | 16,385 (52.7%) | 16,402 (52.8%) | 0.00 | 25076 (48.9%) | 24792 (48.3%) | 0.01 |
| n (%)<br>Electrocardiogram v2; n (%) | 4,189 (46.8%)<br>6,802 (76.0%) | 7,027 (78.5%) | -0.01 | 4,502 (39.8%)<br>8,084 (71.5%) | 4,157 (36.8%)<br>8,613 (76.2%) | -0.11 | 26,290 (84.6%) | 26,741 (86.1%) | -0.04 | 41176 (80.2%) | 42381 (82.6%) | -0.06 |
| Use of glucose test strips; n (%) | 109 (1.2%) | 124 (1.4%) | -0.02 | 114 (1.0%) | 136 (1.2%) | -0.11 | 685 (2.2%) | 746 (2.4%) | -0.04 | 908 (1.8%) | 1006 (2.0%) | -0.06 |
| Dialysis; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 003 (2.2%) | /40 (2.4%) | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| number of different/distinct medication | 0 (0.0%) | 0 (0.0%) | #DIV/0: | 0 (0.0%) | 0 (0.0%) | #510/0: | | | #VALUE: | #VALUE: | #VALUE: | #VALUE: |
| prescriptions | | | | | | | | | | | | |
| mean (sd) | 9.41 (4.42) | 9.45 (4.50) | -0.01 | 9.77 (4.56) | 9.76 (4.56) | 0.00 | 10.93 (4.76) | 10.95 (4.85) | 0.00 | 10.41 (4.66) | 10.43 (4.73) | 0.00 |
| median [IQR] | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 0.00 | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | 0.00 | 10.00 [8.00, 14.00] | 10.00 [8.00, 14.00] | 0.00 | 5.75 (5.45) | 5.75 (5.51) | 0.00 |
| Number of Hospitalizations | 3.00 [0.00, 12.00] | 3.00 (0.00, 12.00) | 0.00 | 3.00 (7.00, 12.00) | 3.00 [7.00, 12.00] | 0.00 | 10.00 [0.00, 11.00] | 10.00 (0.00, 11.00) | 0.00 | 3.73 (3.13) | 3.73 (3.31) | 0.00 |
| mean (sd) | 0.29 (0.55) | 0.29 (0.54) | 0.00 | 0.35 (0.54) | 0.35 (0.55) | 0.00 | 0.65 (0.76) | 0.64 (0.76) | 0.01 | 0.52 (0.68) | 0.52 (0.68) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 0.22 (0.76) | 0.22 (0.76) | 0.00 |
| Number of hospital days | | | | | | | | | | ` , | , , | |
| mean (sd) | 1.34 (3.03) | 1.35 (3.73) | 0.00 | 1.66 (3.30) | 1.62 (3.81) | 0.01 | 3.67 (5.72) | 3.57 (7.18) | 0.02 | 2.82 (4.88) | 2.75 (6.07) | 0.01 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 3.00] | 0.00 [0.00, 3.00] | 0.00 | 2.00 [0.00, 5.00] | 2.00 [0.00, 5.00] | 0.00 | 0.44 (5.29) | 0.44 (6.51) | 0.00 |
| Number of Emergency Department (ED) visits v3 | | | | | | | | | | | | |
| mean (sd) | 0.74 (1.32) | 0.75 (1.35) | -0.01 | 0.64 (2.28) | 0.63 (2.03) | 0.00 | 1.31 (1.95) | 1.31 (1.82) | 0.00 | 1.06 (1.94) | 1.06 (1.80) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 0.22 (2.40) | 0.22 (2.20) | 0.00 |
| Number of Office visits | | | | | | | | | | | | |
| mean (sd) | 5.46 (4.17) | 5.47 (3.88) | 0.00 | 5.89 (4.44) | 5.82 (4.17) | 0.02 | 13.22 (13.02) | 13.19 (12.41) | 0.00 | 10.25 (10.49) | 10.22 (9.98) | 0.00 |
| median [IQR] | 5.00 [3.00, 7.00] | 5.00 [3.00, 7.00] | 0.00 | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | 0.00 | 10.00 [5.00, 17.00] | 10.00 [5.00, 17.75] | 0.00 | 4.17 (10.84) | 4.17 (10.31) | 0.00 |
| Number of Endocrinologist visits | | | | | | | | | | | | |
| mean (sd) | 0.13 (1.20) | 0.11 (0.94) | 0.02 | 0.15 (1.19) | 0.16 (1.21) | -0.01 | 0.26 (1.91) | 0.25 (1.78) | 0.01 | 0.21 (1.66) | 0.21 (1.55) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.82) | 0.00 (1.72) | 0.00 |
| Number of internal medicine/family medicine visits | | | | | | | | | | | | |
| mean (sd) | 9.10 (11.33) | 9.29 (12.40) | -0.02 | 7.60 (11.04) | 7.50 (10.85) | 0.01 | 9.55 (10.63) | 9.49 (10.61) | 0.01 | 9.04 (10.85) | 9.02 (10.99) | 0.00 |
| median [IQR] | 6.00 [2.00, 12.00] | 6.00 [2.00, 12.00] | 0.00 | 4.00 [1.00, 9.00] | 4.00 [1.00, 9.00] | 0.00 | 7.00 [2.00, 13.00] | 7.00 [3.00, 13.00] | 0.00 | 3.47 (12.83) | 3.47 (12.89) | 0.00 |
| Number of Cardiologist visits | | | | | | | | | | | | |
| mean (sd) | 4.73 (5.69) | 4.68 (5.48) | 0.01 | 3.10 (4.72) | 3.09 (4.65) | 0.00 | 6.14 (7.31) | 6.06 (6.74) | 0.01 | 5.22 (6.55) | 5.17 (6.12) | 0.01 |
| median [IQR] | 3.00 [1.00, 7.00] | 3.00 [1.00, 7.00] | 0.00 | 1.00 [0.00, 4.00] | 1.00 [0.00, 4.00] | 0.00 | 4.00 [1.00, 8.00] | 4.00 [2.00, 8.00] | 0.00 | 1.62 (7.18) | 1.62 (6.77) | 0.00 |
| Number electrocardiograms received v2 | | | | | | | | | | | | |
| mean (sd) | 2.14 (2.51) | 2.15 (2.32) | 0.00 | 1.78 (2.15) | 1.77 (1.83) | 0.01 | 2.70 (2.61) | 2.69 (2.43) | 0.00 | 2.40 (2.50) | 2.39 (2.29) | 0.00 |
| median [IQR] | 1.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | -0.41 | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | 0.00 | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.00 | 0.83 (2.83) | 1.01 (2.56) | -0.07 |
| Number of HbA1c tests ordered | | | | | | | | / / | | | | |
| mean (sd) | 0.46 (0.73) | 0.46 (0.72) | 0.00 | 0.21 (0.54) | 0.22 (0.55) | -0.02 | 0.57 (0.81) | 0.57 (0.80) | 0.00 | 0.47 (0.74) | 0.47 (0.74) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (0.82) | 0.00 (0.81) | 0.00 |
| Number of glucose tests ordered | 0.04 (0.04) | 0.40 (0.00) | | 0.40 (0.64) | 0.4.4 (0.00) | | 0.00(4.05) | 0.00 (0.70) | | 0.00 (4.50) | 0.00 (0.70) | |
| mean (sd) | 0.21 (2.91) | 0.19 (0.82) | 0.01 | 0.13 (0.61) | 0.14 (0.89) | -0.01 | 0.22 (1.26) | 0.22 (0.72) | 0.00 | 0.20 (1.59) | 0.20 (0.78) | 0.00 |
| median [IQR] Number of lipid tests ordered | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.63) | 0.00 (0.95) | 0.00 |
| mean (sd) | 0.66 (0.84) | 0.65 (0.79) | 0.01 | 0.29 (0.74) | 0.30 (0.70) | -0.01 | 0.69 (0.77) | 0.69 (0.78) | 0.00 | 0.60 (0.78) | 0.60 (0.76) | 0.00 |
| () | , , | . , | | | | | . , | , , | | | , , | 0.00 |
| median [IQR] Number of creatinine tests ordered | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 0.22 (0.90) | 0.22 (0.88) | 0.00 |
| mean (sd) | 0.07 (0.36) | 0.07 (0.32) | 0.00 | 0.05 (0.32) | 0.05 (0.29) | 0.00 | 0.12 (0.45) | 0.11 (0.43) | 0.02 | 0.10 (0.41) | 0.09 (0.39) | 0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.02 | 0.00 (0.41) | 0.00 (0.43) | 0.02 |
| Number of BUN tests ordered | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 3.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.40) | 0.00 (0.43) | 0.00 |
| mean (sd) | 0.04 (0.28) | 0.04 (0.24) | 0.00 | 0.03 (0.25) | 0.03 (0.23) | 0.00 | 0.08 (0.37) | 0.07 (0.33) | 0.03 | 0.06 (0.33) | 0.06 (0.30) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.33) | 0.00 (0.33) | 0.00 |
| Number of tests for microal burninuria | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 5.00 | 0.00 (0.37) | 0.00 (0.33) | 3.00 |
| mean (sd) | 0.22 (0.66) | 0.22 (0.66) | 0.00 | 0.09 (0.43) | 0.09 (0.41) | 0.00 | 0.17 (0.50) | 0.16 (0.47) | 0.02 | 0.16 (0.52) | 0.16 (0.50) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.58) | 0.00 (0.56) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | [,] | [,] | | [,] | , (,) | | (,) | [,] | **** | () | (0) | =-== |
| digit level Copy | | | | | | | | | | | | |
| mean (sd) | 7.69 (8.86) | 7.57 (8.88) | 0.01 | 3.87 (6.60) | 3.82 (6.57) | 0.01 | 11.49 (12.00) | 11.34 (12.10) | 0.01 | 9.15 (10.51) | 9.03 (10.58) | 0.01 |
| median [IQR] | 5.00 [0.00, 12.00] | 5.00 [0.00, 11.00] | 0.00 | 0.00 [0.00, 5.00] | 0.00 [0.00, 5.00] | 0.00 | 8.00 [0.00, 19.00] | 8.00 [0.00, 18.00] | 0.00 | 2.63 (11.28) | 2.63 (11.34) | 0.00 |

| For PS | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Hemorrhagic stroke+Other cerebrovascular | | | | | | | | | | | | |
| disease+Cerebrovascular procedure (for PS); n (%) | 381 (4.3%) | 367 (4.1%) | 0.01 | 377 (3.3%) | 377 (3.3%) | 0.00 | 1,762 (5.7%) | 1,706 (5.5%) | 0.01 | 2520 (4.9%) | 2450 (4.8%) | 0.00 |
| Occurrence of creatinine tests ordered (for PS); n (%) | 464 (5.2%) | 473 (5.3%) | 0.00 | 438 (3.9%) | 457 (4.0%) | -0.01 | 2,763 (8.9%) | 2,675 (8.6%) | 0.01 | 3665 (7.1%) | 3605 (7.0%) | 0.00 |
| Occurrence of BUN tests ordered (for PS); n (%) | 267 (3.0%) | 278 (3.1%) | -0.01 | 277 (2.5%) | 302 (2.7%) | -0.01 | 1,749 (5.6%) | 1,667 (5.4%) | 0.01 | 2293 (4.5%) | 2247 (4.4%) | 0.00 |
| Occurrence of chronic renal insufficiency w/o CKD | | | | =:: (=:07-) | ( /-/ | | _, (0, | _,, | | | () | |
| (for PS) v2; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 189 (0.6%) | 195 (0.6%) | 0.00 | 189 (0.4%) | 195 (0.4%) | 0.00 |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 | 0 | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Chronic kidney disease Stage 3-6 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 463 (1.5%) | 446 (1.4%) | 0.01 | 463 (0.9%) | 446 (0.9%) | 0.00 |
| Bladder stones+Kidney stones (for PS); n (%) | 84 (0.9%) | 97 (1.1%) | -0.02 | 122 (1.1%) | 126 (1.1%) | 0.00 | 487 (1.6%) | 494 (1.6%) | 0.00 | 693 (1.4%) | 717 (1.4%) | 0.00 |
| Diabetes with peripheral circulatory | | | | | | | | | | | | |
| disorders+Gangrene+Osteomyelitis(for PS) v3 with | 240 (2.6%) | 275 (2.40() | 0.03 | 204 (2.6%) | 204 (2 50() | 0.01 | 4 507 (5 40() | 4 (40 (5 20)) | 0.01 | 24.0.5 (4.20() | 2400 (4 20) | 0.00 |
| ICD10 Copy; n (%) | 318 (3.6%) | 275 (3.1%) | 0.03 | 291 (2.6%) | 284 (2.5%) | 0.01 | 1,587 (5.1%) | 1,640 (5.3%) | -0.01 | 2196 (4.3%) | 2199 (4.3%) | 0.00 |
| Alcohol abuse or dependence+Drug abuse or<br>dependence (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 95 (0.3%) | 84 (0.3%) | 0.00 | 95 (0.2%) | 84 (0.2%) | 0.00 |
| Diabetes with other ophthalmic | - (a.a., | - () | , | - () | - () | | | 0.(0.07-) | | 00 (0.2,-,) | () | |
| manifestations+Retinal detachment, vitreous | | | | | | | | | | | | |
| hemorrhage, vitrectomy+Retinal laser coagulation | | | | | | | | | | | | |
| therapy (for PS); n (%) | 42 (0.5%) | 46 (0.5%) | 0.00 | 174 (1.5%) | 156 (1.4%) | 0.01 | 458 (1.5%) | 465 (1.5%) | 0.00 | 674 (1.3%) | 667 (1.3%) | 0.00 |
| Other atherosclerosis+Cardiac conduction | | | | | | | | | | | | |
| disorders+Other CVD (for PS) v2 Copy; n (%) | 3,857 (43.1%) | 3,825 (42.7%) | 0.01 | 4,510 (39.9%) | 4,497 (39.8%) | 0.00 | 14,213 (45.7%) | 14,081 (45.3%) | 0.01 | 22580 (44.0%) | 22403 (43.7%) | 0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent) +<br>History of CABG or PTCA (for PS) v3; n (%) | 905 (10.1%) | 895 (10.0%) | 0.00 | 640 (5.7%) | 662 (5.9%) | -0.01 | 5,079 (16.3%) | 4,997 (16.1%) | 0.01 | 6624 (12.9%) | 6554 (12.8%) | 0.00 |
| Hyperthyroidism + Hypothyroidism + Other disorders | 903 (10.1%) | 895 (10.0%) | 0.00 | 640 (5.7%) | 002 (3.9%) | -0.01 | 3,079 (10.3%) | 4,997 (10.1%) | 0.01 | 0024 (12.9%) | 0554 (12.6%) | 0.00 |
| of thyroid gland (for PS); n (%) | 1,955 (21.8%) | 1,944 (21.7%) | 0.00 | 1,893 (16.8%) | 1,850 (16.4%) | 0.01 | 5,526 (17.8%) | 5,502 (17.7%) | 0.00 | 9374 (18.3%) | 9296 (18.1%) | 0.01 |
| Delirium + Psychosis (for PS); n (%) | 279 (3.1%) | 261 (2.9%) | 0.01 | 275 (2.4%) | 274 (2.4%) | 0.00 | 1,619 (5.2%) | 1,599 (5.1%) | 0.00 | 2173 (4.2%) | 2134 (4.2%) | 0.00 |
| Any use of Meglitinides (for PS); n (%) | 23 (0.3%) | 20 (0.2%) | 0.02 | 55 (0.5%) | 62 (0.5%) | 0.00 | 155 (0.5%) | 145 (0.5%) | 0.00 | 233 (0.5%) | 227 (0.4%) | 0.01 |
| Any use of AGIs (for PS); n (%) | 10 (0.1%) | 7 (0.1%) | 0.00 | 19 (0.2%) | 12 (0.1%) | 0.03 | 42 (0.1%) | 42 (0.1%) | 0.00 | 71 (0.1%) | 61 (0.1%) | 0.00 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 466 (1.5%) | 448 (1.4%) | 0.01 | 467 (0.9%) | 448 (0.9%) | 0.00 |
| Use of thiazide; n (%) | 1,119 (12.5%) | 1,137 (12.7%) | -0.01 | 1,374 (12.2%) | 1,344 (11.9%) | 0.01 | 4,321 (13.9%) | 4,262 (13.7%) | 0.01 | 6814 (13.3%) | 6743 (13.1%) | 0.01 |
| Use of beta blockers; n (%) | 6,279 (70.2%) | 6,292 (70.3%) | 0.00 | 8,046 (71.2%) | 7,986 (70.7%) | 0.01 | 23,273 (74.9%) | 23,216 (74.7%) | 0.00 | 37598 (73.3%) | 37494 (73.1%) | 0.00 |
| Use of calcium channel blockers; n (%) | 3,638 (40.6%) | 3,637 (40.6%) | 0.00 | 4,634 (41.0%) | 4,646 (41.1%) | 0.00 | 13,887 (44.7%) | 13,904 (44.8%) | 0.00 | 22159 (43.2%) | 22187 (43.2%) | 0.00 |
| All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy; n (%) | 2,126 (23.8%)<br>430 (4.8%) | 2,148 (24.0%)<br>441 (4.9%) | 0.00 | 2,739 (24.2%)<br>738 (6.5%) | 2,739 (24.2%)<br>730 (6.5%) | 0.00 | 9,074 (29.2%)<br>2,444 (7.9%) | 9,159 (29.5%)<br>1,954 (6.3%) | -0.01<br>0.06 | 13939 (27.2%)<br>3612 (7.0%) | 14046 (27.4%)<br>3125 (6.1%) | 0.00<br>0.04 |
| Use of Low Intensity Statins; n (%) | 3,159 (35.3%) | 3,116 (34.8%) | 0.00 | 3,741 (33.1%) | 3,933 (34.8%) | -0.04 | 11,556 (37.2%) | 11,429 (36.8%) | 0.01 | 18456 (36.0%) | 18478 (36.0%) | 0.04 |
| Use of High Intensity Statins; n (%) | 2,354 (26.3%) | 2,408 (26.9%) | -0.01 | 2,939 (26.0%) | 2,814 (24.9%) | 0.03 | 7,959 (25.6%) | 8,167 (26.3%) | -0.02 | 13252 (25.8%) | 13389 (26.1%) | -0.01 |
| Malignant hypertension; n (%) | 463 (5.2%) | 450 (5.0%) | 0.01 | 5,386 (47.7%) | 5,398 (47.8%) | 0.00 | 9,493 (30.6%) | 9,631 (31.0%) | -0.01 | 15342 (29.9%) | 15479 (30.2%) | -0.01 |
| Cardiovascular stress test; n (%) | 38 (0.4%) | 40 (0.4%) | 0.00 | 84 (0.7%) | 73 (0.6%) | 0.01 | 312 (1.0%) | 270 (0.9%) | 0.01 | 434 (0.8%) | 383 (0.7%) | 0.01 |
| Echocardiogram; n (%) | 3,953 (44.2%) | 4,195 (46.9%) | -0.05 | 5,226 (46.2%) | 5,820 (51.5%) | -0.11 | 18,321 (59.0%) | 19,059 (61.3%) | -0.05 | 27500 (53.6%) | 29074 (56.7%) | -0.06 |
| Number of BNP tests | | | | | | | | | | | | |
| mean (sd) | 0.15 (0.52) | 0.15 (0.53) | 0.00 | 0.08 (0.40) | 0.09 (0.40) | -0.03 | 0.25 (0.65) | 0.27 (0.66) | -0.03 | 0.20 (0.58) | 0.21 (0.59) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.63) | 0.00 (0.64) | 0.00 |
| Number of Cardias his markers tests (transin CV MADs MA | realehin CDV) | | | | | | | | | | | |
| Number of Cardiac biomarkers tests (tropnin, CK-MBs, Mymean (sd) | 0.45 (1.43) | 0.49 (1.47) | -0.03 | 0.32 (1.24) | 0.39 (1.40) | -0.05 | 0.36 (0.71) | 0.41 (0.73) | -0.07 | 0.37 (1.00) | 0.42 (1.06) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.26) | 0.00 (1.37) | 0.00 |
| eddi fedd | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.20) | 0.00 (1.57) | 0.00 |
| Number of Ambulatory Blood pressure monitoring tests | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.04) | 0.00 (0.04) | 0.00 | 0.00 (0.03) | 0.00 (0.04) | 0.00 | 0.00 (0.03) | 0.00 (0.04) | 0.00 | 0.00 (0.03) | 0.00 (0.04) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.04) | 0.00 (0.05) | 0.00 |
| N of days on antihypertensive medications during baseline | | 407.05 (50.00) | | 400 70 (50 00) | 400 00 (50 70) | | 447.57 (55.70) | 447.05 (55.04) | | 444 47 (50 57) | 440.07/50.00\ | |
| mean (sd) | 139.61 (62.26) | 137.95 (63.30) | 0.03 | 139.79 (63.30) | 139.00 (63.70) | 0.01<br>0.02 | 147.57 (55.78) | 147.35 (55.84) | 0.00 | 144.47 (58.67) | 143.87 (58.99) | 0.00 |
| median [IQR] 1' N of days in database anytime prior | 74.00 [123.00, 181.00] | 174.00 [117.00, 181.00] | 0.00 | 176.00 [125.00, 181.00] | 175.00 [121.00, 181.00] | 0.02 | 176.00 [144.00, 181.00] | 176.00 [144.00, 181.00] | 0.00 | 107.85 (70.61) | 107.63 (71.01) | 0.00 |
| mean (sd) | 2,041.05 (1,371.23) | 2,042.84 (1,399.19) | 0.00 | 2,552.38 (1,366.73) | 2,530.20 (1,365.03) | 0.02 | 811.15 (547.72) | 817.84 (520.25) | -0.01 | 1409.06 (959.60) | 1408.54 (956.85) | 0.00 |
| ·····car (sa) | 1,782.50 [856.75, | 1,747.50 [822.00, | 0.00 | 2,552.50 (2,500.75) | 2,550.20 (2,505.05) | 0.02 | 011.13 (317.72) | 017.07(320.23) | 0.01 | 1103.00 (333.00) | 1100.51 (550.05) | 0.00 |
| median [IQR] | 3,039.00] | 3,082.00] | 0.03 98 | 8.50 [1,338.00, 3,690.00] 3 | 4.00 [1,285.00, 3,667.00] | 0.01 | 634.00 [462.00, 963.00] | 649.00 [484.00, 971.00] | -0.03 | 1022.66 (1280.79) | 1016.66 (1278.03) | 0.00 |
| Mean Copay for per prescription cost (charges in U.S. \$) (1 | 80-1 day prior) | | | | | | | | | | | |
| mean (sd) | 29.02 (37.48) | 29.19 (41.67) | 0.00 | 18.71 (20.72) | 18.78 (20.05) | 0.00 | 117.00 (89.10) | 118.16 (110.23) | -0.01 | 80.01 (71.73) | 80.76 (88.02) | 0.00 |
| median [IQR] | 18.33 [7.69, 36.56] | 18.77 [8.00, 35.85] | -0.01 | 14.04 [6.59, 24.85] | 14.11 [6.77, 25.00] | 0.00 | 95.83 [68.28, 137.63] | 95.81 [68.80, 135.71] | 0.00 | 27.39 (72.88) | 27.48 (88.90) | 0.00 |
| Missing; n (%) | 194 (2.2%) | 201 (2.2%) | 0.00 | 227 (2.0%) | 242 (2.1%) | -0.01 | 403 (1.3%) | 429 (1.4%) | -0.01 | 824 (1.6%) | 872 (1.7%) | -0.01 |
| Colonoscopy; n (%) | 235 (2.6%) | 238 (2.7%) | -0.01 | 344 (3.0%) | 357 (3.2%) | -0.01 | 1,007 (3.2%) | 974 (3.1%) | 0.01 | 1586 (3.1%) | 1569 (3.1%) | 0.00 |
| Fecal occult blood (FOB) test; n (%) Flu vaccine; n (%) | 274 (3.1%)<br>1,648 (18.4%) | 282 (3.2%)<br>1,646 (18.4%) | -0.01<br>0.00 | 218 (1.9%)<br>1,355 (12.0%) | 214 (1.9%)<br>1,349 (11.9%) | 0.00 | 787 (2.5%)<br>10,078 (32.4%) | 777 (2.5%)<br>10,060 (32.4%) | 0.00<br>0.00 | 1279 (2.5%)<br>13081 (25.5%) | 1273 (2.5%)<br>13055 (25.4%) | 0.00 |
| Mammogram; n (%) | 1,648 (18.4%)<br>810 (9.1%) | 798 (8.9%) | 0.00 | 1,355 (12.0%) | 1,349 (11.9%) 554 (4.9%) | 0.00 | 2,951 (9.5%) | 2,947 (9.5%) | 0.00 | 4352 (8.5%) | 4299 (8.4%) | 0.00 |
| Pap smear; n (%) | 131 (1.5%) | 130 (1.5%) | 0.00 | 179 (1.6%) | 183 (1.6%) | 0.00 | 515 (1.7%) | 531 (1.7%) | 0.00 | 825 (1.6%) | 844 (1.6%) | 0.00 |
| | 151 (1.570) | 150 (1.570) | 0.00 | 2,3 (2.370) | 105 (1.070) | 5.50 | 313 (1.770) | 331 (1.770) | 0.00 | 323 (2.070) | 3 (2.070) | 0.00 |

| | 4.007 (4.4.60) | 4 007 (4 4 40) | | 550 (5.00) | 572 (5.00() | | 5 404 (40 00) | 6 407 (40 70) | | 0440 (45 00) | 0055 (45 70) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Pneumonia vaccine; n (%) PSA test or Prostate exam for DRE; n (%) | 1,307 (14.6%)<br>1,089 (12.2%) | 1,287 (14.4%)<br>1,079 (12.1%) | 0.01<br>0.00 | 660 (5.8%)<br>739 (6.5%) | 672 (5.9%)<br>749 (6.6%) | 0.00 | 6,181 (19.9%)<br>3,184 (10.2%) | 6,107 (19.7%)<br>3,210 (10.3%) | 0.01<br>0.00 | 8148 (15.9%)<br>5012 (9.8%) | 8066 (15.7%)<br>5038 (9.8%) | 0.01<br>0.00 |
| Bone mineral density; n (%) | 309 (3.5%) | 299 (3.3%) | 0.00 | 168 (1.5%) | 158 (1.4%) | 0.00 | 1,103 (3.6%) | 1,076 (3.5%) | 0.00 | 1580 (3.1%) | 1533 (3.0%) | 0.00 |
| Use of Sympatomimetic agents; n (%) | 23 (0.3%) | 24 (0.3%) | 0.00 | 50 (0.4%) | 51 (0.5%) | -0.01 | 76 (0.2%) | 91 (0.3%) | -0.02 | 149 (0.3%) | 166 (0.3%) | 0.00 |
| Use of CNS stimulants; n (%) | 23 (0.3%) | 25 (0.3%) | 0.00 | 49 (0.4%) | 49 (0.4%) | 0.00 | 82 (0.3%) | 68 (0.2%) | 0.02 | 154 (0.3%) | 142 (0.3%) | 0.00 |
| Use of estrogens, progestins, androgens; n (%) | 250 (2.8%) | 225 (2.5%) | 0.02 | 456 (4.0%) | 456 (4.0%) | 0.00 | 856 (2.8%) | 904 (2.9%) | -0.01 | 1562 (3.0%) | 1585 (3.1%) | -0.01 |
| Use of Angiogenesis inhibitors; n (%) | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 4 (0.0%) | 3 (0.0%) | #DIV/0! | ** | 12 (0.0%) | #VALUE! | #VALUE! | 16 (0.0%) | #VALUE! |
| Use of Oral Immunosuppressants; n (%) | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 6 (0.1%) | 2 (0.0%) | 0.04 | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Use of fondaparinux or Bivalirudin; n (%) | 4 (0.0%) | 1 (0.0%) | #DIV/0! | 3 (0.0%) | 3 (0.0%) | #DIV/0! | ** | 11 (0.0%) | #VALUE! | #VALUE! | 15 (0.0%) | #VALUE! |
| ,,, | . (0.07-) | _ () | | - () | - () | , | | == (******) | | | (0.0.0, | |
| Use of other direct thrombin inhibitors (lepirudin, des | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of Ticagrelor ON CED; n (%) | 10 (0.1%) | 14 (0.2%) | -0.03 | 21 (0.2%) | 13 (0.1%) | 0.03 | 12 (0.0%) | 15 (0.0%) | #DIV/0! | 43 (0.1%) | 42 (0.1%) | 0.00 |
| Use of Ticagrelor; n (%) | 22 (0.2%) | 26 (0.3%) | -0.02 | 24 (0.2%) | 18 (0.2%) | 0.00 | 110 (0.4%) | 101 (0.3%) | 0.02 | 156 (0.3%) | 145 (0.3%) | 0.00 |
| Number of D-dimer tests | | | | | | | | | | | | |
| mean (sd) | 0.03 (0.21) | 0.03 (0.19) | 0.00 | 0.02 (0.16) | 0.02 (0.17) | 0.00 | 0.05 (0.23) | 0.05 (0.23) | 0.00 | 0.04 (0.21) | 0.04 (0.21) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.23) | 0.00 (0.24) | 0.00 |
| Numbe of CRP, high-sensitivity CRP tests | | | | | | | | | | | | |
| mean (sd) | 0.06 (0.35) | 0.06 (0.30) | 0.00 | 0.03 (0.22) | 0.03 (0.24) | 0.00 | 0.09 (0.41) | 0.09 (0.45) | 0.00 | 0.07 (0.37) | 0.07 (0.39) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.39) | 0.00 (0.42) | 0.00 |
| Number of PT or aPTTt tests | 0.50 (4.00) | 0.40/4.40\ | | 0.00(4.40) | 0.07 (4.00) | | 0.40/4.04 | 0.40(4.05) | | 0.47(4.04) | 0.45(4.07) | |
| mean (sd) | 0.52 (1.32) | 0.48 (1.43) | 0.03 | 0.39 (1.18) | 0.37 (1.20) | 0.02 | 0.49 (1.24) | 0.48 (1.25) | 0.01 | 0.47 (1.24) | 0.46 (1.27) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.44) | 0.00 (1.47) | 0.00 |
| Number of Bleeding time tests<br>mean (sd) | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.00 (0.01) | 0.00 (0.01) | 0.00 | 0.00 (0.01) | 0.00 (0.01) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | #DIV/0! | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | #DIV/0! | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.01) | 0.00 (0.01) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | #510/0: | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | #DIV/0: | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.01) | 0.00 (0.01) | 0.00 |
| mean (sd) | 3.41 (0.76) | 3.40 (0.76) | 0.01 | 3.29 (0.77) | 3.29 (0.76) | 0.00 | 3.56 (0.74) | 3.55 (0.73) | 0.01 | 3.47 (0.75) | 3.47 (0.74) | 0.00 |
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 1.84 (0.89) | 1.84 (0.88) | 0.00 |
| N of Generic name drugs | () | (,, | | () | (,, | | (,) | (,, | | | () | |
| mean (sd) | 19.22 (14.62) | 19.38 (16.57) | -0.01 | 14.89 (10.15) | 14.82 (11.14) | 0.01 | 20.43 (14.14) | 20.47 (15.60) | 0.00 | 19.00 (13.45) | 19.04 (14.92) | 0.00 |
| median [IQR] | 16.00 [10.00, 24.00] | 15.00 [9.00, 25.00] | 0.06 | 13.00 [8.00, 19.00] | 12.00 [7.00, 19.00] | 0.09 | 17.00 [11.00, 26.00] | 17.00 [10.00, 26.00] | 0.00 | 9.40 (14.86) | 9.00 (16.44) | 0.00 |
| N of Brand name drugs | | | | | | | | | | | | |
| mean (sd) | 4.15 (6.18) | 4.22 (4.32) | -0.01 | 4.70 (5.32) | 4.76 (4.21) | -0.01 | 4.78 (6.13) | 4.92 (5.14) | -0.02 | 4.65 (5.97) | 4.76 (4.81) | 0.00 |
| median [IQR] | 2.00 [0.00, 6.00] | 3.00 [1.00, 6.00] | -0.19 | 3.00 [1.00, 7.00] | 4.00 [2.00, 7.00] | -0.21 | 3.00 [1.00, 7.00] | 3.00 [1.00, 7.00] | 0.00 | 1.67 (6.82) | 2.06 (5.48) | 0.00 |
| Use of clopidogrel; n (%) | 1,027 (11.5%) | 1,017 (11.4%) | 0.00 | 1,382 (12.2%) | 1,356 (12.0%) | 0.01 | 4,482 (14.4%) | 4,428 (14.3%) | 0.00 | 6891 (13.4%) | 6801 (13.3%) | 0.00 |
| Systemic embolism; n (%) | 70 (0.8%) | 67 (0.7%) | 0.01 | 87 (0.8%) | 86 (0.8%) | 0.00 | 324 (1.0%) | 306 (1.0%) | 0.00 | 481 (0.9%) | 459 (0.9%) | 0.00 |
| DVT; n (%) | 23 (0.3%) | 29 (0.3%) | 0.00 | 25 (0.2%) | 24 (0.2%) | 0.00 | 562 (1.8%) | 559 (1.8%) | 0.00 | 610 (1.2%) | 612 (1.2%) | 0.00 |
| PE; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 144 (0.5%) | 141 (0.5%) | 0.00 | 144 (0.3%) | 141 (0.3%) | 0.00 |
| | 2.050 (2.4.00) | 2 442 (24 20) | | 2 5 2 2 (2 4 7 2 ( ) | 2 504 (24 00) | | 40.704/44.40/ | 10.055 (11.50) | | 22.425 (22.20) | 20552 (40 40) | |
| Diabetes: 1 inpatient or 2 outpatient claims within 18 | 3,058 (34.2%) | 3,112 (34.8%) | -0.01 | 3,583 (31.7%) | 3,591 (31.8%) | 0.00 | 13,784 (44.4%) | 13,855 (44.6%) | 0.00 | 20425 (39.8%) | 20558 (40.1%) | -0.01 |
| Intracranial or retroperitoneal hemorrhage: 1 inpatier | 13 (0.1%) | 12 (0.1%) | 0.00 | 15 (0.1%) | 17 (0.2%) | -0.03 | 101 (0.3%) | 99 (0.3%) | 0.00 | 129 (0.3%) | 128 (0.2%) | 0.02 |
| Peptic Ulcer Disease; n (%) | 1,514 (16.9%) | 1,506 (16.8%) | 0.00 | 1,294 (11.5%) | 1,278 (11.3%) | 0.01 | 7,115 (22.9%) | 7,038 (22.7%) | 0.00 | 9923 (19.3%) | 9822 (19.1%) | 0.01 |
| Upper GI bleed; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 22 (0.1%) | 26 (0.1%) | 0.00 | 22 (0.0%) | 26 (0.1%) | -0.04 |
| Lower/ unspecified GI bleed; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 395 (1.3%) | 385 (1.2%) | 0.01 | 395 (0.8%) | 385 (0.8%) | 0.00 |
| Urogenital bleed; n (%) | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 527 (1.7%) | 533 (1.7%) | 0.00 | 527 (1.0%) | 534 (1.0%) | 0.00 |
| Other bleeds; n (%) | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 328 (1.1%) | 314 (1.0%) | 0.01 | 329 (0.6%) | 315 (0.6%) | 0.00 |
| Prior cancer; n (%) | 1,130 (12.6%) | 1,119 (12.5%) | 0.00 | 1,106 (9.8%) | 1,063 (9.4%) | 0.01 | 4,090 (13.2%) | 4,060 (13.1%) | 0.00 | 6326 (12.3%) | 6242 (12.2%) | 0.00 |
| Aspirin; n (%) | 68 (0.8%) | 71 (0.8%) | 0.00 | 186 (1.6%) | 184 (1.6%) | 0.00 | 201 (0.6%) | 201 (0.6%) | 0.00 | 455 (0.9%) | 456 (0.9%) | 0.00 |
| Aspirin/dipyridamole; n (%) | 37 (0.4%) | 32 (0.4%) | 0.00 | 79 (0.7%) | 75 (0.7%) | 0.00 | 180 (0.6%) | 185 (0.6%) | 0.00 | 296 (0.6%) | 292 (0.6%) | 0.00 |
| Other antiplatelet agents; n (%) | 48 (0.5%) | 46 (0.5%) | 0.00 | 62 (0.5%) | 71 (0.6%) | -0.01 | 215 (0.7%) | 224 (0.7%) | 0.00 | 325 (0.6%) | 341 (0.7%) | -0.01 |
| PGP inhibitors; n (%) | 3,868 (43.2%) | 3,887 (43.4%) | 0.00 | 5,184 (45.9%) | 5,203 (46.0%) | 0.00 | 15,745 (50.7%) | 15,746 (50.7%) | 0.00 | 24797 (48.3%) | 24836 (48.4%) | 0.00 |
| Other gastroprotective agents; n (%) | 81 (0.9%) | 86 (1.0%) | -0.01 | 125 (1.1%) | 122 (1.1%) | 0.00 | 461 (1.5%) | 459 (1.5%) | 0.00 | 667 (1.3%) | 667 (1.3%) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.66 (0.84) | 0.65 (0.79) | 0.01 | 0.29 (0.74) | 0.30 (0.70) | -0.01 | 0.72 (0.84) | 0.72 (0.84) | 0.00 | 0.61 (0.82) | 0.62 (0.80) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 0.22 (0.94) | 0.22 (0.91) | 0.00 |
| Proton pump inhibitor; n (%) | 1,891 (21.1%)<br>406 (4.5%) | 1,928 (21.5%)<br>402 (4.5%) | -0.01<br>0.00 | 2,511 (22.2%)<br>429 (3.8%) | 2,460 (21.8%)<br>425 (3.8%) | 0.01<br>0.00 | 8,637 (27.8%)<br>2,128 (6.8%) | 8,657 (27.9%)<br>2,152 (6.9%) | 0.00 | 13039 (25.4%)<br>2963 (5.8%) | 13045 (25.4%)<br>2979 (5.8%) | 0.00<br>0.00 |
| H2 receptor antagonist; n (%) Vitamin K therapy; n (%) | 4 (0.0%) | 402 (4.5%)<br>3 (0.0%) | #DIV/0! | 429 (3.8%)<br>5 (0.0%) | 425 (3.8%) 4 (0.0%) | #DIV/0! | ∠,120 (D.0%)<br>** | ±,±32 (0.97%) | #VALUE! | 2963 (5.8%)<br>#VALUE! | 2979 (5.8%)<br>#VALUE! | #VALUE! |
| Number of neurologist visits | 4 (0.070) | 3 (0.070) | #DIV/U: | 3 (0.0%) | 4 (0.070) | #DIV/U: | | | #YALUL! | #VALUL: | #VALUE! | #VALUE: |
| mean (sd) | 0.32 (1.39) | 0.31 (1.36) | 0.01 | 0.25 (1.17) | 0.25 (1.37) | 0.00 | 0.55 (2.12) | 0.54 (2.05) | 0.00 | 0.44 (1.83) | 0.44 (1.81) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.97) | 0.00 (2.00) | 0.00 |
| Number of INR (prothrombin) tests ordered | (,) | | | | | | () | | | () | ( ) | |
| mean (sd) | 0.37 (1.01) | 0.33 (1.10) | 0.04 | 0.28 (0.89) | 0.26 (0.93) | 0.02 | 0.47 (1.19) | 0.46 (1.21) | 0.01 | 0.41 (1.10) | 0.39 (1.13) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.23) | 0.00 (1.27) | 0.00 |
| Treating prescriber - Cardiologist; n (%) | 5,550 (62.0%) | 5,429 (60.7%) | 0.03 | 5,961 (52.8%) | 5,881 (52.0%) | 0.02 | 21,163 (68.1%) | 20,800 (66.9%) | 0.03 | 32674 (63.7%) | 32110 (62.6%) | 0.02 |
| Treating prescriber - Primary Care Physician; n (%) | 5,841 (65.3%) | 5,877 (65.7%) | -0.01 | 3,792 (33.6%) | 3,789 (33.5%) | 0.00 | 9,315 (30.0%) | 9,328 (30.0%) | 0.00 | 18948 (36.9%) | 18994 (37.0%) | 0.00 |
| Treating prescriber - Other; n (%) | 7,646 (85.4%) | 7,591 (84.8%) | 0.02 | 9,048 (80.1%) | 8,979 (79.5%) | 0.01 | 27,784 (89.4%) | 27,618 (88.9%) | 0.02 | 44478 (86.7%) | 44188 (86.1%) | 0.02 |

| Alpha blockers; n (%)<br>CHADS2 score, 180 days, V | 1,102 (12.3%) | 1,081 (12.1%) | 0.01 | 1,377 (12.2%) | 1,405 (12.4%) | -0.01 | 3,766 (12.1%) | 3,807 (12.3%) | -0.01 | 6245 (12.2%) | 6293 (12.3%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 2.10 (1.19) | 2.11 (1.19) | -0.01 | 2.19 (1.18) | 2.20 (1.19) | -0.01 | 3.73 (1.65) | 3.73 (1.64) | 0.00 | 3.11 (1.48) | 3.11 (1.48) | 0.00 |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.00 | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.00 | 3.00 [3.00, 5.00] | 3.00 [3.00, 5.00] | 0.00 | 1.45 (1.65) | 1.45 (1.65) | 0.00 |
| Use of Prasugrel; n (%) | 25 (0.3%) | 24 (0.3%) | 0.00 | 40 (0.4%) | 30 (0.3%) | 0.02 | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Osc Off Tasagrei, ii (70) | 25 (0.570) | 24 (0.370) | 0.00 | 40 (0.470) | 30 (0.370) | 0.02 | | | #VALUE: | #VALUE: | #VALUE: | #VALUE: |
| Use of Loop Diuretics+other diuretics+other hyperten: | 3,023 (33.8%) | 3,035 (33.9%) | 0.00 | 3,753 (33.2%) | 3,790 (33.5%) | -0.01 | 13,931 (44.8%) | 14,150 (45.5%) | -0.01 | 20707 (40.4%) | 20975 (40.9%) | -0.01 |
| Commercial vs Medicare Advantage- Business Type Code - Co | ORRECT ONE - OPTUM | | | | | | 0 | 0 | | | | |
| Commercial; n (%) | 1461 (16.3%) | 1463 (16.3%) | 0.00 | 9,248 (81.8%) | 9,258 (81.9%) | 0.00 | - | - | #VALUE! | 10,709 (52.9%) | 10,721 (52.9%) | 0.00 |
| Medicare Advantage; n (%) | 7,489 (83.7%) | 7487 (83.7%) | 0.00 | 2,052 (18.2%) | 2,042 (18.1%) | 0.00 | - | - | #VALUE! | 9,541 (47.1%) | 9,529 (47.1%) | 0.00 |
| Commercial vs Medicare Advantage- Business Type Code | | | | | | | | | | | | |
| COM = COMMERCIAL; n (%) | 1,461 (16.3%) | 1,463 (16.3%) | 0.00 | _ | - | #VALUE! | - | - | #VALUE! | 1,461 (16.3%) | 1,463 (16.3%) | 0.00 |
| MCR = MEDICARE; n (%) | 7,489 (83.7%) | 7,487 (83.7%) | 0.00 | _ | - | #VALUE! | - | - | #VALUE! | 7,489 (83.7%) | 7,487 (83.7%) | 0.00 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | _ | - | #VALUE! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| | - () | - () | , | | | | | | | - () | - () | |
| NONE = NO BUSINESS LINE CODE (added in 2015); n ( | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data Type | - | - | | 0 | 0 | | - | - | | | | |
| 1 - Fee For Service; n (%) | - | = | | 1,803 (16.0%) | 1,817 (16.1%) | | - | - | | 1,803 (16.0%) | 1,817 (16.1%) | 0.00 |
| 2 - Encounter; n (%) | - | = | | 249 (2.2%) | 225 (2.0%) | | - | - | | 249 (2.2%) | 225 (2.0%) | 0.00 |
| 3 - Medicare; n (%) | - | = | | 8,539 (75.6%) | 8,523 (75.4%) | | - | - | | 8,539 (75.6%) | 8,523 (75.4%) | 0.00 |
| 4 - Medicare Encounter; n (%) | - | - | | 709 (6.3%) | 735 (6.5%) | | - | - | | 709 (6.3%) | 735 (6.5%) | 0.00 |
| Metropolitan Statistical Area - Urban (any MSA) vs Rural (no | n-MSA) | | | | | | | | | 0 | 0 | 0.00 |
| Urban; n (%) | · - | - | | 8,353 (73.9%) | 8,402 (74.4%) | | = | - | | 8,353 (73.9%) | 8,402 (74.4%) | 0.00 |
| Rural; n (%) | - | - | | 295 (2.6%) | 286 (2.5%) | | = | - | | 295 (2.6%) | 286 (2.5%) | 0.00 |
| Unknown/Missing; n (%) | - | - | | 2,652 (23.5%) | 2,612 (23.1%) | | = | - | | 2,652 (23.5%) | 2,612 (23.1%) | 0.00 |
| | | | | , (====-, | , = (=====, | Dur | a to CMS call suppression n | olicy all values less than 1 | 1 are denoted | , (==:=-, | , = (=====,-, | |

Due to CMS cell suppression policy, all values less than 11 are denoted